| <b>gsk</b> GlaxoSmithKline | Statistical Analysis Plan |
|---|---|
| Detailed Title: | A Phase 1/2, randomized, observer-blind, controlled, multi-center, dose-escalation study to evaluate safety, reactogenicity and immunogenicity of GSK Biologicals' respiratory syncytial virus (RSV) investigational vaccine based on the RSV viral proteins F, N and M2-1 encoded by chimpanzee-derived adenovector (ChAd155-RSV) (GSK3389245A), when administered intramuscularly according to a 0, 1-month schedule to RSV-seropositive infants aged 12 to 23 months |
| eTrack study number and<br>Abbreviated Title | 204838 (RSV PED-002) |
| Scope: | All data pertaining to the above study. |
| Date of Statistical Analysis<br>Plan | Final: 28-Mar-2018 |
| Co-ordinating author: | (Study Statistician) |
| Reviewed by: | PPD (Clinical and Epidemiology Project Lead) PPD (Clinical Research and Development Lead) PPD (Lead statistician) PPD (Lead statistical analyst) PPD (Scientific writer) PPD (Regulatory Affairs) PPD (SERM physician) Mandatory (Public disclosure representative) PPD (Head CLS) PPD (Senior Manager, Immuno Lab Platform3) PPD (Expert Scientist, Biology Molecular) |
| Approved by: | PPD (Lead ADaM CEO Head) PPD (Clinical and Epidemiology Project Lead), PPD (Clinical Research and Development Lead, PPD (Lead statistician), PPD (Lead Scientific writer) PPD (Lead stat Analyst) |

APP 9000058193 Statistical Analysis Plan Template (Effective date: 14 April 2017)

204838 (RSV PED-002) Statistical Analysis Plan Final

## **TABLE OF CONTENTS**

| | | | | PAGE |
|---|---|---|---|---|
| LIS | T OF A | BBREVIA | ATIONS | 10 |
| 1. | DOC | JMENT H | IISTORY | 12 |
| 2. | STUD | Y DESIG | N | 12 |
| 3. | OBJE | CTIVES | | 16 |
| | 3.1. | Primary | objective | 16 |
| | 3.2. | Seconda | ary objectives | 16 |
| | 3.3. | | objectives | |
| 4. | ENDF | POINTS | | 16 |
| | 4.1. | | endpoints | |
| | 4.2. | Seconda | ary endpoints | 17 |
| | 4.3. | Tertiary | endpoints | 18 |
| 5. | ANAI | YSIS SET | TS | 18 |
| ٥. | 5.1. | | on | |
| | 0 | 5.1.1. | | |
| | | 5.1.2. | According-to-protocol cohort for analysis of | |
| | | | immunogenicity | 18 |
| | 5.2. | | for eliminating data from Analysis Sets | |
| | | 5.2.1. | | |
| | | 5.2.2. | Elimination from Per-protocol analysis Set (PPS) | |
| | | | 5.2.2.1. Excluded subjects | |
| | | | 5.2.2.2. Right censored Data | |
| | | | 5.2.2.3. Visit-specific censored Data | 21 |
| | 5.3. | Importai<br>protocol | nt protocol deviation not leading to elimination from per- I analysis set | 22 |
| 6. | СТАТ | ISTICAL | ANALYSES | 22 |
| 0. | 6.1. | | raphy | |
| | 0.1. | 6.1.1. | Analysis of demographics/baseline characteristics planned | t |
| | | _ | in the protocol | |
| | 6.2. | | ogenicity | |
| | | 6.2.1. | Analysis of immunogenicity planned in the protocol | |
| | | | 6.2.1.1. CMI analysis | |
| | | | 6.2.1.2. Humoral immune response | |
| | 6.3. | | s of RSV incidence | |
| | 6.4. | | s of safety | |
| | | 6.4.1. | Analysis of safety planned in the protocol | |
| | | | 6.4.1.1. Within groups assessment | |
| | | 0.40 | 6.4.1.2. Between groups assessment | |
| | | 6.4.2. | Additional considerations | |
| | | | 6.4.2.1. Additional safety analysis | 29 |
| | | | 6.4.2.2. Exclusion of implausible solicited Adverse | 29 |
| | | | ⊏ V H I II | /9 |

| | 6.4.2.3. Combined Solicited and Unsolicited Adverse Events | 29 |
|---|---|---|
| 7. | ANALYSIS INTERPRETATION | 30 |
| 8. | CONDUCT OF ANALYSES | 30 |
| 9. | CHANGES FROM PLANNED ANALYSES | 31 |
| 10. | LIST OF FINAL REPORT TABLES, LISTINGS AND FIGURES | 32 |
| 11. | ANNEX 1 STANDARD DATA DERIVATION RULE AND STATISTICAL METHODS | 33<br>33<br>33<br>34<br>35<br>37 |
| 12. | ANNEX 2: RELEVANT PREFERRED TERMS FOR DETECTION OF AESI | 41 |
| 13. | ANNEX 3: STUDY SPECIFIC MOCK TFL | 47 |

204838 (RSV PED-002) Statistical Analysis Plan Final

## **LIST OF TABLES**

| | | PAGE |
|---|---|---|
| Table 1 | Study groups and epochs foreseen in the study | 14 |
| Table 2 | Implausible Solicited Adverse Events | 29 |
| Table 3 | Endpoints assessed at different analysis time points | 31 |
| Table 4 | Toxicity grading scales for hematology and biochemistry parameters applicable for this study | 38 |
| Table 5 | Case definition of RSV- RTI/LRTI | 39 |

204838 (RSV PED-002) Statistical Analysis Plan Final

## **LIST OF FIGURES**

| | | PAGE |
|---|---|---|
| Figure 1 | Study design | 12 |
| Figure 2 | Individuals results of hemoglobin levels in < group> <exposed set=""></exposed> | 70 |
| Figure 3 | Reverse cumulative distribution curves for anti-RSV-A neutralising antibody titres in each group at baseline and <d60 d365=""> <pps analysis="" at="" day="" for="" immunogenicity="" of="" x=""></pps></d60> | 86 |
| Figure 4 | Individual results of anti-RSV-A neutralising antibody titre at Day <60/365> versus pre-vaccination in <each group=""> and Control group&gt; <pps analysis="" at="" day="" for="" immunogenicity="" of="" x=""></pps></each> | 87 |
| Figure 5 | Boxplots of individual data for CD4+ T-cells expressing at least two markers among CD40L, IL-2, TNF-α, and IFN-γ upon stimulation with <rsv combined="" f="" m2-1="" n=""> peptide pool <from 366="" 61="" day="" pre-vaccination="" to=""> <pps analysis="" at="" day="" for="" immunogenicity="" of="" x=""></pps></from></rsv> | |
| Figure 6 | Co-expression profile of the RSV <f m2-1="" n=""> specific <cd4+> T-cells expressing at least two markers among CD40L, IL-2, TNF-α, and IFN-γ in <rsv-ld group=""> <pps analysis="" at="" day="" for="" immunogenicity="" of="" x=""></pps></rsv-ld></cd4+></f> | 90 |

204838 (RSV PED-002) Statistical Analysis Plan Final

## **LIST OF TEMPLATES**

| | | PAGE |
|---|---|---|
| Template 1 | Number of subjects by country and center <exposed set=""></exposed> | 48 |
| Template 2 | Number of subjects vaccinated, completed and withdrawn with reason for withdrawal – up to Day X <exposed set=""></exposed> | 48 |
| Template 3 | Visit attendance <exposed set=""></exposed> | 49 |
| Template 4 | Number of subjects enrolled into the study as well as the number of subjects excluded from the PPS analysis of immunogenicity at Day X with reasons for exclusion | 49 |
| Template 5 | Summary of demographic characteristics <exposed set=""></exposed> | 50 |
| Template 6 | Summary of vital signs characteristics <exposed set=""></exposed> | 51 |
| Template 7 | Distribution of weight for age Z-score (WAZ) at vaccination <exposed set=""></exposed> | 52 |
| Template 8 | Distribution of height for age Z-score (HAZ) at vaccination <exposed set=""></exposed> | 52 |
| Template 9 | Deviations from specifications for age and intervals between study visits up to Day X <exposed set=""></exposed> | 53 |
| Template 10 | Study Population | 53 |
| Template 11 | Number of enrolled subjects by country | 54 |
| Template 12 | Number of enrolled subjects by age category | 54 |
| Template 13 | Minimum and maximum activity dates <exposed set=""></exposed> | 54 |
| Template 14 | Exposure to study vaccines <exposed set=""></exposed> | 55 |
| Template 15 | Compliance in completing solicited symptoms information <exposed set=""></exposed> | 55 |
| Template 16 | Incidence and nature of symptoms (solicited and unsolicited) reported during the 7-day post-vaccination period (Days 1-7) following each dose and overall <exposed set=""></exposed> | 56 |
| Template 17 | Incidence of solicited local symptoms reported during the 7-day (Days 1-7) post-vaccination period following each dose and overall <exposed set=""></exposed> | 57 |
| Template 18 | Incidence of solicited local symptoms reported during the 7-day (Days 1-7) post-vaccination period following each dose and overall by maximum grading <exposed set=""></exposed> | 58 |

| Template 19 | Incidence of solicited general symptoms reported during the 7-day (Days 1-7) post-vaccination period following each dose and overall <exposed set=""></exposed> | 60 |
|---|---|---|
| Template 20 | Incidence of solicited general symptoms reported during the 7-day (Days 1-7) post-vaccination period following each dose and overall by maximum grading <exposed set=""></exposed> | 62 |
| Template 21 | Maximum Temperature reported during the 7-day (Days 1-7) post-vaccination period – dose X <exposed set=""></exposed> | 65 |
| Template 22 | Percentage of subjects reporting the occurrence of unsolicited symptoms classified by MedDRA Primary System Organ Class and Preferred Term within the 30-day (Days 1-30) post-vaccination period <exposed set=""></exposed> | 65 |
| Template 23 | Number and percentage of subjects taking a concomitant medication during the 7- day (Days 1-7) post -vaccination period <exposed set=""></exposed> | 66 |
| Template 24 | Distribution of change from baseline in hematology and biochemistry with respect to normal laboratory ranges <exposed set=""></exposed> | 67 |
| Template 25 | Summary of hematology and biochemistry results by maximum grade from VISIT X (DX) up to VISIT Y (DY) – post dose 1 of vaccination versus baseline <exposed set=""></exposed> | 68 |
| Template 26 | Descriptive statistics table on eosinophils, basophils, and monocytes counts for subjects <exposed set=""></exposed> | 69 |
| Template 27 | Exploratory comparisons between groups in terms of percentage of subjects reported any Grade 2/3 AE and/or any fever >38.5°C and/or any vaccine-related SAE during the 7-day (Days 1-7) post-vaccination period <exposed set=""></exposed> | 71 |
| Template 28 | Percentage of subjects reporting episode of spontaneous or excessive bleeding (AE of specific interest) classified by MedDRA Primary System Organ Class and Preferred Term within the 30-day (Days 1-30) post-vaccination period <exposed set=""></exposed> | 72 |
| Template 29 | Solicited and unsolicited symptoms classified by MedDRA Primary System Organ Class and Preferred Term within the 30- day (Days 1-30) post-vaccination period including number of events - SAE excluded <exposed set=""></exposed> | 73 |
| Template 30 | Number (%) of subjects with serious adverse events from vaccination dose 1 up to Day X/Study end including number of events reported <exposed set=""></exposed> | 74 |
| Template 31 | Listing of unscheduled safety visit from vaccination dose 1 up to Day X/study end <exposed set=""></exposed> | 75 |

| Template 32 | Listing of SAEs reported from vaccination dose 1 up to Day X visit /study end <exposed set=""></exposed> | 76 |
|---|---|---|
| Template 33 | Listing of AEs related to LRTI and association to RSV infection from vaccination dose 1 up to Day X visit/study end <exposed set=""></exposed> | 77 |
| Template 34 | Listing of RSV-RTI cases identified according to WHO case definitions and RSV-LRTI reported as AESI from vaccination dose 1 up to Day X visit /study end <exposed set=""></exposed> | 78 |
| Template 35 | Listing of AEs related to spontaneous or excessive bleeding together with hemoglobin and platelet count results from vaccination dose 1 up to Day 60 visit <exposed set=""></exposed> | 79 |
| Template 36 | Listing of adverse events, SAEs and solicited symptoms leading to withdrawal from the study or treatment from vaccination dose 1 up to Day X visit/study end <exposed set=""></exposed> | 80 |
| Template 37 | Number and percentage of subjects with anti-RSV-A neutralising antibody titre equal to or above <cut-off> and GMTs <pps analysis="" at="" day="" for="" immunogenicity="" of="" x=""></pps></cut-off> | 81 |
| Template 38 | Vaccine response for anti-RSV-A neutralising antibody titre at each post-vaccination timepoint <pps analysis="" at="" day="" for="" immunogenicity="" of="" x=""></pps> | 82 |
| Template 39 | Distribution of anti-RSV-A neutralising antibody titer <pps analysis="" at="" day="" for="" immunogenicity="" of="" x=""></pps> | 83 |
| Template 40 | Distribution of fold of anti-RSV-A neutralising antibody titer by pre-vaccination titer category <pps analysis="" at="" day="" for="" immunogenicity="" of="" x=""></pps> | 84 |
| Template 41 | Geometric mean of the individual ratio of anti-RSV-A neutralising antibody titers at each post-vaccination timepoint compared to pre-vaccination with 95% CI <pps analysis="" at="" day="" for="" immunogenicity="" of="" x=""></pps> | 85 |
| Template 42 | Descriptive statistics on the frequency of CD4+ T-cells expressing at least two markers among CD40L, IL-2, TNF-α, and IFN-γ upon stimulation with <rsv combined="" f="" m2-1="" n=""> peptide pool <pps analysis="" at="" day="" for="" immunogenicity="" of="" x=""></pps></rsv> | 88 |
| Template 43 | Number and percentage of subjects with at least one RSV infection, RSV-RTI, RSV-LRTI, RSV-severe LRTI, RSV-very severe LRTI, All-cause LRTI and RSV hospitalization from vaccination dose 1 up to D366/D731 visit <exposed set=""></exposed> | 91 |
| Template 44 | Number and percentage of subjects reporting the RSV infection of different severity by number of events experienced between vaccination dose 1 up to D366/D731 visit <exposed set=""></exposed> | 92 |

| Template 45 | Number and percentage of RSV infections and associated disease severity between vaccination dose 1 up to D366/D731 visit <exposed set=""></exposed> | 93 |
|---|---|---|
| Template 46 | Number and percentage of RSV infections requiring hospitalization between vaccination dose 1 up to D366/D731 <exposed set=""></exposed> | 94 |
| Template 47 | Descriptive statistics of viral load calculated on all qRT-PCR confirmed RSV infection episodes with varying disease severity from vaccination dose 1 up to D366/D731 <exposed set=""></exposed> | 95 |
| Template 48 | Descriptive statistics of maximum viral load per subjects based on qRT-PCR confirmed episode with varying disease severity form vaccination dose 1 up to D366/D731 <exposed set=""></exposed> | 96 |
| Template 49 | Frequency of multiple respiratory pathogen for qRT-PCR confirmed RSV-RTI episodes from vaccination dose 1 up to D366/D731 visit <exposed set=""></exposed> | 97 |
| Template 50 | Frequency of multiple respiratory pathogen for confirmed LRTI episodes from vaccination dose 1 up to D366/D731 visit <exposed set=""></exposed> | 98 |
| Template 51 | Listing of RSV-RTI cases identified according to case definitions <exposed set=""></exposed> | 99 |
| Template 52 | Listing of RSV-RTI requiring hospitalization and type of inpatient facility required <exposed set=""></exposed> | 100 |
| Template 53 | Number and percentage of subjects with highest associated severity of RSV infection from vaccination dose 1 up to D366/D731 visit <exposed set=""></exposed> | 101 |
| Template 54 | Number and percentage of subjects reporting the RSV infection of maximum severity by number of events experienced between vaccination dose 1 up to D366/D731 visit <exposed set=""></exposed> | 102 |
| Template 55 | Number (%) of subjects reported solicited local symptoms during the 7-day (Days 1-7) post-vaccination period following each dose and across doses <exposed set=""></exposed> | 103 |
| Template 56 | Number (%) of subjects reported solicited general symptoms during the 7-day (Days 1-7) post-vaccination period following each dose and across dose <exposed set=""></exposed> | 104 |

204838 (RSV PED-002) Statistical Analysis Plan Final

### LIST OF ABBREVIATIONS

AE Adverse event

AESI Adverse Events of Special Interest

ChAd155- Investigational recombinant chimpanzee adenovirus Type 155-

RSV vectored RSV vaccine

CI Confidence Interval

CMI Cell-mediated immunity

CTRS Clinical Trial Registry Summary

ERD Enhanced RSV disease

ES Exposed Set

GMC Geometric mean antibody concentration

GMT Geometric mean antibody titer

ICH International Conference on Harmonisation

IDMC Independent Data Monitoring Committee

iSRC Internal Safety Review Committee

LL Lower Limit of the confidence interval

LLOQ Lower Limit of Quantification

LRTI Lower respiratory tract infection

MedDRA Medical Dictionary for Regulatory Activities

N.A. Not Applicable

PCA Palivizumab Competing Antibodies

PPS Per Protocol Set RR Respiratory rate

RSV Respiratory syncytial virus

RSV-Hd High dose ChAd155-RSV vaccine (5 x 10<sup>10</sup> vp)
RSV-Ld Low dose ChAd155-RSV vaccine (5 x 10<sup>9</sup> vp)

RSV-Md Middle dose ChAd155-RSV vaccine (1.5 x 10<sup>10</sup> vp)

RSV-RTI Respiratory tract infection associated with RSV infection

RTI Respiratory tract infection

SAE Serious adverse event SAP Statistical Analysis Plan

SD Standard Deviation

SHS Study Headline Summary

204838 (RSV PED-002) Statistical Analysis Plan Final

SR Study Report

TFL Tables Figures and Listings

TOC Table of Content

UL Upper Limit of the confidence interval

## 1. DOCUMENT HISTORY

| Date | Description | Protocol Version |
|-------------|---------------|---------------------------|
| 28-MAR-2018 | Final version | Amendment 4 - 10-DEC-2017 |

### 2. STUDY DESIGN

### Figure 1 Study design

Please note that for the analysis for D61, D366 and D731, the study will be converted in cDISC standard. To avoid confusion between analysis planned and table template, all the text and figures have been changed into cDISC, i.e, Day 'DX' is changed to Day 'DX+1'.



Hd: High dose; IDMC: Independent Data Monitoring Committee; ISRC: Internal Safety Review Committee; Ld: low dose; Md: middle dose; R8V: respiratory syncytial virus; 8CR: screening; 8E; safety evaluation

Hd: High dose; IDMC: Independent Data Monitoring Committee; iSRC: Internal Safety Review Committee; Ld: low dose; Md: middle dose; RSV: respiratory syncytial virus; SCR: Screening; SE: solicited events; vp: viral particles.

- ¥ On Day 4 and Day 34, a visit may take place at the investigators clinical facility or the investigator/clinical staff may call the subjects' parent(s)/LAR(s), as appropriate to the circumstances in the judgment of the investigator.
- a Surveillance for RSV-RTI comprises monthly nasal swab collected to detect asymptomatic RSV infections during RSV season and active and passive surveillance contacts for RSV symptomatic RTI (see Section 9.2 of the protocol). Data about RSV–RTI incidence will be reviewed monthly by an IDMC.
- b Within each step, an iSRC will review all accumulating safety data three weeks after the start of vaccination and then about every three weeks (until the IDMC has reviewed all safety data up to 30 days after administration of Dose 2 in Step 3 i.e. Day 61). The IDMC will review all accumulating reactogenicity and safety data monthly throughout the period of vaccination (up to 30 days after administration of Dose 2 in Step 3, i.e. Day 61) and accumulating SAEs until Day 731. Refer to Sections 9.10.2 and 9.10.3 of the protocol.

204838 (RSV PED-002) Statistical Analysis Plan Final

- c Visit 2 (Day 2), Visit 4 (Day 8), Visit 6 (Day 32), Visit 8 (Day 38) and Visit 11 (Day 731) may take place in the subject's home or at the investigators clinical facility as appropriate to the circumstances in the judgment of the investigator.
- d Dose escalation will proceed after administration of two doses of the vaccine to 32 subjects in Step 1. However, in the absence of a significant safety concern detected in the regular monitoring of accumulating safety data on at least 16 subjects, the IDMC may allow for dose escalation to proceed without the requirement of enrolling and evaluating the full group size of 32 subjects. A subsequent dose escalation (from Step 2 to Step 3) will proceed after administration of two doses of the vaccine to between a maximum of 32 to a minimum of 16 subjects in the absence of a significant safety concern detected by the IDMC in the regular monitoring of accumulating safety data. Thus, upon review of the accumulating safety data on a minimum of 16 subjects after administration of two doses of the vaccine, the IDMC may decide that based on the evolving safety profile, sufficient information has been accumulated to allow safe progression to the next sequential dose level. It will be ensured that, as a minimum the IDMC will have reviewed safety data of at least 16 subjects for two doses and given their formal approval prior to enrolling subjects to the next dose level.
- e Only for hematology.
- f Day 8 hematology testing will be performed if any ≥ Grade 1 for platelet decrease is detected on Day 1 after vaccination; to ensure its resolution. Similarly, hematology testing on Day 38 will be performed if any ≥ Grade 1 for platelet decrease is detected on Day 32.
- g Refer to Section 6.6.11.3 of the protocol
- h The IDMC will perform a review when all safety data up to 30 days after administration of Dose 2 in Step 3 (i.e. Day 61) are available.
- i Blood samples for CMI and for humoral immunogenicity may be postponed until after the RSV serostatus is known and eligibility is confirmed up to or on Day 1 (but before vaccination).
- **Experimental design**: Phase I/II, observer-blind, randomized, placebo-controlled, multi-centric, study with two parallel groups per step in a 3-step staggered design
- **Duration of the study**: approximately 24 months:
  - Epoch 001: primary starting at the Screening visit and ending at Visit 9 (Day 61)
  - Epoch 002: follow-up starting at Visit 10 (Day 366) and ending at Visit 11 (Day 731)

Any safety, immunogenicity and disease surveillance data collected beyond Visit 9 (Day 61) will be collected in Epoch 002

- **Primary completion Date**: Visit 9 (Day 61).
- End of Study: Last testing results released of samples collected at Visit 11 (Day 731). \*
  - \* Up to Visit 11 (Day 731), there will be monthly nasal swab to detect asymptomatic RSV infections during the RSV season and if following active or a passive surveillance contacts, subject presents symptoms of RTI, a nasal swab will be collected.
- **Study groups**: Throughout the three steps, infants will be randomized in two groups to receive either ChAd155-RSV vaccine or placebo.

Table 1 Study groups and epochs foreseen in the study

| Ston | Study | Number of | Ago (Min/Max) | Еро | chs |
|---|---|---|---|---|---|
| Step | groups | subjects* | Age (Min/Max) | Epoch 001 | Epoch 002 |
| 1 | RSV-Ld | ~ 16 | 12 months - 23 months | Х | Х |
| | Placebo-Ld | ~ 16 | 12 months - 23 months | Х | Х |
| 2 | RSV-Md | ~ 16 | 12 months - 23 months | Х | Х |
| | Placebo-Md | ~ 16 | 12 months - 23 months | Х | Х |
| 3 | RSV-Hd | ~ 16 | 12 months - 23 months | Х | Х |
| | Placebo-Hd | ~ 16 | 12 months - 23 months | X | Х |

**RSV-Ld**: low dose ChAd155-RSV vaccine (5 x 10<sup>9</sup> vp); **RSV-Md**: middle dose ChAd155-RSV vaccine (1.5 x 10<sup>10</sup> vp); **RSV-Hd**: high dose ChAd155-RSV vaccine (5 x 10<sup>10</sup> vp).

- \*The target will be to enroll up to 96 RSV-seropositive infants aged 12 to 23 months at the time of first vaccination (unless the dose escalation IDMC decision can be made based on the evaluation of accumulating safety data on fewer subjects) to ensure that at least 64 infants receive two doses of study vaccine (ChAd155-RSV or Placebo) (see Section ). Then the number of subjects at each step will be at least 16 (approximately 8 subjects per group) at steps 1 and 2 and 32 (approximately 16 subjects per group at step 3)
- Vaccination schedule: two IM vaccine doses administered according to a 0, 1-month schedule (i.e. at Day 1 and Day 31)
- **Treatment allocation**: infants will be randomized using a randomization system on internet (SBIR) at first vaccination
- **Blinding**: observer-blind in Epoch 001 and single-blind in Epoch 002

### • Sampling schedule:

Blood samples for biochemistry will be taken from all infants at Screening (up to 29) days before first vaccination to Day 1) and on Day 31, and Day 61 (refer to Table 11 of the protocol for the list of parameters to be tested). Blood samples for hematology will be taken from all infants at Screening (up to 29 days before first vaccination to Day 1) and on Day 1, Day 31, Day 32, and Day 61 (refer to Table 11 of the protocol for the list of parameters to be tested). Day 8 hematology testing will be performed if any  $\geq$  Grade 1 for platelet decrease is detected on Day 2 after vaccination, to ensure its resolution. Similarly, hematology testing on Day 38 will be performed if any  $\geq$ Grade 1 for platelet decrease is detected on Day 32. A clinical examination with special attention given to detection of spontaneous bleeding or easy bruising and evidence of bruising or petechiae will be performed by the investigator/study staff on Day 2, Day 4 and Day 8 after each vaccination (i.e. Day 2, Day 4, Day 8, Day 32, Day 34, and Day 38. The visits on Day 4 and Day 34 may be replaced by a phone call by the investigator/study staff to inquire of the infants' general health and to solicit reports of a rash, spontaneous bleeding or easy bruising. On Day 2, and Day 32, special attention will also be given to the detection of petechiae or evidence of petechiae induced by the tourniquet. This special attention to detection of petechiae or evidence of petechiae induced by the tourniquet will also be given on Day 8 and/or Day 38 in case hematology testing will be performed on that day. Further testing may be required to investigate a finding or guide subject management based on the investigators clinical judgment. Subjects' parent(s)/LAR(s) will be instructed to contact the investigator/study staff if their child presents symptoms of spontaneous bleeding or easy bruising or if their child develops a rash in the month following vaccination, in order to detect any thrombocytopenic petechiae or purpura. The

204838 (RSV PED-002) Statistical Analysis Plan Final

investigator will, based on his/her medical judgement, appropriately investigate infants with clinical suspicion of low platelets

- Blood sample for RSV serostatus will be taken from all infants at Screening.
- Blood samples for CMI are limited to those in investigational sites with a laboratory in proximity capable to perform WBS necessary for the CMI assay. In those sites, samples will be taken from all subjects at Screening and on Day 31, Day 61, and Day 366.
  - Note: Blood samples for CMI taken on Day 8 and Day 38 for subjects enrolled under protocol amendment 1 will still be assessed for CMI.
- Blood samples for humoral immunogenicity will be taken from all subjects at Screening and on Day 31, Day 61, and Day 366.
- Blood sample for assessment of mechanism of illness (potential ERD) will be taken from subjects hospitalized for LRTI (only for RSV-positive subjects using a locally available RSV test).
- Nasal swab: there will be monthly nasal swab to detect asymptomatic RSV infections during the RSV season and if following active or a passive surveillance contacts, a subject present symptom of RTI, a nasal swab will be collected.
- **Study visits**: Visit 1 (Day 1), Visit 5 (Day 31), Visit 9 (Day 61) and Visit 10 (Day 366) must be performed at the investigators clinical facility. Visit 2 (Day 2), Visit 4 (Day 8), Visit 6 (Day 32), Visit 8 (Day 38) and Visit 11 (Day 731) (no blood sampling for immune response and no vaccine administration) may take place in the subject's home or at the investigators clinical facility as appropriate to the circumstances in the judgment of the investigator. Visit 3 (Day 4) and Visit 7 (Day 34) may take place at the investigators clinical facility or the investigator/clinical staff may call the subjects' parent(s)/LAR(s), as appropriate to the circumstances in the judgment of the investigator.
- Surveillance for RSV-RTI, difficulty in breathing and wheezing episodes.
  - Surveillance period will be carried out from Visit 1 (after Dose 1) until Visit 11 (Day 731). In order to detect asymptomatic RSV-RTI, monthly nasal swabs for analysis at sponsor laboratory will be performed for all subjects during the RSV season. In order to timely detect RSV-RTI and to ensure cases are timely captured by the study sites, both active and passive surveillance will be conducted:
  - Passive surveillance: Parent(s)/LAR(s) are instructed to contact the investigator/study staff as soon as the subject experiences new RTI symptoms (cough, runny nose or blocked nose) or worsening of RTI symptoms, or in case of difficulty in breathing or wheezing.
  - Active surveillance: parent(s)/LAR(s) of all the subjects will be contacted by the investigator/study staff on a regular basis (weekly during the RSV season and every month outside the RSV season) to identify any potential RSV-RTI and to remind the parent(s)/LAR(s) of the subjects to report any new occurrence of RTI symptoms (cough, runny nose, blocked nose) or worsening of RTI symptoms, or in case of difficulty in breathing or wheezing as soon as possible.

## 3. OBJECTIVES

## 3.1. Primary objective

• To evaluate the safety and reactogenicity of three dose levels of the RSV investigational vaccine when administered as two IM doses according to a 0, 1-month schedule, up to 30 days after Dose 2 (i.e. Day 61) in RSV-seropositive infants aged 12 to 23 months

# 3.2. Secondary objectives

- To evaluate the safety of two IM doses of three dose levels of the RSV investigational vaccine when administered according to a 0, 1-month schedule from study start (Day 1) up to study conclusion (Day 731) in RSV-seropositive infants aged 12 to 23 months
- To evaluate the occurrence of RSV respiratory tract infections in RSV-seropositive infants from Visit 1 (Day 1, after Dose 1) up to study conclusion (Day 731)
- To evaluate the magnitude of the CMI induced by two IM doses of three dose levels of the RSV investigational vaccine when administered according to a 0, 1-month schedule, up to Day 366 in RSV-seropositive infants aged 12 to 23 months.
- To evaluate the humoral immunogenicity induced by two IM doses of three dose levels of the RSV investigational vaccine when administered according to a 0, 1-month schedule, up to Day 366 in RSV-seropositive infants aged 12 to 23 months

# 3.3. Tertiary objectives

- To further evaluate the CMI profile induced by two IM doses of three dose levels of the RSV investigational vaccine when administered according to a 0, 1-month schedule, up to Day 366 in RSV-seropositive infants aged 12 to 23 months
- If deemed necessary, to further characterize the immune response of the RSV investigational vaccine when two IM doses are administered according to a 0, 1-month schedule in RSV-seropositive infants.

### 4. ENDPOINTS

# 4.1. Primary endpoints

- Occurrence of AEs from first vaccination (Day 1) up to Day 61.
  - Occurrence of each solicited local and general AE, during a 7-day follow-up period after each vaccination (i.e. the day of vaccination and 6 subsequent days).
  - Occurrence of any unsolicited AE, during a 30-day follow-up period after each vaccination (i.e. the day of vaccination and 29 subsequent days).

- Occurrence of any SAE from Day 1 up to Day 61.
- Occurrence of episode of spontaneous or excessive bleeding (AE of specific interest), during a 30-day follow-up period after each vaccination.
- Occurrence of any hematological (hemoglobin level, white blood cells and platelets) laboratory abnormalities at Screening, Day 1, Day 8, Day 31, Day 32, Day 38, and Day 61.
- Occurrence of any biochemical (alanine aminotransferase, aspartate aminotransferase and creatinine) laboratory abnormalities at Screening, Day 31, and Day 61

## 4.2. Secondary endpoints

- Occurrence of SAEs from study start (Day 1) up to Day 366.
- Occurrence of RSV-LRTI (AE of specific interest) as from Dose 1 administration up to Day 366.
- Occurrence of RSV-RTI, RSV-LRTI, severe RSV-LRTI (according to standardized case definitions) as from Dose 1 administration up to Day 366.
- Occurrence of SAEs from study start (Day 1) up to study conclusion (Day 731).
- Occurrence of RSV-LRTI (AE of specific interest) as from Dose 1 administration up to study conclusion (Day 731).
- Occurrence of RSV-RTI, RSV-LRTI, severe RSV-LRTI (according to standardized case definitions) as from Dose 1 administration up to study conclusion (Day 731).
- Magnitude of the CMI response to the investigational RSV vaccine, pre-vaccination (Screening), post-Dose 1 (Day 31) and post-Dose 2 (Day 61 and Day 366).
  - CD3+/CD4+ T-cells expressing at least two markers among CD40L, IL-2, TNF-α, and IFN-γ upon stimulation with F, N and M2-1 peptide pools.
- Humoral response to the investigational RSV vaccine, pre-vaccination (Screening), post-Dose 1 (Day 31) and post-Dose 2 (Day 61 and Day 366):
  - Neutralizing antibody titers against RSV-A.
  - RSV F antibody concentrations.
- Humoral response to the investigational RSV vaccine, pre-vaccination (Screening), post-Dose 1 (Day 31) and post-Dose 2 (Day 61):
  - Palivizumab-competing antibody concentrations.

## 4.3. Tertiary endpoints

- CMI response profile (Th1, Th2, Th17) to the investigational RSV vaccine, prevaccination (Screening), post-Dose 1 (Day 31) and post-Dose 2 (Day 61 and Day 366).
  - CD3+/CD4+ and/or CD3+/CD8+ T-cells expressing at least one or any combination of immune marker(s) among CD40L, 41BB, IL-2, TNF-α, IFN-γ, IL-13 and IL-17 upon stimulation with F, N and M2-1 peptide pools.
- Any further exploratory immunology to detect disease-related or vaccine-related immune responses, such as but not limited to:
  - Anti-vector immunity: neutralization. (Analysis for this endpoint will be described in another SAP/AAR).

## 5. ANALYSIS SETS

### 5.1. Definition

### 5.1.1. Total vaccinated cohort

The total vaccinated cohort (TVC) will include all subjects with at least one study vaccine administration documented.

- A safety analysis based on the TVC will include all vaccinated subjects.
- An immunogenicity analysis based on the TVC will include all vaccinated subjects for whom immunogenicity data are available.

The TVC analysis will be performed per treatment actually administered at Dose 1.

# 5.1.2. According-to-protocol cohort for analysis of immunogenicity

The ATP cohort for analysis of immunogenicity will be defined by timepoint and will consist of all subjects from the TVC who complied with eligibility criteria, study procedures up to the end of the study and had immunogenicity results in the epoch as described below.

More specifically, the ATP cohort for analysis of immunogenicity up to Visit 9 (Day 61)/at Visit 10 (Day 366) will include all evaluable subjects:

- Who met all eligibility criteria (i.e. no protocol violation linked to the inclusion/exclusion criteria, including age).
- Who received two dose of study vaccine.
- For whom the administration route and site of the vaccine was as according to protocol.

204838 (RSV PED-002) Statistical Analysis Plan Final

- Who received the vaccine according to protocol procedures.
- Who complied with the vaccination schedule, as specified in Table 5 of the protocol.
- Who did not receive a concomitant medication/product leading to exclusion from an ATP analysis, as described in Section 7.6.2 of the protocol, up to Visit 9 (Day 61)/up to Visit 10 (Day 366).
- Who complied with the timings of the post vaccination blood sampling for immune response evaluation, up to Visit 9 (Day 61) /at Visit 10 (Day 366), as specified in Table 5 of the protocol.
- For whom post-vaccination immunogenicity results are available for at least one assay up to Visit 9 (Day 61) /at Visit 10 (Day 366).

Note that in order to align to ICH and cDISC terminology the Total Vaccinated Cohort and the According to Protocol cohort have been renamed Exposed Set (ES) and Per-Protocol Set (PPS) respectively.

# 5.2. Criteria for eliminating data from Analysis Sets

Elimination codes are used to identify subjects to be eliminated from analysis. Detail is provided below for each set.

### 5.2.1. Elimination from Exposed Set (ES)

Code 1030 (Study vaccine not administered at all) and code 900 (invalid informed consent or fraud data) will be used for identifying subjects eliminated from ES

## 5.2.2. Elimination from Per-protocol analysis Set (PPS)

### 5.2.2.1. Excluded subjects

A subject will be excluded from the PPS for analysis of immunogenicity at Day 61 and Day 366 under the following conditions

| Code | Condition under which the code is used |
|---|---|
| 900 | Invalid informed consent or fraud data (Subjects receiving a code 900 should |
| | not receive any other elimination codes) |
| 1030 | Study vaccine not administered at all (Subjects receiving a code 1030 should |
| | not receive any other elimination codes) |
| 1050 | Randomization failure |
| 1070\$ | Subjects got vaccinated with the correct vaccine but containing a lower volume |
| 1070\$ | Administration not according to protocol for reason specified by the |
| | investigator, other than side, site and route |
| 1070\$ | Site or route of study vaccine administration wrong or unknown |
| 1070\$ | Wrong replacement or study vaccine administered (not compatible with the |
| | vaccine regimen associated to the treatment number) |
| 1070\$ | Administered study vaccine reported as being the correct one but is not |
| | compatible with the vaccine regimen associated to the treatment number |
| 1080 | Vaccine temperature deviation |
| 1090 | Expired vaccine administered |
| 1500\$ | Subjects who have received only one dose of vaccination |
| 2010 | Protocol violation (inclusion/exclusion criteria) |
| 2080 | Subjects did not comply with vaccination schedule |
| | (DOSE 1 to DOSE $2 = 23-36$ (days) |

 $<sup>^{\$}</sup>$ Attribution of code to a subject requires CRDL confirmation Please note that all the elimcode has to be checked for the subject under schedule 1.

# 5.2.2.2. Right censored Data

Data from visit X and subsequent visit will be censored for the PPS analysis under the following conditions. The code \*\*\*\*.Vx will be used to identify subjects whose immunogenicity data should be eliminated from a specific visit onwards. Vx will be V9 and V10 with respect to PPS defined up to Visit 9 and Visit 10, respectively.

| Code | Decode → Condition under which the code is used |
|---|---|
| 1040*.Vx | Administration of concomitant vaccine(s) forbidden in the protocol → A vaccine not foreseen by the study protocol administered from dose 1 and ending 30 days after the last dose of vaccines administration • Applicable visits — For Day 61 PP, to check from Dose 1 up to Day 61 |
| | <ul> <li>For Day 366 PP, to check from Dose 1 up to Day 366</li> </ul> |
| 1060 | Randomization code was broken |

<sup>\*</sup> Attribution of these elimcodes are responsibility of CRDL following review of individual data listings
Please note that all the elimcode has to be checked for the subject under schedule 1 who have received vaccination.

# 5.2.2.3. Visit-specific censored Data

Data at visit X will be censored for the PPS analysis under the following conditions. The code \*\*\*\*.Vx will also be used to identify study withdrawal at visit X. Vx will be V9 and V10 with respect to PPS defined up to Visit 9 and Visit 10, respectively.

| Code | Decode → Condition under which the code is used |
|---|---|
| 2040*.Vx | • Administration of any medication forbidden by the protocol→ |
| | <ul> <li>Any investigational or non-registered product (drug or vaccine)<br/>other than the study vaccines used during the study period.</li> </ul> |
| | <ul> <li>Immunosuppressants or other immune-modifying drugs<br/>administered chronically (i.e., more than 14 days) during the study<br/>period.</li> </ul> |
| | <ul> <li>Immunoglobulins and/or any blood products administered during the study period</li> </ul> |
| | <ul> <li>Administration of long-acting immune-modifying drugs during the<br/>study period.</li> </ul> |
| | Applicable visits |
| | <ul> <li>For Day 61 PP (V9), check from Dose 1 up to Day 61 BS</li> </ul> |
| | <ul> <li>For Day 366 PP (V10), check from Dose 1 up to Day 366 BS</li> </ul> |
| 2050*.Vx | Underlying medical condition forbidden by the protocol |
| | Applicable visits |
| | <ul> <li>For Day 61 PP, to check from Dose 1 up to Day 61</li> </ul> |
| | <ul> <li>For Day 366 PP, to check from Dose 1 up to Day 366</li> </ul> |
| 2060*.Vx | Concomitant infection related to the vaccine which may influence immune response |
| | Applicable visits |
| | <ul> <li>For Day 61 PP (V9), to check from Dose 1 up to Day 61</li> </ul> |
| | <ul> <li>For Day 366 PP (V10), to check from Dose 1 up to Day 366</li> </ul> |
| 2070*.Vx | Concomitant infection not related to the vaccine which may influence immune response |
| | Applicable visits |
| | <ul> <li>For Day 61 PP, to check from Dose 1 up to Day 61</li> </ul> |
| | <ul> <li>For Day 366 PP, to check from Dose 1 up to Day 366</li> </ul> |
| 2090.Vx | Subjects did not comply with immunological blood sample schedule |
| | Applicable visits |
| | <ul> <li>For Day 61 PP, to check for Dose 1 to Visit 5 BS = 23-36 days and Dose 2 to Visit 9 BS = 28-35 days]</li> </ul> |
| | <ul> <li>For Day 366 PP, to check for Dose 1 to Visit 10 BS = 335-395 days]</li> </ul> |

| Code | Decode → Condition under which the code is used |
|---|---|
| 2100.Vx | Serological results not available post-vaccination→ No immunological result at all for the specific blood sample collection timepoint |
| | Applicable visits |
| | <ul> <li>For Day 61 PP, check for availability of atleast one assay [CMI (ICS), Neutra, RSV F IgG or PCA result] at Day 31 and Day 61</li> </ul> |
| | <ul> <li>For Day 366 PP, check for availability of atleast one assay [CMI (ICS), Neutra, RSV F IgG or PCA result] at Day 366</li> </ul> |
| 2120 <sup>!@</sup> .Vx | Obvious incoherence or abnormality or error in data → Incoherence between CRF and results, wrong sample labelling, Central/internal/external lab deviations; incorrect spinning/processing of sample including processing within the time required by protocol; temperature deviations from range defined in protocol and/or SPM - room temperature/refrigerator/freezer; an assessment was completed, but was not completed according to protocol or SPM. |
| | Applicable visits |
| | <ul> <li>For Day 61 PP, check on Day 31 and Day 61 CMI (ICS), Neutra,<br/>RSV F IgG or PCA result</li> </ul> |
| | <ul> <li>For Day 366 PP, check on Day 366 CMI (ICS), Neutra, RSV F IgG<br/>or PCA result</li> </ul> |

<sup>\*</sup> Attribution of these elimcodes are responsibility of CRDL following review of individual data listings
Please note that all the elimcode has to be checked for the subject under schedule 1 who is vaccinated.

@this code need confirmation from lab expert of particular test performed
! Attribution of code to a subject requires CRDL confirmation

# 5.3. Important protocol deviation not leading to elimination from per-protocol analysis set

The following important protocol deviations will be reported by groups:

- Forced randomization: In case of supplies shortage for the next assigned vaccine according to the randomization schedule at the clinical site, the randomization system will use the forced randomization procedure in order to continue to enrol and vaccinate subjects. The system moves seamlessly to the next treatment/randomization number for which vaccine supplies are available. The site will not be aware of the forced randomization event.
- Short follow-up: subjects who completed the last study contact before the minimum length of follow-up requirement
- In case unexpected vaccinations at study start were granted due to regulatory recommendation or medical need, the subjects who had such vaccination could be mentioned.

### 6. STATISTICAL ANALYSES

Note that standard data derivation rule and stat methods are described in annex 1 and will not be repeated below.

## 6.1. Demography

# 6.1.1. Analysis of demographics/baseline characteristics planned in the protocol

The analysis of demographics will be performed on the Exposed Set and on the PPS for analysis of immunogenicity at Day 61 and Day 366 analysis. The analysis of demography will be performed on Exposed Set at Day 731.

Demographic characteristics (age at first vaccination in months, gender, race, country), weight, height or length, and vital signs, and cohort description will be summarized by group using descriptive statistics:

- Frequency tables will be generated for categorical variable such as race.
- Mean, median, standard error and range will be provided for continuous data such as age.

The above analysis will also be done at Day 366 and Day 731 with age at the visit in months.

The weight for age Z score (WAZ) and height or length for age Z score (HAZ) at first vaccination, Day 366 and Day 731 will be calculated on ES. The distribution of subjects will be tabulated as a whole and per group.

Withdrawal status will be summarized by group using descriptive statistics.

- The numbers of withdrawn subjects will be tabulated according to the reason for withdrawal on ES
- The number of subjects enrolled into the study as well as the number of subjects excluded from PPS analyses will be tabulated.

## 6.2. Immunogenicity

# 6.2.1. Analysis of immunogenicity planned in the protocol

The primary analysis will be performed on the PPS for analysis of immunogenicity and a complementary analysis will be performed on Exposed Set. All the immune analysis is within group only.

### **6.2.1.1. CMI** analysis

The analysis will be performed on each group separately, pooled placebo group and pooled RSV group. All the CMI analysis will be performed for each peptide pool (F, N, M2-1) separately and taking all the peptide pool together for subjects who has data available for the three peptide pools.

With respect to secondary objectives, the following parameters will be summarized by group using descriptive statistics (N, geometric mean [GM], minimum [min], 1st quartile [Q1], median, third quartile [Q3], maximum [max]), at each timepoint during which blood samples are collected for CMI in investigational sites with a laboratory in proximity capable to perform WBS necessary for the CMI assay:

- Frequency of CD4+ T-cells expressing at least two markers among CD40L, IL-2, TNF- $\alpha$ , and IFN- $\gamma$  upon stimulation with F, N and M2-1.
- Box plot with individual data for CD4+ T-cells expressing at least two markers among CD40L, IL-2, TNF-α, and IFN-γ upon stimulation with F, N and M2-1 and combined peptide pool will be presented.

With respect to tertiary objectives, the cellular immune response will be further characterized using descriptive analysis of the frequency of CD8+ T-cells and CD4+ T-helper cell profile (Th1, Th2, Th17) expressing at least one or any combination of marker(s) among CD40L, 41BB, IL-2, TNF-α, IFN-γ, IL-13, and IL-17.

The following parameters will be summarized by group using description statistics (N, GM, min, Q1, median, Q3, max), at each timepoint during which blood samples are collected for CMI:

- Frequency of CD4+ and CD8+ T-cells expressing at least one or any combination of immune marker(s) among CD40L, 41BB, IL-2, TNF-α, IFN-γ, IL-13 and IL-17 upon stimulation with F, N and M2-1 peptide pools.
- Tabular presentation of T-helper cell 'Th1' profile Frequency of CD4+ T-cells expressing at least IFN-γ but no IL-13 upon stimulation with F, N and M2-1 peptide pools.
- Tabular presentation of T-helper cell 'Th2' profile: Frequency of CD4+ T-cells expressing at least IL-13 but no IFN-γ upon stimulation with F, N and M2-1 peptide pools.
- Tabular presentation of T-helper cell 'Th17' profile Frequency of CD4+ T-cell expressing atleast IL17 upon stimulation with F, N and M2-1 peptide pools.
- Calculation of 'Th2/Th1 ratio' = Frequency of Th2 T-cells / frequency of Th1 T-cells.
- Separate box plot with individual data for CD4+ and CD8+ T-cells expressing at least one marker among CD40L, 41BB, IL-2, TNF-α, IFN-γ, IL-13 and IL-17 upon stimulation with F, N and M2-1 and combined peptide pools will be presented.

204838 (RSV PED-002) Statistical Analysis Plan Final

- Separate box plot with individual data for CD4+ T-cells expressing at least IFN-γ but no IL-13 (Th1 profile) upon stimulation with F, N and M2-1 and combined peptide pools will be presented.
- Separate box plot with individual data for CD4+ T-cells expressing at least IL-13 but no IFN-γ (Th2 profile) upon stimulation with F, N and M2-1 and combined peptide pools will be presented.
- Separate box plot with individual data for CD4+ T-cells expressing at least IL17(Th17 profile) upon stimulation with F, N and M2-1 and combined peptide pools will be presented.

The need to generate co-expression profile graph for any combination for CD4+ and CD8+ will be evaluated after looking at the descriptive tables.

### 6.2.1.2. Humoral immune response

For each group, at each timepoint that blood samples are collected for humoral immune response against the investigational RSV vaccine (neutralizing antibody titers against RSV-A, RSV F antibody concentrations, and palivizumab-competing antibody concentrations):

- GMTs/GMCs will be tabulated with 95% CI and represented graphically.
- Percentage of subjects above the seropositivity threshold will be tabulated with exact 95% CI.
- Antibody titers/concentrations will be displayed using reverse cumulative curves.
- The distributions of neutralizing antibody titers/concentrations will be tabulated (< 128, 128-256, > 256-512, > 512-1024, > 1024-2048, > 2048-4096, > 4096)
- Percentage of responders in terms of RSV-A neutralizing antibody titers will be tabulated with exact 95% CI.
- Individual post-vaccination versus pre-vaccination results will be plotted using scatter plots. Results of the Placebo groups will be used as a reference.
- Geometric mean of ratios of antibody titers/concentrations at each post-vaccination timepoint over pre-vaccination will be tabulated with 95% CI.
- Distribution of the fold increase of the neutralizing antibody titers will be tabulated by pre-vaccination titer category (percentage of subjects with a fold increase equal to or above 1, 2, 2.5, 3, 4, 6, 8 10, 11 and 12 by pre-vaccination titre category: (< 128, 128-256, > 256-512, > 512-1024, > 1024-2048, > 2048-4096, > 4096, and by cumulative category:  $<128, \ge 128, \ge 256, \ge 512, \ge 1024, \ge 2048, \ge 4096.$ ).
- The kinetics of individual antibody titer/antibody concentration results will be plotted as a function of time for subjects with results available at all timepoints.

If available, any further exploratory immunology results (including, but not limited to anti-vector immunity) will be reported by group and timepoint using descriptive summary statistics will be described separately in Additional analysis request (AAR).

## 6.3. Analysis of RSV incidence

The assessment of RSV analysis incidence and severity will be performed on the Exposed Set on RSV groups, placebo groups, pooled RSV and pooled Placebo groups separately for first RSV season (Day 1-366) and second RSV season (Days 367-731) and overall (Days 1-731).

The analysis will be performed according to all case definitions presented in Table 5.

The proportion of subjects with at least one RSV infection and number of infections experienced by subjects meeting each of the case definition in Table 5 (with 95 % CI) will be calculated by group.

The number of RSV infections within each group and the maximum disease severity of the event will be tabulated. The number of RSV infections within each group and frequency of hospitalization will be tabulated. The number of infections in each group and descriptive analysis of the viral load associated with the maximum disease severity of the event will be tabulated (mean, median, min, max). Descriptive analysis on maximum viral load per subject based on qRT-PCR confirmed RSV infection of maximum severity will be performed.

The viruses identified in the Respiratory Viral Panel will be tabulated to those events where RSV-RTI was identified to describe frequency of co-infections and responsible viruses. These tables will be repeated limited to RVP results of cases of confirmed LRTI and RSV-LRTI.

After looking at the frequency of coinfection of all confirmed LRTI and RSV-LRTI, if there will be more than 10% coinfections (RSV infection with identification of another viral pathogen on RVP), tables will be reproduced including those RSV episodes where co-infection was present and those where no other respiratory viral pathogen was identified. The descriptive analysis on viral load table will not be repeated on subject with at least one episode with maximum viral load.

Listing will be presented for all cases of RSV infection until Day 731 with the details of gender, age at episode, country, site, day of event (i.e days since first visit), classification according to maximum severity of episode as RSV RTI/RSV LRTI/ RSV severe LRTI and RSV very severe LRTI, RSV hospitalization 'Yes/No', SpO2 value, respiratory rate, result of RSV qRT-PCR and RVP result will be presented.

Listings will be generated at Day 731 for all hospitalized cases with gender, age at episode, classification according to maximum severity of episode as (RSV RTI/RSV LRTI/ RSV severe LRTI and RSV very severe LRTI), RVP result, total number of calendar days on which the child was hospitalized, days requiring monitoring/nursing observation, days requiring nasogastric or intravenous fluids, days requiring supplemental oxygen, days requiring respiratory support excluding mechanical ventilation, days requiring mechanical ventilation and days requiring pediatric intensive care unit management.

## 6.4. Analysis of safety

## 6.4.1. Analysis of safety planned in the protocol

### 6.4.1.1. Within groups assessment

The analysis will be based on the ES on each treatment groups separately.

The percentage of subjects with at least one local AE (solicited and unsolicited), with at least one general AE (solicited and unsolicited) and with any AE during the 7-day or 30-day follow-up period will be tabulated with exact 95% confidence interval (CI) after each vaccine dose and overall. The percentage of doses followed by at least one local AE (solicited and unsolicited), by at least one general AE (solicited and unsolicited) and by any AE during the 7-day or 30-day follow-up period will be tabulated, overall vaccination course, with exact 95% CI. The same computations will be done for Grade 3 AEs, for any AEs considered related to vaccination and for any Grade 3 AEs considered related to vaccination.

The percentage of subjects reporting each individual solicited local AE (any grade, Grade 2, Grade 3, resulting in a medically attended visit) and solicited general AE (any grade, Grade 2, Grade 3, any related, Grade 2 related, Grade 3 related, resulting in medically attended visit) during the 7-day follow-up period (Day 1-7) will be tabulated for each group after each vaccine dose and overall. Similarly, the percentage of doses followed by each individual solicited local and general AE and their sub-categories, will be tabulated, overall vaccination course, with exact 95% CI.

For fever, the number and percentage of subjects reporting fever by half degree (°C) cumulative increments during the 7-day follow-up period (Day 0-6) will be tabulated for each group after each vaccine dose and overall. Similar tabulations will be performed for any fever with a causal relationship to vaccination, Grade 3 (> 39.5°C) causally related fever and for any fever resulting in a medically attended visit. In addition, the prevalence of any and Grade 3 fever will be presented graphically over time after vaccination.

The percentage of subjects with unsolicited AEs within 30 days (Day 1-30) after each vaccine dose (overall doses) with its exact 95% CI will be tabulated by group and by MedDRA preferred term. Similar tabulation will be done for Grade 3 unsolicited AEs, for any causally related unsolicited AEs, for Grade 3 causally related unsolicited AEs and for unsolicited AEs resulting in a medically attended visit. The verbatim reports of unsolicited AEs will be reviewed by a physician and the signs and AEs will be coded according to the MedDRA Dictionary Version 20 for Adverse Reaction Terminology. Every verbatim term will be matched with the appropriate Preferred Term.

The percentage of subject with episode of spontaneous or excessive bleeding (AE of specific interest), during a 30-day follow-up period after each vaccination will be tabulated by group according to associated PT code presented in Section 12. The percentage of subjects with RSV-LRTI (AE of specific interest) from Dose 1 up to Day 365 and from Dose 1 up to study conclusion (Day 730) will be tabulated by group according to associated PT code presented in Section 12.

204838 (RSV PED-002) Statistical Analysis Plan Final

The percentage of subjects with SAE within 30 days (Day 1-30) after each vaccine dose with its exact 95% CI will be tabulated by group and by MedDRA preferred term. Similar table will be generated for SAE from Dose 1 up to Day 61, from Dose 1 up to Day 366 and from Dose 1 up to Day 731.

SAEs reported throughout the study and AE of specific interest will be described in detail.

The percentage of subjects using concomitant medication (any medication, any antipyretic/ analgesic and any antipyretic taken prophylactically, respectively) during the 7-day follow-up period (Day 1-7) and during the 30-day follow-up period (Day 1-30) will be summarized by group after each vaccine dose and overall.

For each group and for each hematology and biochemistry parameter:

- The percentage of subjects having hematology and biochemistry results below/above/within the local laboratory normal ranges will be tabulated by timepoint and toxicity grading scale.
- The maximum grading from Screening up to Visit 9 (Day 61) will be tabulated by grading the safety laboratory values according to toxicity criteria Grading scale adapted from [Division of AIDS, 2003], [Division of AIDS, 2004] and [Division of AIDS, 2007].
- For eosinophils, basophils, and monocytes, summary statistics (min, max, standard deviation, mean and median) will be presented as there is no grading provided for these parameters.

### 6.4.1.2. Between groups assessment

Exploratory comparisons between the investigational RSV groups and the Placebo groups will be done in terms of the percentage of subjects, overall doses, reporting any Grade 2/3 AE during the 7-day follow-up period (Day 1-7) after vaccination, and/ or any fever >38.5°C during the 7-day follow-up period (Day 1-7) after vaccination, and/ or any vaccine-related SAE during the 7-day follow-up period (Day 1-7) after vaccination.

The standardized asymptotic 95% CI for the following differences will be computed:

- RSV Ld minus Placebo Ld
- RSV Md minus Placebo Md
- RSV Hd minus Placebo Hd

### 6.4.2. Additional considerations

### 6.4.2.1. Additional safety analysis

For the analysis of safety, the percentage of subjects reporting each individual solicited local AE (any, each grade, resulting in medically attended visit) during the 7-day follow-up period after vaccination will be tabulated based on maximum intensity per subject for each study vaccine for each group. The percentage of subjects reporting each individual solicited general AE (any, each grade, any related, any Grade 2 related, any Grade 3 related, resulting in medically attended visit) during the 7-day follow-up period after vaccination will be based on maximum intensity per subject for each study vaccine for each group.

### 6.4.2.2. Exclusion of implausible solicited Adverse Event

Some local and systemic adverse events will be directly measured by the subject and will not be subject to a reconciliation process, even if they are biologically implausible. Therefore, these implausible measurements will be removed from the analysis but included in listings. Implausible measurements are summarized in the table below:

Table 2 Implausible Solicited Adverse Events

| Parameter | Implausible measurements |
|------------------|---------------------------------------------|
| Body temperature | ≤ 33°C or ≥ 42°C |
| Swelling | For subjects < 6 years: Measurements < 0 mm |

### 6.4.2.3. Combined Solicited and Unsolicited Adverse Events

A summary of subjects with all combined solicited (regardless of their duration) and unsolicited adverse events will be provided. Solicited adverse events will be coded by MedDRA as per the following codes

| Solicited symptom | Lower level term name | Lower level term code | Corresponding Primary Term code |
|---|---|---|---|
| Pain | Pain | 10033371 | 10033371 |
| Redness | Erythema | 10015150 | 10015150 |
| Swelling | Swelling | 10042674 | 10042674 |
| Drowsiness | Drowsiness | 10013649 | 10013649 |
| Fever | Fever | 10016558 | 10016558 |
| Irritability/Fussiness | Irritability | 10022998 | 10022998 |
| Loss of appetite | Appetite lost | 10003028 | 10003028 |

For clintrial.gov and EudraCT posting purposes, a summary of combined solicited and unsolicited non-serious adverse events will be produced by System Organ Class and preferred terms and according to occurrence of each event.

## 7. ANALYSIS INTERPRETATION

All analyses are descriptive. Comparative analyses will be descriptive with the aim to characterize the difference in safety/reactogenicity between groups and should be interpreted with caution considering that there is no adjustment for multiplicity and that group sizes are small for these comparisons.

## 8. CONDUCT OF ANALYSES

## 8.1. Sequence of analyses

The statistical analyses will be performed in 3 steps:

A first analysis will be performed when all data (safety and immunogenicity) up to Day 61 (i.e. data that are as clean as possible) are available. Additional safety data available at the time of this analysis will be described. At this point, the statistician will be unblinded (i.e. individual subject treatment assignments will be available) and the study will be conducted in a single-blind manner, with patients remaining blinded up to study end (Day 731). Summary results may unblind some specific subjects but no individual listings will be provided and the investigators will not have access to the treatment allocation up to study end (Day 731), except in case of emergency unblinding (see Section 9.8 of the protocol).

An analysis will be performed when all data (safety and immunogenicity) up to Visit 10 (Day 366; i.e. data that are as clean as possible) are available. No individual listings will be provided.

The final analysis will be performed when all data up to study conclusion (Day 731) are available. An integrated clinical study report containing all data will be written and made available to the investigators at that time.

If the data for tertiary endpoints (additional exploratory analyses) become available at a later stage, (an) additional analysis/ analyses will be performed. These data will be documented in amendments to the study report and will be made available to the investigators at that time.

| Description | Analysis ID | Disclosure Purpose (CTRS=public posting, SR=study report, internal) | Dry run<br>review<br>needed<br>(Y/N) | Study Headline Summary<br>(SHS)requiring expedited<br>communication to upper<br>management (Yes/No) | Reference for TFL |
|---|---|---|---|---|---|
| Final Analysis | E1_01 | SR | N | Yes | |
| Analysis of epoch 1 | E1_0X | CTRS | Y | Yes | |
| Up to D366 | E1_0X+1 | | N | No | All tables from TFL dated xxxxxx |

Table 3 Endpoints assessed at different analysis time points

| Analysis | Analysis ID | Safety | Immuno | RSV/RTI |
|---|---|---|---|---|
| Epoch 1<br>(Day 60) | | Solicited AE, Unsolicited AE, haematology and biochemistry, AESI(bleeding), SAE from D1-Day 61 | All CMI and Humoral readout from D1-D61 | |
| Up to D366 | | SAE, AESI – | All CMI and Humoral | RSV analysis for 1st season |
| | | D1-D366 | response at D366 | – D1-D366 |
| Final (Day | | SAE, AESI – | None | RSV 2 <sup>nd</sup> season – D367- |
| 731) | | D1-D731 | | D731; Overall (D1-D731) |

## 8.2. Statistical considerations for interim analyses

No interim analysis is planned.

### 9. CHANGES FROM PLANNED ANALYSES

Following are the changes in the planned analysis:-

- The naming of the cohort has been changed per cDISC standards.
- Per cDISC standard, the day of first vaccination is now changed from Day 0 to Day 1.
- The study design diagram has been adapted as per cDISC format
- In secondary endpoints, specific safety endpoints for Day 1 up to D366 has been added as follows: -
  - Occurrence of SAEs from study start (Day 1) up to Day 366.
  - Occurrence of RSV-LRTI (AE of specific interest) as from Dose 1 administration up to Day 366.
  - Occurrence of RSV-RTI, RSV-LRTI, severe RSV-LRTI (according to standardized case definitions) as from Dose 1 administration up to Day 366.
- For the immunogenicity analysis, the analysis will be performed on both PPS and ES without any condition on percentage of subjects excluded
- For inclusion of subjects in PPS for analysis of immunogenicity, subjects should have received both the doses and not atleast one dose.

# 10. LIST OF FINAL REPORT TABLES, LISTINGS AND FIGURES

The TFL TOC provides the list of tables/listings and figures needed for the study report. It also identifies the tables eligible for each analyses and their role (synopsis, in-text, post-text, SHS, CTRS,...). Note that all TFL aimed to be included as post-text are noted as post-text even if these are tabulation of individual data such as listing of SAE. The post-text material contains all source material for the study report and accordingly a post-text table may be redundant with an in-text table.

The mock tables referred under column named 'layout' can be found in legacy-GSK SDD dedicated folder for standard tables and in Section 12 (Annex 2) for study specific mock table/figure/listing. The latter table/figure/listing are identified by the prefix SS\_ in the TFL Toc.

The following group names and pooled group names will be used in the TFLs, to be in line with the T-domains:

| Group<br>order in<br>tables | Group label in tables | Group definition for footnote | Pooled<br>Groups<br>label in<br>tables | Pooled definition for footnote |
|---|---|---|---|---|
| 1 | RSV-Ld | Low dose ChAd155-RSV vaccine (5 x 109 vp) | RSV | ChAd155-RSV vaccine (low/ middle/high dose pooled groups) |
| 2 | RSV-Md | Middle dose ChAd155-RSV vaccine (1.5 x 1010 vp) | RSV | ChAd155-RSV vaccine (low/ middle/high dose pooled groups) |
| 3 | RSV-Hd | High dose ChAd155-RSV vaccine (5 x 10 <sup>10</sup> vp) | RSV | ChAd155-RSV vaccine (low/ middle/high dose pooled groups) |
| 4 | Placebo-Ld | Non-active control (0.5 ml) | Placebo | Non active control (0.15/0.5 ml pooled groups) |
| 5 | Placebo-Md | Non-active control (0.15 ml) | Placebo | Non active control (0.15/0.5 ml pooled groups) |
| 6 | Placebo-Hd | Non-active control (0.5 ml) | Placebo | Non active control (0.15/0.5 ml pooled groups) |
| 7^ | Pooled | Pooled RSV + Placebo | Pooled | Pooled RSV + Placebo |

<sup>&</sup>lt;sup>^</sup>The pooled group is not in the treatment dataset but will be created for generating some tables during D366 analysis.

# 11. ANNEX 1 STANDARD DATA DERIVATION RULE AND STATISTICAL METHODS

# 11.1. cDISC specification

The analysis planned at D61, D366 and D731 is planned in cDISC format. In cDISC format, the day of vaccination is mentioned as Day 1 rather than Day 0 per protocol. Accordingly, all the timepoint will be mentioned as Day X +1. The analysis will be performed adjusting for it so that correct interval will be selected.

## 11.2. Statistical Method References

The exact two-sided 95% CIs for a proportion within a group will be the Clopper-Pearson exact CI [Clopper CJ, Pearson ES. The use of confidence or fiducial limits illustrated in the case of binomial. *Biometrika*. 1934; 26:404-413].

The standardised asymptotic two-sided 95% CI for the group difference in proportions is based on the method described in the following paper: Robert G. Newcombe, interval estimation for the difference between independent proportions: comparison of eleven methods, *Statist Med.* 1998; 17, 873-890]. The standardised asymptotic method used is the method six.

### 11.3. Standard data derivation

### 11.3.1. Date derivation

- SAS date derived from a character date: In case day is missing, 15 is used. In case day & month are missing, 30June is used.
- Onset day for an event (ae, medication, vaccination, ...): The onset day is the number of days between the last study vaccination & the onset/start date of the event. This is 1 for an event starting on the same day as a vaccination. See SAS date derived in case the start date of the event is incomplete.
- Duration: Duration of an event is expressed in days. It is the number of days between the start & the stop dates + 1. Therefore, duration is 1 day for an event starting & ending on the same day.
- Association of an event to the primary epoch: An adverse event belongs to the primary epoch, if the onset date is before and including Visit 9 (Day 60). Any safety data collected beyond Visit 9 (Day 60) will be collected in Epoch 002.

### 11.3.2. Dose number

- The study dose number is defined in reference to the number of study visits at which vaccination occurred. More specifically dose 1 refers to all vaccines administered at the first vaccination visit while dose 2 corresponds to all vaccinations administered at the second vaccination visit even if this is the first time a product is administered to the subject.
- Relative dose: the relative dose for an event (AE, medication, vaccination) is the most recent study dose given before an event. In case the event takes place on the day a study dose is given, the related dose will be that of the study dose, even if the event actually took place before vaccination. For instance, if an adverse event begins on the day of the study vaccination but prior to administration of the vaccine, it will be assigned to this dose. In case a study dose is not administered and an event occurs after the subsequent study dose (eg 2<sup>nd</sup> study dose), the relative dose of the event will be study dose associated to the subsequent study dose (eg dose 2).
- The number of doses for a product is the number of times the product was administered to a subject.
- The incidence per dose is the number of vaccination visits at which an event was reported among all vaccination visits.

## 11.3.3. Demography

- Age: Age at the reference activity, computed as the number of units between the date of birth and the reference activity. Note that due to incomplete date, the derived age may be incorrect by 1 month when month is missing from the birthdate. This may lead to apparent inconsistency between the derived age and the eligibility criteria/the age category used for randomization.
- Conversion of weight to kg: The following conversion rule is used:

Weight in Kilogramm= weight in Pounds / 2.2

Weight in Kilogramm = weight in oncs / 35.27

The result is rounded to 2 decimals.

• Conversion of height to cm: The following conversion rule is used:

Height in Centimetres = Height in Feet \* 30.48

Height in Centimetres = Height in Inch \* 2.54

The result is rounded to the unit (ie no decimal).

• Conversion of temperature to °C: The following conversion rule is used:

Temperature in °Celsius = ((Temperature in °Fahrenheit -32) \*5)/9

The result is rounded to 1 decimal.

- Calculation of weight for age Z-score (WAZ) for each subject (rounded to 2 decimal):
  - WAZ = (Weight of subject -median weight)/Standard deviation for weight
- Calculation of height for age Z-score (HAZ) for each subject (rounded to 2 decimal):
  - HAZ = (Height of subject -median height)/Standard deviation for height

## 11.3.4. Immunogenicity

- For a given subject and given immunogenicity measurement, missing or non-evaluable measurements will not be replaced. Therefore, an analysis will exclude subjects with missing or non-evaluable measurements. Kinetics will be plotted on subjects with results available at all timepoints.
- The Geometric Mean Concentrations/Titres (GMC/Ts) calculations are performed by taking the anti-log of the mean of the log titre transformations. Antibody titres below the cut-off of the assay will be given an arbitrary value of half the cut-off of the assay for the purpose of GMT calculation.
- The 95% CI for the mean of log-transformed titer will be first obtained assuming that log-transformed values were normally distributed with unknown variance. The 95% CI for the GMTs/GMCs will be then obtained by exponential-transformation of the 95% CI for the mean of log-transformed titer.
- A seronegative subject is a subject whose antibody titre is below the cut-off value of the assay. A seropositive subject is a subject whose antibody titre is greater than or equal to the cut-off value of the assay.
- An exploratory definition of vaccine response to the RSV neutralising antibodies will be as:
  - At least a 4-fold increase from pre-vaccination if pre-vaccination neutralising antibody titre <128.</li>
  - At least a 3-fold increase from pre-vaccination if pre-vaccination neutralising antibody titre in [128-256].
  - At least a 2.5-fold increase from pre-vaccination if pre-vaccination neutralising antibody titre in [256-1024].
  - At least 1-fold from pre-vaccination if pre-vaccination neutralising antibody titre >1024

Please note that other definition of vaccine response will be also be explored but interest might be limited considering this is not target population.

• Assay cut-off for the humoral immunity will be per the following table

| Component | Method | Unit | Cut-off |
|---|---|---|---|
| Respiratory Syncytial Virus A Ab | NEUTRALIZATION | ED60 | 8 |
| Respiratory Syncytial Virus F protein Ab.lgG (Anti-RSV PreF antibody) | ELISA | EU/ml | 10 |
| Respiratory Syncytial Virus F protein Ab.lgG (Palivizumab competing Ab) | ELISA | μg/ml | 9.6 |

• Considering the cut-off for the neutralising antibody against RSV-A is below the assay's LLOQ [32], the following rules will be applied for derivation of seropostivity status and GMT:

| Assay | Raw result | Derivation for<br>seropositivity<br>status | Derivation for<br>GMT<br>calculation | Derivation for fold-<br>increase between Post and<br>Pre-vaccination titres |
|---|---|---|---|---|
| RSV-A | <cut-off< td=""><td>NEG</td><td>Cut-off/2</td><td>LLOQ/2</td></cut-off<> | NEG | Cut-off/2 | LLOQ/2 |
| neutralising<br>Antibody | [cut-off-LLOQ [ | POS | Cut-Off | LLOQ/2 |
| Aillibody | ≥LLOQ | POS | Exact value | Exact value |

- The cut-off for the PCA assay is set at the level of the assay LLOQ (9.60 μg/mL). For results below the cut-off (LLOQ), an arbitrary value of half of the cut-off will be considered for calculation of GMC and fold increase.
- All CI computed will be two-sided 95% CI.
- CMI: CD4+ and/or CD8+ T-cells, by ICS using WBS
  - All results available in the database (events/per million of cells) will be dividing by 10000 in order to express the results in percentage (%).
  - The derived variable that will be used for the analysis will be:
    - the frequency of RSV F/N/M2-1 specific and combined (RSV F/N/M2-1) CD4+ T-cells expressing at least two marker among CD40L, IL-2, TNF-α, and IFN-γ;
    - the frequency of CD4<sup>+</sup> and CD8<sup>+</sup> T-cells expressing at least one or any combination of immune marker(s) among CD40L, 41BB, IL-2, TNF-α, IFN-γ, IL-13 and IL-17 upon stimulation with F, N and M2-1 peptide pools and combined peptide pools.
  - Those derived variables will be obtained as follows: sum of all specific responses of interest minus the sum of corresponding background responses. All values less or equal to zero will be set to 1 for the purpose of GM calculation.
  - Co-expression profile: for each CD4+/CD8+ any combination of markers, the RSV F/N/M2-1 specific response will be obtained by subtracting the background value to the RSV value (stimulation with RSV F/N/M2-1 peptides), and by setting to 1 all values less than or equal to zero for the purpose of GM calculation and graphical representation.
  - The log-transformation of the percentage of RSV F/N/M2-1specific CD4+/CD8+ T-cells will be applied, and the GM calculations will be performed by taking the anti-log of the mean of the log transformations.
  - For calculation of Th2/Th1 ratio has to be done by taking average of Th2 and Th1 profile at the individual level after adjusting on background.
#### 11.3.5. Safety

- For a given subject and the analysis of solicited symptoms during the 7 day follow-up period after vaccination, missing or non-evaluable measurements will not be replaced. Therefore, the analysis of the solicited symptoms based on the ES will include only vaccinated subjects with documented safety data (*i.e.*, symptom screen completed). More specifically the following rules will be used:
  - Subjects who documented the absence of a solicited symptom after one dose will be considered not having that symptom after that dose.
    - Subjects who documented the presence of a solicited symptom and fully or partially recorded daily measurement over the solicited period will be included in the summaries at that dose and classified according to their maximum observed daily recording over the solicited period.
    - Subjects who documented the presence of a solicited symptom after one dose without having recorded any daily measurement will be considered as having symptom and will be considered in subjects who experiences the symptom but will not be considered in the specific information by grade.
    - Doses without symptom sheets documented will be excluded.
- For analysis of unsolicited AEs, SAEs and for the analysis of concomitant medications, all vaccinated subjects will be considered. Subjects who did not report an event or concomitant medication will be considered as subjects without the event or the concomitant medication respectively.
- Related dose: The related dose for an event (e.g., AE, medication, vaccination...) is the study dose given before an event. In case the event takes place on a day a study dose is given, the related dose will be that of the study dose even if the event actually took place before. For instance, for a conc. medication started on the day of study dose 2 but before dose 2 administrations, the related dose will be dose 2.
- The maximum intensity of local injection site redness and swelling will be scored at GSK Biologicals as follows:

0 · None

1: < 5 mm

2:5 to 20 mm

3: > 20 mm

• Fever is defined as temperature ≥ 37.5°C / 99.5°F for oral, axillary or tympanic route, or ≥ 38.0°C / 100.4°F for rectal route. The preferred route for recording temperature in this study will be axillary. For the analysis, temperatures will be coded as follows:

| Grade | Temperature (oral, axillary or tympanic route) | Temperature (rectal route) |
|---|---|---|
| 0 | < 37.5°C | < 38°C |
| 1 | ≥ 37.5°C - ≤ 38.5°C | ≥ 38°C - ≤ 39°C |
| 2 | > 38.5°C - ≤ 39.5°C | > 39°C - ≤ 40°C |
| 3 | > 39.5°C | > 40°C |

- Conversion of temperature to °C
  - Temperature in °Celsius = ((Temperature in °Fahrenheit -32) \*5)/9.
  - The result is rounded to 1 decimal.
- Note that for all tables described in this section, the way the percentage of subjects will be derived will depend on the event analysed (see table below for details). As a result, the N value will differ from one table to another.

| Event | N used for deriving % per subject for Vaccination phase | N used for deriving % per dose for<br>Vaccination phase |
|---|---|---|
| Concomitant vaccination | All subjects with study vaccine administered | All study visits with study vaccine administered |
| Solicited<br>general<br>symptom | All subjects with at least one solicited general symptom documented as either present or absent (i.e., symptom screen completed) | All study visits with study vaccine administered and with at least one solicited general symptom documented as either present or absent (i.e., symptom screen completed) |
| Solicited local symptom | All subjects with at least one solicited local symptom documented as either present or absent (i.e., symptom screen completed) | All study visits with study vaccine administered and with at least one solicited local symptom documented as either present or absent (i.e., symptom screen completed) |
| Unsolicited symptom | All subjects with study vaccine administered | All study visits with study vaccine administered |
| Concomitant medication | All subjects with study vaccine administered | All study visits with study vaccine administered |

- All CI computed will be two-sided 95% CI.
- Grading of haematological and biochemical parameters will be assessed as per the following tables: -

Table 4 Toxicity grading scales for hematology and biochemistry parameters applicable for this study

| Component | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
|---|---|---|---|---|
| Hemoglobin (g/dL) | 9.0 to < 10.5 | 8.0 to < 9.0 | 7.0 to < 8.0 | < 7.0 |
| Leukocytes decreased (cell/mm³) | 2500 to < 3500 | 1500 to < 2500 | 1000 to < 1500 | < 1000 |
| Platelets decreased (cell//mm³) | 75000 to < 150000 | 50000 to < 75000 | 25000 to < 50000 | < 25000 |
| Alanine Aminotransferase (increase by factor) | 1.1 to < 2.0 xULN | 2.0 to < 3.0 xULN | $3.00 \text{ to} \leq 8.0 \text{ xULN}$ | > 8.0 xULN |
| Aspartate Aminotransferase (increase by factor) | 1.1 to < 2.0 xULN | 2.0 to < 3.0 xULN | $3.00 \text{ to} \leq 8.0 \text{ xULN}$ | > 8.0 xULN |
| Creatinine (mg/dL) | 0.6 to < 0.9 | 0.9 to < 1.2 | $1.2 \text{ to} \leq 1.5$ | > 1.5 |
| Absolute neutrophil count decreased (cell/mm³) | 1000 to < 1300 | 750 to < 1000 | 500 to < 750 | < 500 |
| Absolute lymphocyte count decreased (cell/mm³) | 600 to < 650 | 500 to < 600 | 350 to < 500 | < 350 |
| Eosinophil | N.A | N.A | N.A | N.A |
| Basophil | N.A | N.A | N.A | N.A |
| Monocyte | N.A | N.A | N.A | N.A |

Grading scale adapted from [, 2003], [, 2004] and [, 2007].

**ULN**: upper limit of normal

#### 11.3.6. RTI and LRTI

• For the analysis of RTI and LRTI, all cases will be definitively classified as either RSV-RTI, RSV-LRTI, RSV-severe LRTI or RSV-very severe LRTI according to standardized case definitions (see table below) based on the available WHO case definitions, and the association to RSV infection will be assessed by quantitative PCR as primary analysis.

Table 5 Case definition of RSV- RTI/LRTI

| RSV infection | Symptomatic and/or asymptomatic RSV infection |
|---|---|
| RSV-RTI | Runny nose OR blocked nose OR cough |
| | AND |
| | Confirmed RSV infection <sup>4</sup> |
| RSV-LRTI | History of cough OR difficulty breathing <sup>1</sup> |
| | AND |
| | SpO <sub>2</sub> < 95% <sup>2</sup> , OR RR increase <sup>3</sup> |
| | AND |
| | Confirmed RSV infection <sup>4</sup> |
| RSV-severe LRTI | Meeting the case definition of RSV-LRTI |
| | AND |
| | SpO <sub>2</sub> < 93% <sup>2</sup> , OR lower chest wall in-drawing |
| RSV-very severe LRTI | Meeting the case definition of RSV-LRTI |
| | AND |
| | SpO <sub>2</sub> < 90% <sup>2</sup> , OR inability to feed, OR failure to respond / unconscious |
| RSV hospitalization | Confirmed RSV infection 5 |
| | AND |
| | Hospitalized for acute medical condition <sup>6</sup> |
| All-cause LRTI | History of cough OR difficulty breathing <sup>1</sup> |
| | AND |
| | SpO <sub>2</sub> < 95% <sup>2</sup> , OR RR increase <sup>3</sup> |

Definition based on [Modjarrad, 2016]

LRTI = lower respiratory tract infections; RR = respiratory rate; RTI = respiratory tract infections;

SpO<sub>2</sub> = blood oxygen saturatin

- For the analysis of RSV-RTI episode, the start date of an RTI episode will be defined as the first day of any occurrence of cough, runny nose, blocked nose, and a new case requires an interval of at least 7 symptom free days since the last episode of RTI that was diagnosed.
- For the analysis of RSV-LRTI or severe or very severe LRTI the start date of the LRTI episode is defined as the point at which the first symptoms of cough, or difficulty breathing were observed and a new case requires an interval of at least 7 symptom free days since the last episode of LRTI that was diagnosed.

<sup>&</sup>lt;sup>1</sup> Based on history reported by parents/LARs and includes difficulty breathing (e.g. showing signs of wheezing or stridor, tachypnoea, flaring [of nostrils], chest in-drawing, apnoea) associated with nasal obstruction

<sup>&</sup>lt;sup>2</sup> For blood oxygen saturation (SpO<sub>2</sub>), the lowest value monitored will be used

<sup>&</sup>lt;sup>3</sup> RR increase defined as  $\geq$  40/minute (12 months of age or above)

<sup>&</sup>lt;sup>4</sup> RSV infection confirmed on nasal swab positive for RSV A or B by quantitative Reverse Transcription Polymerase Chain Reaction (qRT-PCR)

<sup>&</sup>lt;sup>5</sup> RSV sampling and testing is based on medical judgment of medical practitioner or driven by algorithm

<sup>6</sup> Hospitalization is defined as a medical decision that the infant requires admission for observation or treatment

- End date of the RTI episode is defined as the point at which the child is considered symptom-free of cough, runny nose, blocked nose, wheezing, and difficulty breathing.
- For molecular biology (qRT-PCR test), the following cut-off will be applied: -

| System | Component | Method | Unit | Cut-off |
|---|---|---|---|---|
| Nasal swab | RSV-A RNA | Quantitative real-time PCR (qRT-PCR) | Copies/ml | 1123 |
| Nasal swab | RSV-B RNA | Quantitative real-time PCR (qRT-PCR) | Copies/ml | 1467 |

• For calculation of viral load for RSV-A/B, all reported values will be included. Subject infected by either RSV-A or RSV-B or both will be included for calculation. Total viral load = Viral load for RSV-A + Viral load for RSV-B. LOD for RSV-A and RSV-B are 1123 and 1467 copies/ml, respectively. Following rule will be applied: -

| Raw result | Derivation for positivity | Derivation for viral<br>load calculation |
|---|---|---|
| <lod< td=""><td>NEG</td><td>LOD/2</td></lod<> | NEG | LOD/2 |
| ≥LOD | POS | Exact value |

#### 11.3.7. Number of decimals displayed

The following decimal description from the decision rules will be used for the demography, immunogenicity and safety/reactogenicity.

| Display Table | Parameters | Number of decimal digits |
|---|---|---|
| Demographic characteristics | Mean, median age | 1 |
| Demographic characteristics | SD (age) | 1 |
| Reactogenicity | Mean, Min, Q1, Median, Q3, Max for duration | 1 |
| All summaries | % of count, including LL & UL of CI | 1 |
| All summaries | % of difference, including LL & UL of CI | 2 |

### 12. ANNEX 2: RELEVANT PREFERRED TERMS FOR DETECTION OF AESI

Any of the below listed preferred term reported as an Expedited Adverse Event must be immediately escalated to the CRDL or Central Safety Physician to assess or confirm the need for an urgent IDMC review.

The list of preferred terms and associated PT codes is given below:

#### **HAEMATOMA**

| HALMATOMA | 1 |
|------------------------------------|----------|
| Preferred term | PT code |
| abdominal wall haematoma | 10067383 |
| administration site haematoma | 10075100 |
| adrenal haematoma | 10059194 |
| aortic intramural haematoma | 10067975 |
| application site haematoma | 10068317 |
| arterial intramural haematoma | 10074971 |
| auricular haematoma | 10003797 |
| basal ganglia haematoma | 10077031 |
| brain stem haematoma | 10073230 |
| breast haematoma | 10064753 |
| broad ligament haematoma | 10006375 |
| bursal haematoma | 10077818 |
| catheter site haematoma | 10055662 |
| cephalhaematoma | 10008014 |
| cerebellar haematoma | 10061038 |
| cerebral haematoma | 10053942 |
| cervix haematoma uterine | 10050020 |
| chest wall haematoma | 10076597 |
| colonic haematoma | 10009996 |
| deep dissecting haematoma | 10074718 |
| extradural haematoma | 10015769 |
| eyelid haematoma | 10064976 |
| haematoma | 10018852 |
| haematoma evacuation | 10060733 |
| haematoma infection | 10051564 |
| hepatic haematoma | 10019676 |
| incision site haematoma | 10059241 |
| infusion site haematoma | 10065463 |
| injection site haematoma | 10022066 |
| instillation site haematoma | 10073609 |
| intestinal haematoma | 10069829 |
| intra-abdominal haematoma | 10056457 |
| intracerebral haematoma evacuation | 10062025 |

204838 (RSV PED-002) Statistical Analysis Plan Final

| intracranial haematoma 10059491 intraocular haematoma 10071934 laryngeal haematoma 10066304 mediastinal haematoma 10049941 mediastinal haematoma 10075577 mesenteric haematoma 10075577 mesenteric haematoma 10075027 oesophageal intramural haematoma 100774786 oral mucosa haematoma 10074779 ovarian haematoma 10074779 ovarian haematoma 10054974 perlic haematoma 10054974 perlic haematoma 10070656 perineal haematoma 10074520 periorbital haematoma 10074520 periorbital haematoma 10074542 periorbeal haematoma 100749450 peritoneal haematoma 10058095 pharyngeal haematoma 10068121 post procedural haematoma 10063188 pulmonary haematoma 10058095 pretroperitoneal haematoma 10058095 spinal epidural haematoma 10058060 scrotal haematoma 10076051 spinal epidura | | |
|---|---|---|
| laryngeal haematoma 10070885 lip haematoma 10066304 mediastinal haematoma 10049941 medical device site haematoma 10075577 mesenteric haematoma 10071557 nasal septum haematoma 10075027 oesophageal intramural haematoma 10074779 ovarian haematoma 10074779 ovarian haematoma 1003263 paranasal sinus haematoma 10069702 pelvic haematoma 10070656 perineal haematoma 10034520 periorbital haematoma 10034520 periorbital haematoma 100749450 peritoneal haematoma 100734544 periorseal haematoma 10058095 pharyngeal haematoma 10068121 post procedural haematoma 10068121 post procedural haematoma 10054991 renal haematoma 10058360 scrotal haematoma 10076051 spinal cord haematoma 10076051 spinal epidural haematoma 10050162 spinal subdural haematoma 10065304 subcut | intracranial haematoma | 10059491 |
| lip haematoma 10066304 mediastinal haematoma 10049941 medical device site haematoma 10075577 mesenteric haematoma 10071557 nasal septum haematoma 10075027 oesophageal intramural haematoma 10074786 oral mucosa haematoma 10074779 ovarian haematoma 10034263 paranasal sinus haematoma 10054974 perlie haematoma 10054974 penile haematoma 10070656 perineal haematoma 10034520 periorbital haematoma 10034520 periorbital haematoma 10074950 peritoneal haematoma 10073454 periorbital haematoma 10049450 peritoneal haematoma 10058095 pharyngeal haematoma 10068121 post procedural haematoma 10068121 post procedural haematoma 10054991 renal haematoma 10074991 renal haematoma 10076051 spinal cord haematoma 10076051 spinal epidural haematoma 10076051 spinal subdu | intraocular haematoma | 10071934 |
| mediastinal haematoma 10049941 medical device site haematoma 10075577 mesenteric haematoma 10071557 nasal septum haematoma 10075027 oesophageal intramural haematoma 1007486 oral mucosa haematoma 10074779 ovarian haematoma 10069702 pelvic haematoma 10054974 penile haematoma 10070656 perineal haematoma 10034520 periorbital haematoma 10073441 perirenal haematoma 10073441 perirenal haematoma 10073441 perirenal haematoma 10058095 pharyngeal haematoma 10068121 post procedural haematoma 10054991 renal haematoma 10054991 renal haematoma 1005895 retroperitoneal haematoma 1005895 retroperitoneal haematoma 1005895 retroperitoneal haematoma 10058960 scrotal haematoma 10076051 spinal epidural haematoma 10076051 spinal subdural haematoma 10050164 splenic haematoma 10076701 subcutaneous haematoma 10042345 subdural haematoma 10042345 subdural haematoma 10042361 subgaleal haematoma 10071935 tongue haematoma 10063875 vaccination site haematoma 10069472 vaginal haematoma 1006990 vitreous haematoma 10071936 | laryngeal haematoma | 10070885 |
| medical device site haematoma 10075577 mesenteric haematoma 10071557 nasal septum haematoma 10075027 oesophageal intramural haematoma 10074786 oral mucosa haematoma 10074779 ovarian haematoma 10069702 pelvic haematoma 10054974 penile haematoma 10034520 periorbital haematoma 10034520 periorbital haematoma 10073444 periosteal haematoma 10073454 peritoneal haematoma 10073454 peritoneal haematoma 10073454 peritoneal haematoma 1007341 perirenal haematoma 1007341 peritoneal haematoma 10058095 pharyngeal haematoma 10068121 post procedural haematoma 10063188 pulmonary haematoma 10054991 renal haematoma 10054991 renal haematoma 10054991 retroperitoneal haematoma 10038459 retroperitoneal haematoma 10076051 spinal epidural haematoma 10076051 spinal epidural haematoma 10050162 spinal subdural haematoma 10050164 splenic haematoma 10065304 subarachnoid haematoma 10076701 subcutaneous haematoma 10042345 subdural haematoma 10042345 subdural haematoma 10042345 subdural haematoma 10043959 uterine haematoma 10063875 vaccination site haematoma 10069472 vaginal haematoma 1006990 vitreous haematoma 10071936 | lip haematoma | 10066304 |
| mesenteric haematoma 10071557 nasal septum haematoma 10075027 oesophageal intramural haematoma 10077486 oral mucosa haematoma 10074779 ovarian haematoma 10033263 paranasal sinus haematoma 10069702 pelvic haematoma 10054974 penile haematoma 10070656 perineal haematoma 10034520 periorbital haematoma 10034544 periosteal haematoma 10077341 perirenal haematoma 10058095 pharyngeal haematoma 10068121 post procedural haematoma 10054991 renal haematoma 10054991 renal haematoma 10058360 scrotal haematoma 10058360 scrotal haematoma 10076051 spinal epidural haematoma 10050162 spinal subdural haematoma 10065304 subarachnoid haematoma 10076701 subcutaneous haematoma 10042345 subdural haematoma 10076701 subcutaneous haematoma 10042361 subgaleal haematoma 10071935 tongue haematoma 10043959 uterine haematoma 10043959 vitreous haematoma 10046909 vitreous haematoma 10046909 vitreous haematoma 10046909 | mediastinal haematoma | 10049941 |
| nasal septum haematoma10075027oesophageal intramural haematoma10077486oral mucosa haematoma10074779ovarian haematoma10033263paranasal sinus haematoma10069702pelvic haematoma10070656perineal haematoma10034520periorbital haematoma10034544periosteal haematoma10077341perirenal haematoma10049450peritoneal haematoma10058095pharyngeal haematoma10068121post procedural haematoma10054991renal haematoma10038459retroperitoneal haematoma10058360scrotal haematoma10076051spinal cord haematoma10076051spinal epidural haematoma10050162spinal subdural haematoma10050164splenic haematoma10041646spontaneous haematoma10045304subcutaneous haematoma10042361subdural haematoma10042361subgaleal haematoma10042361subretinal haematoma10049510subretinal haematoma10043959uterine haematoma10069875vaccination site haematoma10046909vitreous haematoma10046909vitreous haematoma10071936 | medical device site haematoma | 10075577 |
| oesophageal intramural haematoma oral mucosa haematoma 10074779 ovarian haematoma 10033263 paranasal sinus haematoma 10069702 pelvic haematoma 10054974 penile haematoma 10070656 perineal haematoma 10034520 periorbital haematoma 10034544 periosteal haematoma 10077341 perirenal haematoma 10077341 perirenal haematoma 10058095 pharyngeal haematoma 10068121 post procedural haematoma 10068121 post procedural haematoma 10068121 post procedural haematoma 10058095 retroperitoneal haematoma 100584991 renal haematoma 10058459 retroperitoneal haematoma 10058360 scrotal haematoma 10076051 spinal epidural haematoma 10076051 spinal epidural haematoma 10050162 spinal subdural haematoma 10041646 spontaneous haematoma 10076701 subcutaneous haematoma 10076701 subcutaneous haematoma 10042345 subdural haematoma 10042361 subgaleal haematoma 10071935 tongue haematoma 10043959 uterine haematoma 10046909 vitreous haematoma 10046909 vitreous haematoma 10046909 vitreous haematoma 10071935 | mesenteric haematoma | 10071557 |
| oral mucosa haematoma 10074779 ovarian haematoma 10033263 paranasal sinus haematoma 10069702 pelvic haematoma 10054974 penile haematoma 10070656 perineal haematoma 10034520 periorbital haematoma 10034544 periosteal haematoma 10077341 perirenal haematoma 10049450 peritoneal haematoma 10058095 pharyngeal haematoma 10068121 post procedural haematoma 10063188 pulmonary haematoma 10054991 renal haematoma 10038459 retroperitoneal haematoma 10038459 retroperitoneal haematoma 10076051 spinal epidural haematoma 10050162 spinal subdural haematoma 1005164 splenic haematoma 10041646 spontaneous haematoma 10042361 subgaleal haematoma 10042345 subgaleal haematoma 10076701 subcutaneous haematoma 10042361 subgaleal haematoma 10071935 tongue haematoma 10043959 uterine haematoma 10069472 vaginal haematoma 10046909 vitreous haematoma 10046909 | nasal septum haematoma | 10075027 |
| ovarian haematoma 10033263 paranasal sinus haematoma 10069702 pelvic haematoma 10054974 penile haematoma 10070656 perineal haematoma 10034520 periorbital haematoma 10034544 periosteal haematoma 10077341 perirenal haematoma 10058095 pharyngeal haematoma 10068121 post procedural haematoma 10063188 pulmonary haematoma 100584991 renal haematoma 100584991 renal haematoma 100584991 retroperitoneal haematoma 10058360 scrotal haematoma 10076051 spinal cord haematoma 10076051 spinal subdural haematoma 10050162 spinal subdural haematoma 10065304 splenic haematoma 10041646 spontaneous haematoma 10042361 subgaleal haematoma 10042361 subgaleal haematoma 1007935 tongue haematoma 10043959 uterine haematoma 10063875 vaccination site haematoma 10069472 vaginal haematoma 10046909 vitreous haematoma 10071936 | oesophageal intramural haematoma | 10077486 |
| paranasal sinus haematoma 10054974 pelvic haematoma 10054974 penile haematoma 10070656 perineal haematoma 10034520 periorbital haematoma 10034544 periosteal haematoma 10077341 perirenal haematoma 10049450 peritoneal haematoma 10058095 pharyngeal haematoma 10068121 post procedural haematoma 10054991 renal haematoma 100584991 renal haematoma 10058459 retroperitoneal haematoma 10058360 scrotal haematoma 10076051 spinal cord haematoma 10050162 spinal subdural haematoma 10050164 splenic haematoma 10041646 spontaneous haematoma 10041646 spontaneous haematoma 10042361 subgaleal haematoma 10042361 subgaleal haematoma 1007935 tongue haematoma 10043959 uterine haematoma 10069372 vaginal haematoma 10069472 vaginal haematoma 10046909 vitreous haematoma 10071936 | oral mucosa haematoma | 10074779 |
| pelvic haematoma 10054974 penile haematoma 10070656 perineal haematoma 10034520 periorbital haematoma 10034544 periosteal haematoma 10077341 perirenal haematoma 10049450 peritoneal haematoma 10058095 pharyngeal haematoma 10068121 post procedural haematoma 10063188 pulmonary haematoma 10054991 renal haematoma 10038459 retroperitoneal haematoma 10038459 retroperitoneal haematoma 10039749 spinal cord haematoma 10076051 spinal epidural haematoma 10050162 spinal subdural haematoma 10041646 spontaneous haematoma 10076701 subcutaneous haematoma 10042345 subdural haematoma 10042361 subgaleal haematoma 10042361 subgaleal haematoma 10071935 tongue haematoma 10069570 vaccination site haematoma 10069472 vaginal haematoma 10046909 vitreous haematoma 10071936 | ovarian haematoma | 10033263 |
| penile haematoma 10070656 perineal haematoma 10034520 periorbital haematoma 10034544 periosteal haematoma 10077341 perirenal haematoma 10049450 peritoneal haematoma 10058095 pharyngeal haematoma 10068121 post procedural haematoma 10054991 renal haematoma 10054991 renal haematoma 10058360 scrotal haematoma 10038459 retroperitoneal haematoma 10039749 spinal cord haematoma 10076051 spinal epidural haematoma 10050162 spinal subdural haematoma 10050164 splenic haematoma 10065304 subarachnoid haematoma 10076701 subcutaneous haematoma 10042345 subdural haematoma 10042361 subgaleal haematoma 10071935 tongue haematoma 10063875 vaccination site haematoma 10069972 vaginal haematoma 1006909 vitreous haematoma 10071936 | paranasal sinus haematoma | 10069702 |
| perineal haematoma 10034520 periorbital haematoma 10034544 periosteal haematoma 10077341 perirenal haematoma 10049450 peritoneal haematoma 10058095 pharyngeal haematoma 10068121 post procedural haematoma 10063188 pulmonary haematoma 10054991 renal haematoma 10058360 scrotal haematoma 10038459 retroperitoneal haematoma 10076051 spinal cord haematoma 10050162 spinal subdural haematoma 10050164 splenic haematoma 10041646 spontaneous haematoma 10076701 subcutaneous haematoma 10042345 subdural haematoma 10042361 subgaleal haematoma 10071935 tongue haematoma 10063875 vaccination site haematoma 10069972 vaginal haematoma 10046909 vitreous haematoma 10071936 | pelvic haematoma | 10054974 |
| periorbital haematoma 10034544 periosteal haematoma 10077341 perirenal haematoma 10049450 peritoneal haematoma 10058095 pharyngeal haematoma 10068121 post procedural haematoma 10054991 renal haematoma 10054991 renal haematoma 10038459 retroperitoneal haematoma 10058360 scrotal haematoma 10039749 spinal cord haematoma 10076051 spinal epidural haematoma 10050162 spinal subdural haematoma 10050164 splenic haematoma 10041646 spontaneous haematoma 10076701 subcutaneous haematoma 10042345 subdural haematoma 10042361 subgaleal haematoma 10079510 subretinal haematoma 10071935 tongue haematoma 10063875 vaccination site haematoma 10069972 vaginal haematoma 10046909 vitreous haematoma 10071936 | penile haematoma | 10070656 |
| periosteal haematoma 10077341 perirenal haematoma 10049450 peritoneal haematoma 10058095 pharyngeal haematoma 10068121 post procedural haematoma 10054991 renal haematoma 10054991 renal haematoma 10038459 retroperitoneal haematoma 10038360 scrotal haematoma 10039749 spinal cord haematoma 10076051 spinal epidural haematoma 10050162 spinal subdural haematoma 10050164 splenic haematoma 10065304 subarachnoid haematoma 10076701 subcutaneous haematoma 10042345 subdural haematoma 10042361 subgaleal haematoma 10069510 subretinal haematoma 10071935 tongue haematoma 10063875 vaccination site haematoma 1006909 vitreous haematoma 10046909 vitreous haematoma 10071936 | perineal haematoma | 10034520 |
| perirenal haematoma 10049450 peritoneal haematoma 10058095 pharyngeal haematoma 10068121 post procedural haematoma 10063188 pulmonary haematoma 10054991 renal haematoma 10038459 retroperitoneal haematoma 10058360 scrotal haematoma 10039749 spinal cord haematoma 10076051 spinal epidural haematoma 10050162 spinal subdural haematoma 10050164 splenic haematoma 10041646 spontaneous haematoma 10065304 subarachnoid haematoma 10076701 subcutaneous haematoma 10042345 subdural haematoma 10042361 subgaleal haematoma 10071935 tongue haematoma 10063875 vaccination site haematoma 1006999 vitreous haematoma 10046909 vitreous haematoma 10071936 | periorbital haematoma | 10034544 |
| peritoneal haematoma 10058095 pharyngeal haematoma 10068121 post procedural haematoma 10063188 pulmonary haematoma 10054991 renal haematoma 10038459 retroperitoneal haematoma 10058360 scrotal haematoma 10039749 spinal cord haematoma 10076051 spinal epidural haematoma 10050162 spinal subdural haematoma 10050164 splenic haematoma 10041646 spontaneous haematoma 10065304 subarachnoid haematoma 10076701 subcutaneous haematoma 10042345 subdural haematoma 10042361 subgaleal haematoma 10071935 tongue haematoma 10063875 vaccination site haematoma 10046909 vitreous haematoma 10046909 | periosteal haematoma | 10077341 |
| pharyngeal haematoma 10068121 post procedural haematoma 10063188 pulmonary haematoma 10054991 renal haematoma 10038459 retroperitoneal haematoma 10058360 scrotal haematoma 10039749 spinal cord haematoma 10076051 spinal epidural haematoma 10050162 spinal subdural haematoma 10050164 splenic haematoma 10065304 subarachnoid haematoma 10076701 subcutaneous haematoma 10042345 subdural haematoma 10042361 subgaleal haematoma 10071935 tongue haematoma 10063875 vaccination site haematoma 1006999 vitreous haematoma 10046909 vitreous haematoma 10071936 | perirenal haematoma | 10049450 |
| post procedural haematoma 10063188 pulmonary haematoma 10054991 renal haematoma 10038459 retroperitoneal haematoma 10058360 scrotal haematoma 10039749 spinal cord haematoma 10076051 spinal epidural haematoma 10050162 spinal subdural haematoma 10050164 splenic haematoma 10041646 spontaneous haematoma 10076701 subcutaneous haematoma 10042345 subdural haematoma 10042345 subdural haematoma 10069510 subretinal haematoma 10071935 tongue haematoma 10063875 vaccination site haematoma 10046909 vitreous haematoma 10071936 | peritoneal haematoma | 10058095 |
| pulmonary haematoma 10054991 renal haematoma 10038459 retroperitoneal haematoma 10058360 scrotal haematoma 10039749 spinal cord haematoma 10076051 spinal epidural haematoma 10050162 spinal subdural haematoma 10050164 splenic haematoma 10041646 spontaneous haematoma 10065304 subarachnoid haematoma 10076701 subcutaneous haematoma 10042345 subdural haematoma 10042361 subgaleal haematoma 10071935 tongue haematoma 10063875 vaccination site haematoma 10069472 vaginal haematoma 10046909 vitreous haematoma 10071936 | pharyngeal haematoma | 10068121 |
| renal haematoma 10038459 retroperitoneal haematoma 10058360 scrotal haematoma 10039749 spinal cord haematoma 10076051 spinal epidural haematoma 10050162 spinal subdural haematoma 10050164 splenic haematoma 10041646 spontaneous haematoma 10065304 subarachnoid haematoma 10076701 subcutaneous haematoma 10042345 subdural haematoma 10042361 subgaleal haematoma 10071935 tongue haematoma 10043959 uterine haematoma 10069472 vaginal haematoma 10046909 vitreous haematoma 10071936 | post procedural haematoma | 10063188 |
| retroperitoneal haematoma 10058360 scrotal haematoma 10039749 spinal cord haematoma 10076051 spinal epidural haematoma 10050162 spinal subdural haematoma 10050164 splenic haematoma 10041646 spontaneous haematoma 10065304 subarachnoid haematoma 10076701 subcutaneous haematoma 10042345 subdural haematoma 10042361 subgaleal haematoma 10069510 subretinal haematoma 10071935 tongue haematoma 10063875 vaccination site haematoma 10069472 vaginal haematoma 10046909 vitreous haematoma 10071936 | pulmonary haematoma | 10054991 |
| scrotal haematoma 10039749 spinal cord haematoma 10076051 spinal epidural haematoma 10050162 spinal subdural haematoma 10050164 splenic haematoma 10041646 spontaneous haematoma 10065304 subarachnoid haematoma 10076701 subcutaneous haematoma 10042345 subdural haematoma 10042361 subgaleal haematoma 10069510 subretinal haematoma 10071935 tongue haematoma 10063875 vaccination site haematoma 10069472 vaginal haematoma 10046909 vitreous haematoma 10071936 | renal haematoma | 10038459 |
| spinal cord haematoma 10076051 spinal epidural haematoma 10050162 spinal subdural haematoma 10050164 splenic haematoma 10041646 spontaneous haematoma 10065304 subarachnoid haematoma 10076701 subcutaneous haematoma 10042345 subdural haematoma 10042361 subgaleal haematoma 10069510 subretinal haematoma 10071935 tongue haematoma 10063875 vaccination site haematoma 10069472 vaginal haematoma 10046909 vitreous haematoma 10071936 | retroperitoneal haematoma | 10058360 |
| spinal epidural haematoma 10050162 spinal subdural haematoma 10050164 splenic haematoma 10041646 spontaneous haematoma 10065304 subarachnoid haematoma 10076701 subcutaneous haematoma 10042345 subdural haematoma 10042361 subgaleal haematoma 10069510 subretinal haematoma 10071935 tongue haematoma 10063875 vaccination site haematoma 10069472 vaginal haematoma 10046909 vitreous haematoma 10071936 | scrotal haematoma | 10039749 |
| spinal subdural haematoma 10050164 splenic haematoma 10041646 spontaneous haematoma 10065304 subarachnoid haematoma 10076701 subcutaneous haematoma 10042345 subdural haematoma 10042361 subgaleal haematoma 10069510 subretinal haematoma 10071935 tongue haematoma 10063875 vaccination site haematoma 10069472 vaginal haematoma 10046909 vitreous haematoma 10071936 | spinal cord haematoma | 10076051 |
| splenic haematoma 10041646 spontaneous haematoma 10065304 subarachnoid haematoma 10076701 subcutaneous haematoma 10042345 subdural haematoma 10042361 subgaleal haematoma 10069510 subretinal haematoma 10071935 tongue haematoma 10063875 vaccination site haematoma 10069472 vaginal haematoma 10046909 vitreous haematoma 10071936 | spinal epidural haematoma | 10050162 |
| spontaneous haematoma 10065304 subarachnoid haematoma 10076701 subcutaneous haematoma 10042345 subdural haematoma 10042361 subgaleal haematoma 10069510 subretinal haematoma 10071935 tongue haematoma 10043959 uterine haematoma 10063875 vaccination site haematoma 10069472 vaginal haematoma 10046909 vitreous haematoma 10071936 | spinal subdural haematoma | 10050164 |
| subarachnoid haematoma 10076701 subcutaneous haematoma 10042345 subdural haematoma 10042361 subgaleal haematoma 10069510 subretinal haematoma 10071935 tongue haematoma 10043959 uterine haematoma 10063875 vaccination site haematoma 10069472 vaginal haematoma 10046909 vitreous haematoma 10071936 | splenic haematoma | 10041646 |
| subcutaneous haematoma10042345subdural haematoma10042361subgaleal haematoma10069510subretinal haematoma10071935tongue haematoma10043959uterine haematoma10063875vaccination site haematoma10069472vaginal haematoma10046909vitreous haematoma10071936 | spontaneous haematoma | 10065304 |
| subdural haematoma10042361subgaleal haematoma10069510subretinal haematoma10071935tongue haematoma10043959uterine haematoma10063875vaccination site haematoma10069472vaginal haematoma10046909vitreous haematoma10071936 | subarachnoid haematoma | 10076701 |
| subgaleal haematoma10069510subretinal haematoma10071935tongue haematoma10043959uterine haematoma10063875vaccination site haematoma10069472vaginal haematoma10046909vitreous haematoma10071936 | subcutaneous haematoma | 10042345 |
| subretinal haematoma10071935tongue haematoma10043959uterine haematoma10063875vaccination site haematoma10069472vaginal haematoma10046909vitreous haematoma10071936 | subdural haematoma | 10042361 |
| tongue haematoma 10043959 uterine haematoma 10063875 vaccination site haematoma 10069472 vaginal haematoma 10046909 vitreous haematoma 10071936 | subgaleal haematoma | 10069510 |
| uterine haematoma10063875vaccination site haematoma10069472vaginal haematoma10046909vitreous haematoma10071936 | subretinal haematoma | 10071935 |
| vaccination site haematoma10069472vaginal haematoma10046909vitreous haematoma10071936 | tongue haematoma | 10043959 |
| vaginal haematoma10046909vitreous haematoma10071936 | uterine haematoma | 10063875 |
| vitreous haematoma 10071936 | vaccination site haematoma | 10069472 |
| | vaginal haematoma | 10046909 |
| vulval haematoma 10047756 | vitreous haematoma | 10071936 |
| | vulval haematoma | 10047756 |

#### **HAEMORRHAGE**

| HALMORRIAGE | |
|----------------------------------------|----------|
| Preferred term | PT code |
| abdominal wall haemorrhage | 10067788 |
| acute haemorrhagic conjunctivitis | 10067817 |
| administration site haemorrhage | 10075101 |
| adrenal haemorrhage | 10001361 |
| anal haemorrhage | 10049555 |
| anastomotic haemorrhage | 10056346 |
| angina bullosa haemorrhagica | 10064223 |
| application site haemorrhage | 10072694 |
| arterial haemorrhage | 10060964 |
| basal ganglia haemorrhage | 10067057 |
| bone marrow haemorrhage | 10073581 |
| brain stem haemorrhage | 10006145 |
| brain stem microhaemorrhage | 10071205 |
| breast haemorrhage | 10006254 |
| bronchial haemorrhage | 10065739 |
| catheter site haemorrhage | 10051099 |
| central nervous system haemorrhage | 10072043 |
| cerebellar haemorrhage | 10008030 |
| cerebellar microhaemorrhage | 10071206 |
| cerebral haemorrhage | 10008111 |
| cerebral microhaemorrhage | 10067277 |
| cervix haemorrhage uterine | 10050022 |
| ciliary body haemorrhage | 10057417 |
| conjunctival haemorrhage | 10010719 |
| diverticulitis intestinal haemorrhagic | 10013541 |
| diverticulum intestinal haemorrhagic | 10013560 |
| duodenitis haemorrhagic | 10013865 |
| ear haemorrhage | 10014009 |
| encephalitis haemorrhagic | 10014589 |
| gastric haemorrhage | 10017788 |
| gastroduodenal haemorrhage | 10053768 |
| gastrointestinal haemorrhage | 10017955 |
| genital haemorrhage | 10061178 |
| haemarthrosis | 10018829 |
| haematemesis | 10018830 |
| haematochezia | 10018836 |
| haematotympanum | 10063013 |
| haematuria | 10018867 |
| haemorrhage | 10055798 |
| haemorrhage coronary artery | 10055803 |

204838 (RSV PED-002) Statistical Analysis Plan Final

| Г | 1 |
|------------------------------------|----------|
| haemorrhage intracranial | 10018985 |
| haemorrhage subcutaneous | 10018999 |
| haemorrhage subepidermal | 10019001 |
| haemorrhage urinary tract | 10055847 |
| haemorrhagic anaemia | 10052293 |
| haemorrhagic diathesis | 10062713 |
| haemorrhagic disorder | 10019009 |
| haemorrhagic infarction | 10019013 |
| haemorrhagic ovarian cyst | 10060781 |
| haemorrhagic pneumonia | 10077933 |
| haemorrhagic thyroid cyst | 10072256 |
| haemorrhagic urticaria | 10059499 |
| injection site haemorrhage | 10022067 |
| internal haemorrhage | 10075192 |
| intestinal haemorrhage | 10059175 |
| intra-abdominal haemorrhage | 10061249 |
| intraventricular haemorrhage | 10022840 |
| iris haemorrhage | 10057418 |
| joint microhaemorrhage | 10077666 |
| lacrimal haemorrhage | 10069930 |
| large intestinal haemorrhage | 10052534 |
| laryngeal haemorrhage | 10065740 |
| lip haemorrhage | 10049297 |
| lower gastrointestinal haemorrhage | 10050953 |
| lymph node haemorrhage | 10074270 |
| mediastinal haemorrhage | 10056343 |
| mesenteric haemorrhage | 10060717 |
| mouth haemorrhage | 10028024 |
| mucocutaneous haemorrhage | 10076048 |
| mucosal haemorrhage | 10061298 |
| muscle haemorrhage | 10028309 |
| myocardial haemorrhage | 10048849 |
| naevus haemorrhage | 10062955 |
| ocular retrobulbar haemorrhage | 10057571 |
| oesophageal haemorrhage | 10030172 |
| optic disc haemorrhage | 10030919 |
| optic nerve sheath haemorrhage | 10030941 |
| ovarian haemorrhage | 10065741 |
| pancreatic haemorrhage | 10033625 |
| papillary muscle haemorrhage | 10059164 |
| parathyroid haemorrhage | 10059051 |
| | 10033031 |

204838 (RSV PED-002) Statistical Analysis Plan Final

| | T |
|------------------------------------|----------|
| pelvic haemorrhage | 10063678 |
| penile haemorrhage | 10034305 |
| pericardial haemorrhage | 10034476 |
| periorbital haemorrhage | 10071697 |
| peritoneal haemorrhage | 10034666 |
| petechiae | 10034754 |
| pharyngeal haemorrhage | 10034827 |
| pituitary haemorrhage | 10049760 |
| post procedural haemorrhage | 10051077 |
| procedural haemorrhage | 10071229 |
| prostatic haemorrhage | 10036960 |
| pulmonary alveolar haemorrhage | 10037313 |
| pulmonary haemorrhage | 10037394 |
| putamen haemorrhage | 10058940 |
| rectal haemorrhage | 10038063 |
| renal haemorrhage | 10038460 |
| respiratory tract haemorrhage | 10038727 |
| retinal haemorrhage | 10038867 |
| retroperitoneal haemorrhage | 10038980 |
| scleral haemorrhage | 10050508 |
| skin haemorrhage | 10064265 |
| small intestinal haemorrhage | 10052535 |
| soft tissue haemorrhage | 10051297 |
| spermatic cord haemorrhage | 10065742 |
| spinal cord haemorrhage | 10048992 |
| spinal epidural haemorrhage | 10049236 |
| spinal subarachnoid haemorrhage | 10073564 |
| spinal subdural haemorrhage | 10073563 |
| splenic haemorrhage | 10041647 |
| spontaneous haemorrhage | 10074557 |
| subarachnoid haemorrhage | 10042316 |
| subdural haemorrhage | 10042364 |
| testicular haemorrhage | 10051877 |
| thalamus haemorrhage | 10058939 |
| thoracic haemorrhage | 10062744 |
| thyroid haemorrhage | 10064224 |
| tongue haemorrhage | 10049870 |
| tracheal haemorrhage | 10062543 |
| upper gastrointestinal haemorrhage | 10046274 |
| ureteric haemorrhage | 10065743 |
| urethral haemorrhage | 10049710 |
| urinary bladder haemorrhage | 10046528 |

| urogenital haemorrhage | 10050058 |
|------------------------------|----------|
| uterine haemorrhage | 10046788 |
| vaccination site haemorrhage | 10069475 |
| vaginal haemorrhage | 10046910 |
| venous haemorrhage | 10065441 |
| vitreous haemorrhage | 10047655 |
| vulval haemorrhage | 10063816 |

#### **THROMBOCYTOPENIA**

| Preferred term | PT code |
|---------------------------|----------|
| bleeding time abnormal | 10049227 |
| bleeding time prolonged | 10005140 |
| coagulation test abnormal | 10063557 |
| platelet count abnormal | 10035526 |
| platelet count decreased | 10035528 |
| platelet disorder | 10035532 |
| platelet dysfunction | 10073391 |
| thrombocytopenia | 10043554 |
| thrombocytopenic purpura | 10043561 |

#### LOWER RESPIRATORY TRACT INFECTION

| Preferred term | PT code |
|-------------------------------------------|----------|
| atypical pneumonia | 10003757 |
| bronchitis | 10006451 |
| bronchitis viral | 10053160 |
| haemorrhagic pneumonia | 10077933 |
| lower respiratory tract infection | 10024968 |
| lower respiratory tract infection viral | 10065188 |
| lung infection | 10061229 |
| pneumonia | 10035664 |
| pneumonia respiratory syncytial viral | 10035732 |
| pulmonary sepsis | 10051739 |
| respiratory syncytial virus bronchiolitis | 10038718 |
| respiratory syncytial virus bronchitis | 10069811 |
| respiratory tract infection | 10062352 |
| respiratory tract infection viral | 10062106 |

#### 13. ANNEX 3: STUDY SPECIFIC MOCK TFL

The data display, title and footnote is for illustration purpose and will be adapted to the study specificity as indicated in the TFL TOC. Note that there may be few changes between the study specific SAP mock TFL and the final TFLs as editorial/minor changes do not require a SAP amendment.

#### 13.1. List of individual data listing

Following individual data listing will be generated

Appendix Table I.A - Elimination codes

Appendix Table I.B – Demography

Appendix Table IBii - Physical examination/vital signs

Appendix Table I.Ci - Dates of birth, Informed consent, Vaccination and blood sampling, Contact

Appendix Table I.Cii - Reason for visit not done

Appendix Table I.D - General medical history - Physical examination

Appendix Table I.Ei – Study Conclusion

Appendix Table I.Eii – Screening conclusion

Appendix Table I.F – Notes (this appendix is provided for info only and should not be used for the clinical report)

Appendix Table I.G / I.H - Vaccination procedure

Appendix Table I.I - Reason for not administration of vaccine

Appendix Table I.J - Reason for non-eligibility

Appendix Table I.Ki – Previous history of vaccination

Appendix Table I.Kii - Previous history of disease

Appendix Table II.Ai - Solicited local adverse events

Appendix Table II.B - Solicited general adverse events

Appendix Table II.Ci - Unsolicited adverse events within (30) days post-vaccination

Appendix Table II.Cii - Unsolicited adverse events after (30) days post-vaccination

Appendix Table II.Di - Concomitant medications

Appendix Table II.Dii - Concomitant vaccinations

Appendix Table III.A – Immunogenicity - HI

Appendix Table III.B – Immunogenicity- CMI

Appendix Table IV.A – Haematology and Biochemistry

Appendix Table IIIA – Altitude of the site

Appendix Table IIE –Detection of Episodes and Limb Examination

Appendix Table IIF - Surveillance Contact

Appendix Table IIG - Assessment of RTI Episode

Appendix Table IIH - RTI Symptoms

Appendix Table IIJ - Signs and Symptoms of RSV-LRTI

Appendix Table IIK - Chest X-Ray Observations

Appendix Table IIL- Inpatient Care

Appendix Table IIIA – Local RSV Result

Appendix Table IIIB – Nasal Swab (qRT-PCR Result)

Appendix IIIC – Blood culture result

Appendix IIID- Re-screening

#### 13.2. Template of Tables and Figures

#### Template 1 Number of subjects by country and center <Exposed Set>

| | | | <each group=""><br/>N=XXXX</each> | | | Total<br>N=XXXX | |
|---|---|---|---|---|---|---|---|
| Country | Center | n | % | n | % | n | % |
| <each country=""></each> | <each center=""></each> | XXX | XX.X | XXX | XX.X | XXX | XX.X |
| | All | XXX | XX.X | XXX | XX.X | XXX | XX.X |

#### <each group>:

RSV-Ld = Low dose ChAd155-RSV vaccine (5 x 109 vp)

RSV-Md = Middle dose ChAd155-RSV vaccine (1.5 x 10<sup>10</sup> vp)

RSV-Hd = High dose ChAd155-RSV vaccine (5 x 10<sup>10</sup> vp)

Placebo-Ld = Non-active control (0.5 ml)

Placebo-Md = Non-active control (0.15 ml)

Placebo-Hd = Non-active control (0.5 ml)

n = number of subjects in a given center or country

N = total number of subjects

 $% = n/N \times 100$ 

Center = GSK Biologicals assigned center number

### Template 2 Number of subjects vaccinated, completed and withdrawn with reason for withdrawal – up to Day X <Exposed set>

| | <each group=""><br/>N=XXXX</each> | <each group=""><br/>N=XXXX</each> | Total<br>N=XXXX |
|---|---|---|---|
| | n | n | n |
| Number of subjects vaccinated | xxx | XXX | XXX |
| End of study status | | | |
| [EACH CATEGORY] | xxx | XXX | XXX |
| Reasons for withdrawal: | | | |
| [REASONS] | xxx | XXX | XXX |

#### <each group>:

RSV-Ld = Low dose ChAd155-RSV vaccine (5 x 109 vp)

RSV-Md = Middle dose ChAd155-RSV vaccine (1.5 x 10<sup>10</sup> vp)

RSV-Hd = High dose ChAd155-RSV vaccine (5 x  $10^{10}$  vp)

Placebo-Ld = Non-active control (0.5 ml)

Placebo-Md = Non-active control (0.15 ml)

Placebo-Hd = Non-active control (0.5 ml)

Vaccinated = number of subjects who were vaccinated in the study

Completed = number of subjects who completed last study visit

Withdrawn = number of subjects who did not come for the last study visit

#### Template 3 Visit attendance <Exposed set>

| | | <each group=""><br/>N=XXX</each> | |
|---|---|---|---|
| Visit | Status | n | % |
| INFORMED CONSENT | Completed | | |
| RANDOMIZATION | Completed | | |
| <each visit=""></each> | Attended | | |
| | Not attended yet | | |
| | Permanent discontinuation prior to this visit | | |
| | Not attended | | |
| CONCLUSION | Completed | | |

#### <each group>:

RSV-Ld = Low dose ChAd155-RSV vaccine (5 x 109 vp)

RSV-Md = Middle dose ChAd155-RSV vaccine (1.5 x 10<sup>10</sup> vp)

RSV-Hd = High dose ChAd155-RSV vaccine (5 x 10<sup>10</sup> vp)

Placebo-Ld = Non-active control (0.5 ml)

Placebo-Md = Non-active control (0.15 ml)

Placebo-Hd = Non-active control (0.5 ml)

N = Number of subjects in each group or in total

Conclusion = date of last visit or withdrawal

Template 4 Number of subjects enrolled into the study as well as the number of subjects excluded from the PPS analysis of immunogenicity at Day X with reasons for exclusion

| | | Tota | ıl | <eac< th=""><th>ch group&gt;</th></eac<> | ch group> |
|---|---|---|---|---|---|
| Title | Total <each< th=""><th>s</th></each<> | s | | | |
| Enrolled Set | | | | | |
| Invalid informed consent or fraudulent data (code 900) | | | | | |
| Study vaccine dose not administered but subject number allocated (code 1030) | | | | | |
| Exposed set | | | | | |
| <reason &="" code="" elimination="" for=""></reason> | | | | | |
| <reason &="" code="" elimination="" for=""></reason> | | | | | |
| PPS for analysis of immunogenicity at Day X | | | | | |

#### <each group>:

RSV-Ld = Low dose ChAd155-RSV vaccine (5 x 109 vp)

RSV-Md = Middle dose ChAd155-RSV vaccine (1.5 x 10<sup>10</sup> vp)

RSV-Hd = High dose ChAd155-RSV vaccine (5 x  $10^{10}$  vp)

Placebo-Ld = Non-active control (0.5 ml)

Placebo-Md = Non-active control (0.15 ml)

Placebo-Hd = Non-active control (0.5 ml)

Note: Subjects may have more than one elimination code assigned

n = number of subjects with the elimination code assigned excluding subjects who have been assigned a lower elimination code number

s = number of subjects with the elimination code assigned

% = percentage of subjects in the considered PPS relative to the Exposed set

#### Template 5 Summary of demographic characteristics <Exposed set>

| | <each group=""> N=XXXX</each> | | <each group=""><br/>N=XXXX</each> | | | otal<br>(XXX |
|---|---|---|---|---|---|---|
| | Value or n | % | Value or n | % | Value or n | % |
| Age in months at <timepoint></timepoint> | | | | | | |
| N with data | XXX | | XXX | | XXX | |
| Mean | XXX.X | | XXX.X | | XXX.X | |
| SD | XXX.X | | XXX.X | | XXX.X | |
| Median | xxx.x | | XXX.X | | XXX.X | |
| Minimum | XXX | | XXX | | XXX | |
| Maximum | XXX | | XXX | | XXX | |
| Gender | | | | | | |
| <each gender=""></each> | XXX | XX.X | XXX | XX.X | xxx | XX.X |
| | XXX | XX.X | XXX | XX.X | XXX | XX.X |
| Ethnicity | | | | | | |
| <each ethnicity=""></each> | xxx | XX.X | XXX | XX.X | XXX | XX.X |
| | xxx | XX.X | XXX | XX.X | XXX | XX.X |
| Geographic Ancestry | | | | | | |
| <each ancestry="" geographic=""></each> | XXX | XX.X | XXX | XX.X | XXX | XX.X |
| | XXX | XX.X | XXX | XX.X | XXX | XX.X |
| Country | | | | | | |
| <each country=""></each> | xxx | XX.X | XXX | XX.X | xxx | XX.X |
| | xxx | XX.X | XXX | XX.X | xxx | XX.X |

#### <each group>:

RSV-Ld = Low dose ChAd155-RSV vaccine (5 x 109 vp)

RSV-Md = Middle dose ChAd155-RSV vaccine (1.5 x 10<sup>10</sup> vp)

RSV-Hd = High dose ChAd155-RSV vaccine (5 x 10<sup>10</sup> vp)

Placebo-Ld = Non-active control (0.5 ml)

Placebo-Md = Non-active control (0.15 ml)

Placebo-Hd = Non-active control (0.5 ml)

N = total number of subjects

n/% = number / percentage of subjects in a given category

Value = value of the considered parameter

N with data = number of subjects with documentation of the corresponding data

SD = standard deviation

#### Template 6 Summary of vital signs characteristics <Exposed set>

| | | | <each group=""><br/>N =</each> | Total<br>N = |
|---|---|---|---|---|
| Visit | Characteristics | Parameters | Value | Value |
| <each visit=""></each> | Height (Cm) | N with data | | |
| | | Mean | | |
| | | SD | | |
| | | Median | | |
| | | Minimum | | |
| | | Maximum | | |
| | Weight (Kg) | N with data | | |
| | | Mean | | |
| | | SD | | |
| | | Median | | |
| | | Minimum | | |
| | | Maximum | | |
| | Heart rate (Beats per minute) | N with data | | |
| | | Mean | | |
| | | SD | | |
| | | Median | | |
| | | Minimum | | |
| | | Maximum | | |
| | Respiratory rate (Breadth per minute) | N with data | | |
| | | Mean | | |
| | | SD | | |
| | | Median | | |
| | | Minimum | | |
| | | Maximum | | |
| | Temperature/(Axillary) (°C) | N with data | | |
| | | Mean | | |
| | | SD | | |
| | | Median | | |
| | | Minimum | | |
| | | Maximum | | |

#### <each group>:

RSV-Ld = Low dose ChAd155-RSV vaccine (5 x 109 vp)

RSV-Md = Middle dose ChAd155-RSV vaccine (1.5 x 10<sup>10</sup> vp)

RSV-Hd = High dose ChAd155-RSV vaccine (5  $\times$  10<sup>10</sup> vp)

Placebo-Ld = Non-active control (0.5 ml)

Placebo-Md = Non-active control (0.15 ml)

Placebo-Hd = Non-active control (0.5 ml)

N = total number of subjects

N with data = number of subjects with documentation of the corresponding data

Value = value of the considered parameter

SD = standard deviation

#### Template 7 Distribution of weight for age Z-score (WAZ) at vaccination <Exposed Set>

| | | | Each group<br>N = | | |
|---|---|---|---|---|---|
| Visit | Characteristics | n | % | n | % |
| Day 1 | Normal (-1 < WAZ < 0) | | | | |
| | Mildly underweight (-2 <waz<-1)< td=""><td></td><td></td><td></td><td></td></waz<-1)<> | | | | |
| | Moderately underweight (-3 <waz<-2)< td=""><td></td><td></td><td></td><td></td></waz<-2)<> | | | | |
| | Severely underweight (WAZ<-3) | | | | |
| Day 366 | Normal (-1 < WAZ < 0) | | | | |
| | Mildly underweight (-2 <waz<-1)< td=""><td></td><td></td><td></td><td></td></waz<-1)<> | | | | |
| | Moderately underweight (-3 <waz<-2)< td=""><td></td><td></td><td></td><td></td></waz<-2)<> | | | | |
| | Severely underweight (WAZ<-3) | | | | |

<group>

RSV-Ld = Low dose ChAd155-RSV vaccine (5 x 109 vp)

RSV-Md = Middle dose ChAd155-RSV vaccine (1.5 x 10<sup>10</sup> vp)

RSV-Hd = High dose ChAd155-RSV vaccine (5 x  $10^{10}$  vp)

Placebo-Ld = Non-active control (0.5 ml)

Placebo-Md = Non-active control (0.15 ml)

Placebo-Hd = Non-active control (0.5 ml)

N = Total number of subjects

n = number of subjects in each category

% = n / Number of subjects with available results x 100

For weight for age Z score calculation of each subject, median = XX and SD = YY

Template 8 Distribution of height for age Z-score (HAZ) at vaccination <Exposed Set>

| | | Each group<br>N = | | Total<br>N = | |
|---|---|---|---|---|---|
| Visit | Characteristics | n | % | n | % |
| Day 1 | Normal (-1 < HAZ < 0 ) | | | | |
| | Mildly stunted (-2 <haz<-1)< td=""><td></td><td></td><td></td><td></td></haz<-1)<> | | | | |
| | Moderately stunted (-3 <haz<-2)< td=""><td></td><td></td><td></td><td></td></haz<-2)<> | | | | |
| | Severely stunted (HAZ<-3) | | | | |
| Day 366 | Normal (-1 < HAZ < 0 ) | | | | |
| | Mildly stunted (-2 <haz<-1)< td=""><td></td><td></td><td></td><td></td></haz<-1)<> | | | | |
| | Moderately stunted (-3 <haz<-2)< td=""><td></td><td></td><td></td><td></td></haz<-2)<> | | | | |
| | Severely stunted (HAZ<-3) | | | | |

<group>

RSV-Ld = Low dose ChAd155-RSV vaccine (5 x 109 vp)

RSV-Md = Middle dose ChAd155-RSV vaccine (1.5 x 10<sup>10</sup> vp)

RSV-Hd = High dose ChAd155-RSV vaccine (5 x  $10^{10}$  vp)

Placebo-Ld = Non-active control (0.5 ml)

Placebo-Md = Non-active control (0.15 ml)

Placebo-Hd = Non-active control (0.5 ml)

N = Total number of subjects

n = number of subjects in each category

% = n / Number of subjects with available results x 100

For height for age Z score calculation of each subject, median = XX and SD = YY

### Template 9 Deviations from specifications for age and intervals between study visits up to Day X <Exposed Set>

| | | Age | SCR-<br>Dose:1 | Dose:1-<br>VISIT3<br>(D4) | Dose:1-<br>VISIT4<br>(D8) | Dose:1-<br>Dose:2 | Dose:2-<br>VISIT7<br>(D34) | Dose:2-<br>VISIT8<br>(D38) | Dose:2-<br>VISIT9<br>(D61) | Dose:1-<br>VISIT10<br>(D366) | Dose:1-<br>VISIT11<br>(D731) |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Group | | Protocol | Protocol | Protocol | Protocol | Protocol | Protocol | Protocol | Protocol | Protocol | Protocol |
| | | from 12 | from 1 to | from 3 to | from 7 to | from 23 | from 3 to | from 7 to | from 28 to | from 335 | from 700 |
| | | to 23 | 30 days | 4 days | 10 days | to 36 | 4 days | 10 days | 35 days | to 395 | to 760 |
| | | months | | | | days | - | | | days | days |
| <each< td=""><td>N</td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td></each<> | N | | | | | | | | | | |
| group> | | | | | | | | | | | |
| | n | | | | | | | | | | |
| | % | | | | | | | | | | |
| | range | | | | | | | | | | |

#### <each group (pooled groups)>:

RSV-Ld = Low dose ChAd155-RSV vaccine (5 x 109 vp)

RSV-Md = Middle dose ChAd155-RSV vaccine (1.5 x 10<sup>10</sup> vp)

RSV-Hd = High dose ChAd155-RSV vaccine (5 x  $10^{10}$  vp)

Placebo-Ld = Non-active control (0.5 ml)

Placebo-Md = Non-active control (0.15 ml)

Placebo-Hd = Non-active control (0.5 ml)

N = total number of subjects with available results

n/% = number / percentage of subjects with results outside of the interval

range = minimum-maximum for age and intervals

Please note - On Day 3 and Day 33, a visit may take place at the investigators clinical facility or the investigator/clinical staff may call the subjects' parent(s)/LAR(s), as appropriate to the circumstances in the judgment of the investigator

#### **Template 10 Study Population**

| | <each group=""></each> | <each group=""> N=XXXX</each> | Total<br>N=XXXX |
|---|---|---|---|
| Number of subjects | | | |
| Planned, N | XXX | XXX | XXX |
| Randomised, N <cohort name=""></cohort> | XXX | XXX | xxx |
| Completed, n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| <unknown></unknown> | XXX | XXX | XXX |
| Demographics | | | |
| N <cohort name=""></cohort> | XXX | XXX | XXX |
| Females:Males | XXX:XXX | XXX:XXX | XXX:XXX |
| Mean Age, <unit> (SD)</unit> | xxx.x (xxx.x) | xxx.x (xxx.x) | xxx.x (xxx.x) |
| Median Age, <unit> (minimum, maximum)</unit> | xxx (xxx,xxx) | xxx (xxx,xxx) | xxx (xxx,xxx) |
| <most category="" frequent="" of="" race=""></most> | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| <second category="" frequent="" most="" of="" race=""></second> | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| <third category="" frequent="" most="" of="" race=""></third> | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |

#### <each group>:

RSV-Ld = Low dose ChAd155-RSV vaccine (5 x 109 vp)

RSV-Md = Middle dose ChAd155-RSV vaccine (1.5 x 10<sup>10</sup> vp)

RSV-Hd = High dose ChAd155-RSV vaccine (5 x 10<sup>10</sup> vp)

Placebo-Ld = Non-active control (0.5 ml)

Placebo-Md = Non-active control (0.15 ml)

Placebo-Hd = Non-active control (0.5 ml)

N = Total number of subjects

SD = Standard deviation

#### Template 11 Number of enrolled subjects by country

| | <each group=""><br/>N =</each> | Total<br>N = |
|-----------------|--------------------------------|--------------|
| Characteristics | n | n |
| Country | | |

#### <each group>:

RSV-Ld = Low dose ChAd155-RSV vaccine (5 x 109 vp)

RSV-Md = Middle dose ChAd155-RSV vaccine (1.5 x 10<sup>10</sup> vp)

RSV-Hd = High dose ChAd155-RSV vaccine (5 x 10<sup>10</sup> vp)

Placebo-Ld = Non-active control (0.5 ml)

Placebo-Md = Non-active control (0.15 ml)

Placebo-Hd = Non-active control (0.5 ml)

N = Number of enrolled subjects

n= number of enrolled subjects included in each group or in total for a given country or for all countries

#### Template 12 Number of enrolled subjects by age category

| | | <each group=""><br/>N =</each> | Total<br>N = |
|---|---|---|---|
| Characteristics | Categories | n | n |
| Age category | 1=Infants and toddlers (28 days-23 month) | | |
| | Missing | | |

#### <each group>:

RSV-Ld = Low dose ChAd155-RSV vaccine (5 x 109 vp)

RSV-Md = Middle dose ChAd155-RSV vaccine  $(1.5 \times 10^{10} \text{ vp})$ 

RSV-Hd = High dose ChAd155-RSV vaccine (5 x 10<sup>10</sup> vp)

Placebo-Ld = Non-active control (0.5 ml)

Placebo-Md = Non-active control (0.15 ml)

Placebo-Hd = Non-active control (0.5 ml)

N = Number of enrolled subjects

n= number of enrolled subjects included in each group or in total for a given age category or for all age categories Missing = age at dose 1 unknown

#### Template 13 Minimum and maximum activity dates <Exposed set>

| | | <each group=""></each> | <each group=""></each> | Overall |
|---|---|---|---|---|
| Visit Description | Parameter | Date | Date | Date |
| <each consent="" inform=""></each> | Minimum | | | |
| | Maximum | | | |
| [Randomisation] | Minimum | | | |
| | Maximum | | | |
| <each visit=""></each> | Minimum | | | |
| | Maximum | | | |

#### <each group>:

RSV-Ld = Low dose ChAd155-RSV vaccine (5 x 109 vp)

RSV-Md = Middle dose ChAd155-RSV vaccine (1.5 x 10<sup>10</sup> vp)

RSV-Hd = High dose ChAd155-RSV vaccine (5 x 10<sup>10</sup> vp)

Placebo-Ld = Non-active control (0.5 ml)

Placebo-Md = Non-active control (0.15 ml)

Placebo-Hd = Non-active control (0.5 ml)

#### Template 14 Exposure to study vaccines < Exposed Set>

| | | ach group><br>N=XXXX | | ach group><br>N=XXXX | N | Total<br>N=XXXX |
|---|---|---|---|---|---|---|
| Number of subjects receiving | n | % | n | % | n | % |
| Exactly 1 Dose | | | | | | |
| Exactly 2 Doses | | | | | | |
| At least 1 Dose | | | | | | |
| Total number of doses administered during the study | | | | | | |

RSV-Ld = Low dose ChAd155-RSV vaccine (5 x 109 vp)

RSV-Md = Middle dose ChAd155-RSV vaccine (1.5 x 10<sup>10</sup> vp)

RSV-Hd = High dose ChAd155-RSV vaccine (5 x  $10^{10}$  vp)

Placebo-Ld = Non-active control (0.5 ml)

Placebo-Md = Non-active control (0.15 ml)

Placebo-Hd = Non-active control (0.5 ml)

N = number of subjects in each group or in total included in the considered cohort

n = number of subjects/doses in the given category

% = percentage of subjects in the given category

Template 15 Compliance in completing solicited symptoms information <Exposed Set>

| | | | <each gro<="" th=""><th>oup&gt;</th><th colspan="5"><each group=""></each></th></each> | oup> | <each group=""></each> | | |
|---|---|---|---|---|---|---|---|
| DOSE | Symptom information | N | n | Compliance (%) | N | n | Compliance (%) |
| DOSE <each dose="" number=""></each> | General SS | | | | | | |
| | Local SS | | | | | | |
| TOTAL | General SS<br>Local SS | | | | | | |

RSV-Ld = Low dose ChAd155-RSV vaccine (5 x 109 vp)

RSV-Md = Middle dose ChAd155-RSV vaccine  $(1.5 \times 10^{10} \text{ vp})$ 

RSV-Hd = High dose ChAd155-RSV vaccine (5 x 10<sup>10</sup> vp)

Placebo-Ld = Non-active control (0.5 ml)

Placebo-Md = Non-active control (0.15 ml)

Placebo-Hd = Non-active control (0.5 ml)

N=Number of administered doses

n = number of doses with SS returned

General SS = Symptom screens used for the collection of general solicited AEs

Local SS = Symptom screens used for the collection of local solicited AEs

Compliance (%) =  $(n / N) \times 100$ 

204838 (RSV PED-002) Statistical Analysis Plan Final

## Template 16 Incidence and nature of symptoms (solicited and unsolicited) reported during the 7-day post-vaccination period (Days 1-7) following each dose and overall <Exposed Set>

| | | <e< th=""><th>ac</th><th>h gr</th><th>oup&gt;</th><th></th><th><e< th=""><th>acl</th><th>h gr</th><th>oup&gt;</th><th></th><th></th><th>Loc</th><th>cal s</th><th>ympto</th><th>ms</th></e<></th></e<> | ac | h gr | oup> | | <e< th=""><th>acl</th><th>h gr</th><th>oup&gt;</th><th></th><th></th><th>Loc</th><th>cal s</th><th>ympto</th><th>ms</th></e<> | acl | h gr | oup> | | | Loc | cal s | ympto | ms |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | % CI | | | | 95 | % CI | | | | 95 | % CI |
| Dose | Symptoms | N | n | % | LL | UL | N | n | % | LL | UL | N | n | % | LL | UL |
| Dose 1 | Any symptom | | | | | | | | | | | | | | | |
| | General symptoms | | | | | | | | | | | | | | | |
| | Local symptoms | | | | | | | | | | | | | | | |
| Dose 2 | Any symptom | | | | | | | | | | | | | | | |
| | General symptoms | | | | | | | | | | | | | | | |
| | Local symptoms | | | | | | | | | | | | | | | |
| Overall/dose | Any symptom | | | | | | | | | | | | | | | |
| | General symptoms | | | | | | | | | | | | | | | |
| | Local symptoms | | | | | | | | | | | | | | | |
| Overall/subject | Any symptom | | | | | | | | | | | | | | | |
| - | General symptoms | | | | | | | | | | | | | | | |
| | Local symptoms | | | | | | | | | | | | | | | |

RSV-Ld = Low dose ChAd155-RSV vaccine (5 x 109 vp)

RSV-Md = Middle dose ChAd155-RSV vaccine (1.5 x 10<sup>10</sup> vp)

RSV-Hd = High dose ChAd155-RSV vaccine (5 x 10<sup>10</sup> vp)

Placebo-Ld = Non-active control (0.5 ml)

Placebo-Md = Non-active control (0.15 ml)

Placebo-Hd = Non-active control (0.5 ml)

For each dose:

N = number of subjects with the corresponding documented dose

n/% = number/percentage of subjects presenting at least one type of symptom following the corresponding dose For overall/dose:

N = number of documented dose

n/% = number/percentage of doses followed by at least one type of symptom

For overall/subject:

N = number of documented dose

n/% = number/percentage of subjects presenting at least one type of symptom

95% CI = exact 95% confidence interval, LL = Lower Limit, UL = Upper Limit

204838 (RSV PED-002) Statistical Analysis Plan Final

## Template 17 Incidence of solicited local symptoms reported during the 7-day (Days 1-7) post-vaccination period following each dose and overall <Exposed Set>

| | | | | <each group=""></each> | | | |
|---|---|---|---|---|---|---|---|
| | | | | | | 9: | 5 % CI |
| Dose | Symptom | Туре | N | n | % | LL | UL |
| DOSE 1 | Pain | All | | | | | |
| | | ≥ Grade 2 | | | | | |
| | | Grade 3 | | | | | |
| | | Medical advice | | | | | |
| | Redness (mm) | All | | | | | |
| | | ≥ 5 | | | | | |
| | | >20 | | | | | |
| | | Medical advice | | | | | |
| | Swelling (mm) | All | | | | | |
| | | ≥ 5 | | | | | |
| | | >20 | | | | | |
| | | Medical advice | | | | | |
| DOSE 2 | Pain | | | | | | |
| | Redness (mm) | | | | | | |
| | Swelling (mm) | | | | | | |
| OVERALL/DOSE | Pain | | | | | | |
| | Redness (mm) | | | | | | |
| | Swelling (mm) | | | | | | |
| OVERALL/SUBJECT | Pain | | | | | | |
| | Redness (mm) | | | | | | |
| | Swelling (mm) | | | | | | |

#### <each group>:

RSV-Ld = Low dose ChAd155-RSV vaccine (5 x 109 vp)

RSV-Md = Middle dose ChAd155-RSV vaccine (1.5 x 10<sup>10</sup> vp)

RSV-Hd = High dose ChAd155-RSV vaccine (5 x 10<sup>10</sup> vp)

Placebo-Ld = Non-active control (0.5 ml)

Placebo-Md = Non-active control (0.15 ml)

Placebo-Hd = Non-active control (0.5 ml)

For each dose:

N = number of subjects with the corresponding documented dose

n/% = number/percentage of subjects reporting the type of symptom at least once following the corresponding dose For Overall/dose:

N = number of documented dose

n/% = number/percentage of doses followed by at least one type of symptom

For Overall/subject:

N = number of subjects with at least one documented dose

n/% = number/percentage of subjects reporting the type of symptom at least once

95%CI= Exact 95% confidence interval; LL = lower limit, UL = upper limit

The maximum intensity of local injection site redness/swelling was coded as follows:

1: > 0.1 mm to < 5 mm

 $2: \geq 5 \text{ mm to} \leq 20 \text{ mm}$ 

3: > 20 mm

204838 (RSV PED-002) Statistical Analysis Plan Final

# Template 18 Incidence of solicited local symptoms reported during the 7-day (Days 1-7) post-vaccination period following each dose and overall by maximum grading <Exposed Set>

| | | | | | <eac< th=""><th colspan="4">ch group&gt;</th></eac<> | ch group> | |
|---|---|---|---|---|---|---|---|
| | Γ- | I | | | 95 % C | | |
| Oose | Symptom | Туре | N | n | % | LL | UL |
| OSE 1 | Pain | All | | | | | |
| | | Grade 1 | | | | | |
| | | Grade 2 | | | | | |
| | | Grade 3 | | | | | |
| | | Medical advice | | | | | |
| | Redness (mm) | All | | | | | |
| | | ≥0.1 - <5.0 | | | | | |
| | | ≥5.0 - ≤20.0 | | | | | |
| | | >20 | | | | | |
| | | Medical advice | | | | | |
| | Swelling (mm) | All | | | | | |
| | | ≥0.1 - <5.0 | | | | | |
| | | ≥5.0 - ≤20.0 | | | | | |
| | | >20 | | | | | |
| | | Medical advice | | | | | |
| OOSE 2 | Pain | All | | | | | |
| | | Grade 1 | | | | | |
| | | Grade 2 | | | | | |
| | | Grade 3 | | | | | |
| | | Medical advice | | | | | |
| | Redness (mm) | All | | | | | |
| | redices (iiiii) | ≥0.1 - <5.0 | | | | | |
| | | ≥5.0 - ≤20.0 | | | | | |
| | | >20 | | | | | |
| | | Medical advice | | | | | |
| | Constling (mass) | | | | | | |
| | Swelling (mm) | All | | | | | |
| | | ≥0.1 - <5.0 | | | | | |
| | | ≥5.0 - ≤20.0 | | | | | |
| | | >20 | | | | | |
| N/EDALL/DOOF | D : | Medical advice | | | | | |
| OVERALL/DOSE | Pain | All | | | | | |
| | | Grade 1 | | | | | |
| | | Grade 2 | | | | | |
| | | Grade 3 | | | | | |
| | | Medical advice | | | | | |
| | Redness (mm) | All | | | | | |
| | | ≥0.1 - <5.0 | | | | | |
| | | ≥5.0 - ≤20.0 | | | | | |
| | | >20 | | | | | |
| | | Medical advice | | | | | |
| | Swelling (mm) | All | | | | | |
| | | ≥0.1 - <5.0 | | | | $\perp$ | |
| | | ≥5.0 - ≤20.0 | | | | $\perp$ | |
| | | >20 | | | | | |
| | | Medical advice | | | | | |

204838 (RSV PED-002) Statistical Analysis Plan Final

| | | | | | <eac< th=""><th>ch gro</th><th>up&gt;</th></eac<> | ch gro | up> |
|---|---|---|---|---|---|---|---|
| | | | | | | | 95 % CI |
| Dose | Symptom | Туре | N | n | % | LL | UL |
| OVERALL/SUBJECT | Pain | All | | | | | |
| | | Grade 1 | | | | | |
| | | Grade 2 | | | | | |
| | | Grade 3 | | | | | |
| | | Medical advice | | | | | |
| | Redness (mm) | All | | | | | |
| | () | ≥0.1 - <5.0 | | | | | |
| | | ≥5.0 - ≤20.0 | | | | | |
| | | >20 | | | | | |
| | | Medical advice | | | | | |
| | Swelling (mm) | All | | | | | |
| | | ≥0.1 - <5.0 | | | | | |
| | | ≥5.0 - ≤20.0 | | | | | |
| | | >20 | | | | | |
| | | Medical advice | | | | | |

RSV-Ld = Low dose ChAd155-RSV vaccine (5 x 109 vp)

RSV-Md = Middle dose ChAd155-RSV vaccine (1.5 x 10<sup>10</sup> vp)

RSV-Hd = High dose ChAd155-RSV vaccine (5 x 10<sup>10</sup> vp)

Placebo-Ld = Non-active control (0.5 ml)

Placebo-Md = Non-active control (0.15 ml)

Placebo-Hd = Non-active control (0.5 ml)

For each dose:

N = number of subjects with the corresponding documented dose

n/% = number/percentage of subjects reporting the type of symptoms as maximum intensity during the follow-up period

For Overall/dose:

N = number of documented dose

n/% = number/percentage of doses followed by the type of symptom as maximum intensity during the follow-up period For Overall/subject:

N = number of documented dose

n/% = number/percentage of subjects reporting the type of symptom as maximum intensity during the follow-up period CI = Exact 95% confidence interval; LL = lower limit, UL = upper limit

The maximum intensity of local injection site redness/swelling was coded as follows:

- 1: > 0.1 mm to < 5 mm
- $2: \geq 5 \text{ mm to} \leq 20 \text{ mm}$
- 3: > 20 mm

204838 (RSV PED-002) Statistical Analysis Plan Final

## Template 19 Incidence of solicited general symptoms reported during the 7-day (Days 1-7) post-vaccination period following each dose and overall <Exposed Set>

| | | | | | <each gr<="" th=""><th></th><th></th></each> | | |
|---|---|---|---|---|---|---|---|
| | | | | | le: | | 5 % CI |
| Oose | Symptom | Туре | N | n | % | LL | UL |
| OSE 1 | Drowsiness | All | | | | | |
| | | ≥ Grade 2 | | | | | |
| | | Grade 3 | | | | | |
| | | Related | | | | | |
| | | ≥ Grade 2*Related | | | | | |
| | | Grade 3*Related | | | | | |
| | | Medical advice | | | | | |
| | Irritability/Fussiness | All | | | | | |
| | | ≥ Grade 2 | | | | | |
| | | Grade 3 | | | | | |
| | | Related | | | | | |
| | | ≥ Grade 2*Related | | | | | |
| | | Grade 3*Related | | | | | |
| | | Medical advice | | | | | |
| | Loss of appetite | All | | | | | |
| | zooo o. apponto | ≥ Grade 2 | | | | | |
| | | Grade 3 | | | | | |
| | | Related | | | | | |
| | | ≥ Grade 2*Related | | | | | |
| | | Grade 3*Related | | | | | |
| | | Medical advice | | | | | |
| | Fever (Axillary) (°C) | All (≥37.5) | | | | | |
| | rever (Axillary) ( C) | >37.5 | | | | | |
| | | >38.0 | | | | | |
| | | >38.5 | | | | | |
| | | >39.0 | | | | | |
| | | >39.5 | | | | | |
| | | Related | | | | | |
| | | >38.5*Related | | | | | |
| | | >39.5*Related | | | | | |
| 2005.0 | | Medical advice | | | | | |
| OOSE 2 | Drowsiness | | | | | | |
| | Irritability/Fussiness | | | | | | |
| | Loss of appetite | | | | | | |
| | Fever (Axillary) (°C) | | | | | | |
| OVERALL/DOSE | Drowsiness | | | | | | |
| | Irritability/Fussiness | | | | | | |
| | Loss of appetite | | | | | | |
| | Fever (Axillary) (°C) | | | | | | |
| OVERALL/SUBJECT | Drowsiness | | | | | | |
| | Irritability/Fussiness | | | | | | |
| | Loss of appetite | | | | | | |
| | Fever (Axillary) (°C) | | | | | | |

#### <each group>:

RSV-Ld = Low dose ChAd155-RSV vaccine (5 x 109 vp)

RSV-Md = Middle dose ChAd155-RSV vaccine (1.5 x 10<sup>10</sup> vp)

RSV-Hd = High dose ChAd155-RSV vaccine ( $5 \times 10^{10} \text{ vp}$ )

Placebo-Ld = Non-active control (0.5 ml)

204838 (RSV PED-002) Statistical Analysis Plan Final

Placebo-Md = Non-active control (0.15 ml)

Placebo-Hd = Non-active control (0.5 ml)

For each dose:

N = number of subjects with the corresponding documented dose

n/% = number/percentage of subjects reporting the symptom at least once following the corresponding dose For Overall/dose:

N = number of documented dose

n/% = number/percentage of doses followed by at least one type of symptom

For Overall/subject:

N = number of subjects with at least one documented dose

n/% = number/percentage of subjects reporting the type of symptom at least once

95%CI= Exact 95% confidence interval; LL = lower limit, UL = upper limit

Temperatures were coded as follows:

1: ≥ 37.5 °C to ≤ 38.5 °C

 $2: > 38.5 \,^{\circ}\text{C} \text{ to} \le 39.5 \,^{\circ}\text{C}$ 

2. > 30.5 °C to ≤ 39. 3: > 39.5°C

204838 (RSV PED-002) Statistical Analysis Plan Final

# Template 20 Incidence of solicited general symptoms reported during the 7-day (Days 1-7) post-vaccination period following each dose and overall by maximum grading <Exposed Set>

| | | | | ach | ch group<br>95 % | | |
|---|---|---|---|---|---|---|---|
| Dose | Symptom | Туре | N | n | 0/_ | LL | UL |
| OOSE 1 | Drowsiness | All | IN | " | /0 | LL | UL |
| JOSE 1 | Diowsiness | Grade 1 | | | | | - |
| | | Grade 2 | | | | | - |
| | | Grade 3 | | | | | - |
| | | Related | | | | | _ |
| | | | | | | | - |
| | | Grade 2 Related | | | | | _ |
| | | Grade 3 Related | | | | | _ |
| | Indiah III. / Francisco | Medical advice | | | | | _ |
| | Irritability / Fussiness | All | | | | | - |
| | | Grade 1 | | | | | _ |
| | | Grade 2 | | | | | |
| | | Grade 3 | | | | | |
| | | Related | | | | | |
| | | Grade 2 Related | | | | | |
| | | Grade 3 Related | | | | | |
| | | Medical advice | | | | | |
| | Loss Of Appetite | All | | | | | |
| | | Grade 1 | | | | | |
| | | Grade 2 | | | | | |
| | | Grade 3 | | | | | |
| | | Related | | | | | |
| | | Grade 2 Related | | | | | |
| | | Grade 3 Related | | | | | - |
| | | Medical advice | | | | | |
| | Temperature/(Axillary) (°C) | All | | | | | + |
| | romporatoro/(romary) ( o) | ≥37.5 - ≤38.5 | | | | | + |
| | | >38.5 - ≤39.5 | | | | | + |
| | | >39.5 | | | | | + |
| | | Related | | | | | - |
| | | >38.5 - ≤39.5*Related | | | | | - |
| | | >39.5*Related | | | | | - |
| | | Medical advice | | | | | - |
| OCE 1 | Drawainasa | All | | | | | - |
| OOSE 2 | Drowsiness | | | | | | - |
| | | Grade 1 | | | | | - |
| | | Grade 2 | | | | | - |
| | | Grade 3 | | | | | - |
| | | Related | | | | | _ |
| | | Grade 2 Related | | | | | - |
| | | Grade 3 Related | | | | | |
| | | Medical advice | | | | | |
| | Irritability / Fussiness | All | | | | | |
| | | Grade 1 | | | | | |
| | | Grade 2 | | | | | |
| | | Grade 3 | | | | | |
| | | Related | | | | | |
| | | Grade 2 Related | | | | | |
| | | Grade 3 Related | | | | | |
| | | Medical advice | | | | | 1 |

204838 (RSV PED-002) Statistical Analysis Plan Final

| | | | | E | acl | n gro | up |
|---|---|---|---|---|---|---|---|
| | | | | | | 95 | % CI |
| Dose | Symptom | Туре | N | n | % | LL | UL |
| | Loss Of Appetite | All | | | | | |
| | | Grade 1 | | | | | |
| | | Grade 2 | | | | | |
| | | Grade 3 | | | | | |
| | | Related | | | | | |
| | | Grade 2 Related | | | | | |
| | | Grade 3 Related | | | | | |
| | | Medical advice | | | | | |
| | Temperature/(Axillary) (°C) | All | | | | | |
| | | ≥37.5 - ≤38.5 | | | | | |
| | | >38.5 - ≤39.5 | | | | | |
| | | >39.5 | | | | | |
| | | Related | | | | | |
| | | >38.5 - ≤39.5*Related | | | | | |
| | | >39.5*Related | | | | | 1 |
| | | Medical advice | | | | | |
| N/EDALL/DOSE | Droweinose | All | | | | 1 | |
| OVERALL/DOSE | Drowsiness | | | - | | 1 | |
| | | Grade 1 | | | | 1 | |
| | | Grade 2 | | | | | |
| | | Grade 3 | | | | | |
| | | Related | | | | | |
| | | Grade 2 Related | | | | | |
| | | Grade 3 Related | | | | | |
| | | Medical advice | | | | | |
| | Irritability / Fussiness | All | | | | | |
| | initability / 1 d33inc33 | Grade 1 | | | | | |
| | | Grade 2 | | | | | |
| | | Grade 3 | | | | | |
| | | Related | | | | | |
| | | Grade 2 Related | | | | | |
| | | Grade 3 Related | | | | | |
| | | Medical advice | | | | | |
| | Loss Of Appetite | All | | | | | |
| | | Grade 1 | | | | | |
| | | Grade 2 | | | | | |
| | | Grade 3 | | | | | |
| | | Related | | | | | |
| | | Grade 2 Related | | | | | |
| | | Grade 3 Related | | | | | |
| | | Medical advice | | | | | |
| | Temperature/(Axillary) (°C) | All | | | | | |
| | . , , , , | ≥37.5 - ≤38.5 | | | | | |
| | | >38.5 - ≤39.5 | | | | | |
| | | >39.5 | | | | | |
| | | Related | | | | 1 | |
| | | | | - | | 1 | |
| | | >38.5 - ≤39.5*Related | | - | | 1 | |
| | | >39.5*Related | | | | 1 | |
| | | Medical advice | | | | | |
| OVERALL/SUBJECT | Drowsiness | All | | | L | | |
| | | Grade 1 | | | | 1 | |
| | | Grade 2 | | | | | |
| | | Grade 3 | | | | 1 | |
| | | Related | | <del> </del> | 1 | | 1 |

204838 (RSV PED-002) Statistical Analysis Plan Final

| | | | | E | acl | n gro | |
|---|---|---|---|---|---|---|---|
| | | | | | | 95 | % C |
| Dose | Symptom | Туре | N | n | % | LL | UL |
| | | Grade 2 Related | | | | | |
| | | Grade 3 Related | | | | | |
| | | Medical advice | | | | | |
| | Irritability / Fussiness | All | | | | | |
| | | Grade 1 | | | | | |
| | | Grade 2 | | | | | |
| | | Grade 3 | | | | | |
| | | Related | | | | | |
| | | Grade 2 Related | | | | | |
| | | Grade 3 Related | | | | | |
| | Loss Of Appetite | Medical advice | | | | | |
| | | All | | | | | |
| | | Grade 1 | | | | | |
| | | Grade 2 | | | | | |
| | | Grade 3 | | | | | |
| | | Related | | | | | |
| | | Grade 2 Related | | | | | |
| | | Grade 3 Related | | | | | |
| | | Medical advice | | | | | |
| | Temperature/(Axillary) (°C) | All | | | | | |
| | | ≥37.5 - ≤38.5 | | | | | |
| | | >38.5 - ≤39.5 | | | | | |
| | | >39.5 | | | | | |
| | | Related | | | | | |
| | | >38.5 - ≤39.5*Related | | | | | |
| | | >39.5*Related | | | | | |
| | | Medical advice | | | | | |

RSV-Ld = Low dose ChAd155-RSV vaccine (5 x 109 vp)

RSV-Md = Middle dose ChAd155-RSV vaccine (1.5 x 10<sup>10</sup> vp)

RSV-Hd = High dose ChAd155-RSV vaccine (5 x 10<sup>10</sup> vp)

Placebo-Ld = Non-active control (0.5 ml)

Placebo-Md = Non-active control (0.15 ml)

Placebo-Hd = Non-active control (0.5 ml)

For each dose:

N = number of subjects with the corresponding documented dose

n/% = number/percentage of subjects reporting the type of symptom as maximum intensity during the follow-up period For Overall/dose:

N = number of documented dose

n/% = number/percentage of doses followed by the type of symptoms as maximum intensity during the follow-up period For Overall/subject:

N = number of subjects with at least one documented dose

n/% = number/percentage of subjects reporting the type of symptoms as maximum intensity during the follow-up period 95%CI = Exact 95% confidence interval; LL = lower limit, UL = upper limit

Temperatures were coded as follows:

1: ≥ 37.5 °C to ≤ 38.5 °C

 $2: > 38.5 \,^{\circ}\text{C} \text{ to} \le 39.5 \,^{\circ}\text{C}$ 

3: > 39.5°C

Template 21 Maximum Temperature reported during the 7-day (Days 1-7) post-vaccination period – dose X <Exposed Set>

| | | E | | | Each group<br>N = | | | Total<br>N = | |
|---|---|---|---|---|---|---|---|---|---|
| | | | | 9 | 95% CI | | | 9: | 5% CI |
| Characteristics | Categories | n | % | LL | UL | n | % | LL | UL |
| Maximum temperature | No fever | | | | | | | | |
| | Unknown temperature | | | | | | | | |
| | [37.5-37.9] | | | | | | | | |
| | [38.0-38.4] | | | | | | | | |
| | [38.5-38.9] | | | | | | | | |
| | [39.0-39.4] | | | | | | | | |
| | [39.5-39.9] | | | | | | | | |
| | [40.0 | | | | | | | | |

N = number of subjects with documented dose

n/% = number/percentage of subjects in a given category

95%CI = Exact 95% confidence interval; LL = lower limit, UL = upper limit

Template 22 Percentage of subjects reporting the occurrence of unsolicited symptoms classified by MedDRA Primary System Organ Class and Preferred Term within the 30-day (Days 1-30) post-vaccination period <Exposed Set>

| | | | acł<br>I = | ı gr | oup |
|---|---|---|---|---|---|
| | | | | | 5%<br>CI |
| Gastrointestinal disorders (10017947) General disorders and administration site conditions (10018065) Inmune system disorders (10021428) | Preferred Term (CODE) | n | % | LL | UL |
| At least one symptom | | | | | |
| Gastrointestinal disorders (10017947) | Diarrhoea (10012735) | | | | |
| ,<br> | Teething (10043183) | | | | |
| | Vomiting (10047700) | | | | |
| General disorders and administration site conditions (10018065) | Pyrexia (10037660) | | | | |
| Immune system disorders (10021428) | Seasonal allergy (10048908) | | | | |
| Infections and infestations (10021881) | Conjunctivitis (10010741) | | | | |
| , , | Otitis media (10033078) | | | | |
| | Paronychia (10034016) | | | | |
| | Tonsillitis (10044008) | | | | |
| | Tonsillitis streptococcal (10044013) | | | | |
| | Viral upper respiratory tract infection (10047482) | | | | |
| Injury, poisoning and procedural complications (10022117) | Arthropod bite (10003399) | | | | |
| , , , , , | Face injury (10050392) | | | | |
| | Head injury (10019196) | | | | |
| Skin and subcutaneous tissue disorders (10040785) | Miliaria (10027627) | | | | |

RSV-Ld = Low dose ChAd155-RSV vaccine (5 x 109 vp)

RSV-Md = Middle dose ChAd155-RSV vaccine (1.5 x 10<sup>10</sup> vp)

RSV-Hd = High dose ChAd155-RSV vaccine (5 x  $10^{10}$  vp)

Placebo-Ld = Non-active control (0.5 ml)

Placebo-Md = Non-active control (0.15 ml)

Placebo-Hd = Non-active control (0.5 ml)

At least one symptom = at least one symptom experienced (regardless of the MedDRA Preferred Term)

N = number of subjects included in the considered cohort in each group

n/% = number/percentage of subjects reporting the symptom at least once

95% CI = exact 95% confidence interval; LL = Lower Limit, UL = Upper Limit

204838 (RSV PED-002) Statistical Analysis Plan Final

## Template 23 Number and percentage of subjects taking a concomitant medication during the 7- day (Days 1-7) post -vaccination period <Exposed Set>

| | | | | <each g<="" th=""><th>group&gt;</th><th></th></each> | group> | |
|---|---|---|---|---|---|---|
| | | | | | | 95% CI |
| Dose | Туре | N | n | % | LL | UL |
| DOSE 1 | Any | | | | | |
| | Any antipyretics | | | | | |
| | Prophylactic antipyretics | | | | | |
| DOSE 2 | Any | | | | | |
| | Any antipyretics | | | | | |
| | Prophylactic antipyretics | | | | | |
| OVERALL/DOSE | Any | | | | | |
| | Any antipyretics | | | | | |
| | Prophylactic antipyretics | | | | | |
| OVERALL/SUBJECT | Any | | | | | |
| | Any antipyretics | | | | | |
| | Prophylactic antipyretics | | | | | |

#### <each group>:

RSV-Ld = Low dose ChAd155-RSV vaccine (5 x 109 vp)

RSV-Md = Middle dose ChAd155-RSV vaccine (1.5 x 10<sup>10</sup> vp)

RSV-Hd = High dose ChAd155-RSV vaccine (5 x 10<sup>10</sup> vp)

Placebo-Ld = Non-active control (0.5 ml)

Placebo-Md = Non-active control (0.15 ml)

Placebo-Hd = Non-active control (0.5 ml)

For each dose:

N = total number of subjects with the corresponding administered dose

n/% = number/percentage of subjects took the specified type of concomitant medication at least once during the considered period

For Overall/dose:

N = number of administered doses

n/% = number/percentage of doses after which the specified type of concomitant medication was taken at least once during the considered period

For Overall/subject:

N = total number of subjects with at least one administered dose

n/% = number/percentage of subjects who took the specified type of concomitant medication at least once during the considered period

95%CI = Exact 95% confidence interval; LL = lower limit, UL = upper limit

### Template 24 Distribution of change from baseline in hematology and biochemistry with respect to normal laboratory ranges <Exposed Set>

| | | | | < | each | group > |
|---|---|---|---|---|---|---|
| Laboratory parameter | Timing | Range indicator at Baseline (SCR) | Range indicator at timing | N | n | % |
| Alanine Aminotransferase | PI(D2) | Unknown | Unknown | | | |
| | | | Below | | | |
| | | | Within | | | |
| | | | Above | | | |
| | | Below | Unknown | | | |
| | | Bel | | | | |
| | | | Within | | | |
| | | | Above | | | |
| | | Within | Unknown | | | |
| | | | Below | | | |
| | | | Within | | | |
| | | | Above | | | |
| | | Above | Unknown | | | |
| | | Belo | Below | | | |
| | | | Within | | | |
| | | | Above | | | |
| | PI (D8) | | | | | |
| | PI (D31) | | | | | |
| | PII (D32) | | | | | |
| | PII (D38) | | | | | |
| | PII (D61) | | | | | |
| | UNSCH1 | | | | | |
| | UNSCH2 | | | | | |
| Aspartate Aminotransferase | | | | | | |
| Creatinine | | | | | | |
| -<br>Hemoglobin | | | | | | |
| Leukocytes (White Blood Cells) | | | | | | |
| Neutrophil | | | | | | |
| Platelets | | | | | | |

#### <each group>:

RSV-Ld = Low dose ChAd155-RSV vaccine (5 x 109 vp)

RSV-Md = Middle dose ChAd155-RSV vaccine (1.5 x 10<sup>10</sup> vp)

RSV-Hd = High dose ChAd155-RSV vaccine (5 x  $10^{10}$  vp)

Placebo-Ld = Non-active control (0.5 ml)

Placebo-Md = Non-active control (0.15 ml)

Placebo-Hd = Non-active control (0.5 ml)

N = number of subjects with available results for the specified laboratory parameter and timing in a given baseline category

n/% = number/percentage of subjects in the specified category

Below = below the normal laboratory range defined for the specified laboratory parameter

Within = within the normal laboratory range defined for the specified laboratory parameter

Above = above the normal laboratory range defined for the specified laboratory parameter

SCR= Screening

PI (D2): Post-vaccination dose 1 at Day 2

PI (D8): Post-vaccination dose 1 at Day 8

PI (D31): Post-vaccination dose 1 at Day 31

PII (D32): Post-vaccination dose 2 at Day 32

PII (D38): Post-vaccination dose 2 at Day 38

PII (D61): Post-vaccination dose 2 at Day 61 UNSCH: Unscheduled visit for safety

Template 25 Summary of hematology and biochemistry results by maximum grade from VISIT X (DX) up to VISIT Y (DY) – post dose 1 of vaccination versus baseline <Exposed Set>

| | | | <each group=""></each> | | |
|---|---|---|---|---|---|
| Laboratory parameter | Baseline<br>(SCR) | Visit 2 to Visit X | N | n | % |
| Hemoglobin (decrease) | Unknown | Unknown | | | |
| | | Grade 0 | | | |
| | | Grade 1 | | | |
| | | Grade 2 | | | |
| | | Grade 3 | | | |
| | | Grade 4 | | | |
| | Grade 0 | | | | |
| | Grade 1 | | | | |
| | Grade 2 | | | | |
| | Total | | | | |
| Leukocytes (White Blood Cells) (decrease) | | | | | |
| Neutrophil (decrease) | | | | | |
| Platelets | | | | | |
| Alanine Aminotransferase | | | | | |
| Aspartate Aminotransferase | | | | | |
| Creatinine | | | | | |

#### <each group>:

RSV-Ld = Low dose ChAd155-RSV vaccine (5 x 109 vp)

RSV-Md = Middle dose ChAd155-RSV vaccine (1.5 x 1010 vp)

RSV-Hd = High dose ChAd155-RSV vaccine (5 x 1010 vp)

Placebo-Ld = Non-active control (0.5 ml)

Placebo-Md = Non-active control (0.15 ml)

Placebo-Hd = Non-active control (0.5 ml)

N = number of subjects with at least one available result for the specified laboratory parameter and follow-up period n/% = number/percentage of subjects reporting at least once the laboratory event when the maximum grading over the follow-up period is considered

SCR=Screening

204838 (RSV PED-002) Statistical Analysis Plan Final

### Template 26 Descriptive statistics table on eosinophils, basophils, and monocytes counts for subjects <Exposed Set>

| | | | Each Group<br>N= | | |
|-------------|-----------|-----------|------------------|----|--------|
| | | | | | 95% CI |
| Parameters | Timing | Parameter | Value | LL | UL |
| Eosinophils | SCR | n | | | |
| • | | Mean | | | |
| | | 95% CI | | | |
| | | Q1 | | | |
| | | Median | | | |
| | | Q3 | | | |
| | | Min/Max | | | |
| | PI(D2) | | | | |
| | PI (D8) | | | | |
| | PI (D31) | | | | |
| | PII (D32) | | | | |
| | PII (D38) | | | | |
| Basophils | | | | | |
| Monocytes | | | | | |

RSV-Ld = Low dose ChAd155-RSV vaccine (5 x  $10^9$  vp)

RSV-Md = Middle dose ChAd155-RSV vaccine  $(1.5 \times 10^{10} \text{ vp})$ 

RSV-Hd = High dose ChAd155-RSV vaccine (5 x 10<sup>10</sup> vp)

Placebo-Ld = Non-active control (0.5 ml)

Placebo-Md = Non-active control (0.15 ml)

Placebo-Hd = Non-active control (0.5 ml)

N = number of subjects in each group

n= Number of subjects with result available

SD=Standard Deviation

Q1, Q2 and Q3 = 1st, 2nd (median) and 3rd quantiles

Min/Max = Minimum/Maximum

95% CI = exact 95% confidence interval, LL = Lower Limit, UL = Upper Limit

Figure 2 Individuals results of hemoglobin levels in < group> <Exposed Set>



Note: This figure is shown as an example.

204838 (RSV PED-002) Statistical Analysis Plan Final

# Template 27 Exploratory comparisons between groups in terms of percentage of subjects reported any Grade 2/3 AE and/or any fever >38.5°C and/or any vaccine-related SAE during the 7-day (Days 1-7) post-vaccination period <Exposed Set>

| | | | | | | | | Difference in percentage<br>(Group 1 minus Group 2) | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | | 95 | % CI |
| Group 1 | N | n | % | Group 2 | N | n | % | Difference | % | LL | UL |
| RSV_Ld | | | | Placebo_Ld | | | | RSV_Ld - Placebo_Ld | | | |
| RSV_Md | | | | Placebo_Md | | | | RSV_Md - Placebo_Md | | | |
| RSV Hd | | | | Placebo Hd | | | | RSV Hd - Placebo Hd | | | |

#### <each group>:

RSV-Ld = Low dose ChAd155-RSV vaccine (5 x 109 vp)

RSV-Md = Middle dose ChAd155-RSV vaccine (1.5 x 10<sup>10</sup> vp)

RSV-Hd = High dose ChAd155-RSV vaccine (5 x 10<sup>10</sup> vp)

Placebo-Ld = Non-active control (0.5 ml)

Placebo-Md = Non-active control (0.15 ml)

Placebo-Hd = Non-active control (0.5 ml)

N = Number of subjects with the administered dose

n/% = number/percentage of subjects reporting a specified symptom

95% CI = Standardized asymptotic 95% confidence interval, LL = Lower Limit, UL = Upper Limit

204838 (RSV PED-002) Statistical Analysis Plan Final

# Template 28 Percentage of subjects reporting episode of spontaneous or excessive bleeding (AE of specific interest) classified by MedDRA Primary System Organ Class and Preferred Term within the 30-day (Days 1-30) post-vaccination period <Exposed Set>

| | | E | | gro<br>N = | up |
|---|---|---|---|---|---|
| | | | | 95 | % CI |
| Primary System Organ Class (CODE) | Preferred Term (CODE) | n* r | 1 % | LL | UL |
| At least one symptom | , i | | | | |
| Gastrointestinal disorders (10017947) | Diarrhoea (10012735) | | | | |
| , | Teething (10043183) | | | | |
| | Vomiting (10047700) | | | | |
| General disorders and administration site conditions (10018065) | Pyrexia (10037660) | | | | |
| Immune system disorders (10021428) | Seasonal allergy (10048908) | | | | |
| Infections and infestations (10021881) | Conjunctivitis (10010741) | | | | |
| | Otitis media (10033078) | | | | |
| | Paronychia (10034016) | | | | |
| | Tonsillitis (10044008) | | | | |
| | Tonsillitis streptococcal (10044013) | | | | |
| | Viral upper respiratory tract infection (10047482) | | | | |
| Injury, poisoning and procedural complications (10022117) | Arthropod bite (10003399) | | | | |
| ,, , | Face injury (10050392) | | | | |
| | Head injury (10019196) | | | | |
| Skin and subcutaneous tissue disorders (10040785) | Miliaria (10027627) | | | | |

RSV-Ld = Low dose ChAd155-RSV vaccine (5 x 109 vp)

RSV-Md = Middle dose ChAd155-RSV vaccine (1.5 x 10<sup>10</sup> vp)

RSV-Hd = High dose ChAd155-RSV vaccine (5 x  $10^{10}$  vp)

Placebo-Ld = Non-active control (0.5 ml)

Placebo-Md = Non-active control (0.15 ml)

Placebo-Hd = Non-active control (0.5 ml)

At least one symptom = at least one symptom experienced (regardless of the MedDRA Preferred Term)

N = number of subjects with at least one administered dose

n\* = number of events reported

n/% = number/percentage of subjects reporting the symptom at least once

95% CI = exact 95% confidence interval; LL = Lower Limit, UL = Upper Limit
204838 (RSV PED-002) Statistical Analysis Plan Final

# Template 29 Solicited and unsolicited symptoms classified by MedDRA Primary System Organ Class and Preferred Term within the 30-day (Days 1-30) post-vaccination period including number of events - SAE excluded <Exposed Set>

| | | | <each gr<br="">N =</each> | oup> |
|---|---|---|---|---|
| Primary System Organ Class (CODE) | Preferred Term (CODE) | n* | n | % |
| At least one symptom | , | | | |
| <each soc=""></each> | <each pt="" term=""></each> | | | |

#### <each group>:

RSV-Ld = Low dose ChAd155-RSV vaccine (5 x 109 vp)

RSV-Md = Middle dose ChAd155-RSV vaccine (1.5 x 10<sup>10</sup> vp)

RSV-Hd = High dose ChAd155-RSV vaccine (5 x  $10^{10}$  vp)

Placebo-Ld = Non-active control (0.5 ml)

Placebo-Md = Non-active control (0.15 ml)

Placebo-Hd = Non-active control (0.5 ml)

At least one symptom = at least one symptom experienced (regardless of the MedDRA Preferred Term)

N = number of subjects with the administered dose

n\* = number of events reported

n/% = number/percentage of subjects reporting the symptom at least once

204838 (RSV PED-002) Statistical Analysis Plan Final

## Template 30 Number (%) of subjects with serious adverse events from vaccination dose 1 up to Day X/Study end including number of events reported <Exposed Set>

| | | | <ea< th=""><th>ch gro<br/>N =</th><th>up&gt;</th></ea<> | ch gro<br>N = | up> |
|---|---|---|---|---|---|
| Type of Event | Primary System Organ Class | Preferred Term (CODE) | n* | n | % |
| SAE | At least one symptom | | | | |
| | <each soc=""></each> | <each pt="" term=""></each> | | | |
| Related SAE | At least one symptom | | | | |
| | <each soc=""></each> | <each pt="" term=""></each> | | | |
| Fatal SAE | At least one symptom | | | | |
| | <each soc=""></each> | <each pt="" term=""></each> | | | |
| Related fatal SAE | At least one symptom | | | | |
| | <each soc=""></each> | <each pt="" term=""></each> | | | |

#### <each group>:

RSV-Ld = Low dose ChAd155-RSV vaccine (5 x 109 vp)

RSV-Md = Middle dose ChAd155-RSV vaccine (1.5 x 10<sup>10</sup> vp)

RSV-Hd = High dose ChAd155-RSV vaccine (5 x  $10^{10}$  vp)

Placebo-Ld = Non-active control (0.5 ml)

Placebo-Md = Non-active control (0.15 ml)

Placebo-Hd = Non-active control (0.5 ml)

N = number of subjects with the administered dose

n\* = number of events reported

n/% = number/percentage of subjects reporting the symptom at least once

204838 (RSV PED-002) Statistical Analysis Plan Final

#### Template 31 Listing of unscheduled safety visit from vaccination dose 1 up to Day X/study end <Exposed Set>

| Group | Sub.<br>No. | Gender | Country | Race | VISIT | Date of previous safety sample | Timing | Laboratory parameter | Result | Unit | Grade |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | <timepoint previous="" safety="" to="" unsched=""></timepoint> | Hemoglobin | | | |
| | | | | | | | | Platelet count | | | |
| | | | | | | | UNSCHED SAFETY 1 | Hemoglobin | | | |
| | | | | | | | | Platelet count | | | |

#### <each group>:

RSV-Ld = Low dose ChAd155-RSV vaccine (5 x 109 vp)

RSV-Md = Middle dose ChAd155-RSV vaccine (1.5 x 10<sup>10</sup> vp)

RSV-Hd = High dose ChAd155-RSV vaccine (5 x 10<sup>10</sup> vp)

Placebo-Ld = Non-active control (0.5 ml)

Placebo-Md = Non-active control (0.15 ml)

Placebo-Hd = Non-active control (0.5 ml)

Please note the listing will be generated on group blinded at D61 and D366 analysis

28-MAR-2018 

204838 (RSV PED-002) Statistical Analysis Plan Final

#### Template 32 Listing of SAEs reported from vaccination dose 1 up to Day X visit /study end <Exposed Set>

| Group | Sub.<br>No. | Sex | Country | Race | Age at<br>onset<br>(Month) | Verbatim | Preferred<br>term | Primary<br>System<br>Organ<br>Class | MED<br>type | Dose | Day of onset | Duration | Intensity Causality | AMADILLI | criteria | Potential<br>AESI<br>(preferred<br>term) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|

#### <each group>:

RSV-Ld = Low dose ChAd155-RSV vaccine (5 x 109 vp)

RSV-Md = Middle dose ChAd155-RSV vaccine (1.5 x 10<sup>10</sup> vp)

RSV-Hd = High dose ChAd155-RSV vaccine (5 x 10<sup>10</sup> vp)

Placebo-Ld = Non-active control (0.5 ml)

Placebo-Md = Non-active control (0.15 ml)

Placebo-Hd = Non-active control (0.5 ml)

Potential AESI: AEs potentially related to spontaneous or excessive bleeding or LRTI will be identified based on the list of preferred terms described in section 11 –Annex

Please note the listing will be generated on group blinded at D61 and D366 analysis

28-MAR-2018 

204838 (RSV PED-002) Statistical Analysis Plan Final

Template 33 Listing of AEs related to LRTI and association to RSV infection from vaccination dose 1 up to Day X visit/study end <Exposed Set>

| Group | Sub. | Age at<br>onset<br>(month) | Verbatim | Preferred<br>term | Dose | lot | <br>End<br>date | Duration | Intensity | Causality | Local<br>RSV test<br>result | sample<br>for local | test | Central<br>test<br>RSV B | Date of<br>sample<br>for<br>central<br>testing | AESI |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|

RSV-Ld = Low dose ChAd155-RSV vaccine (5 x 109 vp)

RSV-Md = Middle dose ChAd155-RSV vaccine (1.5 x 10<sup>10</sup> vp)

RSV-Hd = High dose ChAd155-RSV vaccine (5 x  $10^{10}$  vp)

Placebo-Ld = Non-active control (0.5 ml)

Placebo-Md = Non-active control (0.15 ml)

Placebo-Hd = Non-active control (0.5 ml)

AESI: AEs of Special Interest - LRTI identified by the Investigator

\*AEs related to LRTI will be identified based on the list of preferred terms described in in section 12 -Annex 2

28-MAR-2018 

204838 (RSV PED-002) Statistical Analysis Plan Final

Template 34 Listing of RSV-RTI cases identified according to WHO case definitions and RSV-LRTI reported as AESI from vaccination dose 1 up to Day X visit /study end <Exposed Set>

| Grou | Sub.<br>No. | 1: | Surveillance<br>type | date of | End<br>date of<br>episode | SpO2 | IRespiratory | Local<br>RSV<br>test | for | Central | Central<br>test<br>RSV B | tor | | RSV-<br>LRTI | RSV-<br>severe<br>I RTI | RSV-<br>very<br>severe<br>LRTI | All-<br>cause<br>LRTI | AESI | Hospitalization |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | | | | | Yes/No | Yes/No | Yes/No | Yes/No | Yes/NO | Yes/No | Yes/No |

#### <each group>:

RSV-Ld = Low dose ChAd155-RSV vaccine (5 x 109 vp)

Placebo-Ld = Non-active control (0.5 ml)

RSV-Md = Middle dose ChAd155-RSV vaccine (1.5 x 10<sup>10</sup> vp)

Placebo-Md = Non-active control (0.15 ml)

RSV-Hd = High dose ChAd155-RSV vaccine (5 x  $10^{10}$  vp)

Placebo-Hd = Non-active control (0.5 ml)

AESI: AEs of Special Interest - LRTI identified by the Investigator

28-MAR-2018 

204838 (RSV PED-002) Statistical Analysis Plan Final

Template 35 Listing of AEs related to spontaneous or excessive bleeding together with hemoglobin and platelet count results from vaccination dose 1 up to Day 60 visit <Exposed Set>

| Group | Sub. No. | Age at onset (month) | Verbatim | Preferred term* | Previous<br>Dose | Day<br>of<br>onset | Duration | Intensity | Start date | End date | AESI | Date of sample | Laboratory parameter | Raw<br>result | Unit |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XX | XX | | XX | XX | XX | XX | | | XX | XX | | XX | Hemoglobin | | |
| | | | | | | | | | | | | | Platelet | | |
| | | | | | | | | | | | | | count | | |
| | | | | | | | | | | | | XX | Hemoglobin | | |
| | | | | | | | | | | | | | Platelet | | |
| | | | | | | | | | | | | | count | | |

RSV-Ld = Low dose ChAd155-RSV vaccine (5 x 109 vp)

RSV-Md = Middle dose ChAd155-RSV vaccine (1.5 x 10<sup>10</sup> vp)

RSV-Hd = High dose ChAd155-RSV vaccine (5 x 10<sup>10</sup> vp)

Placebo-Ld = Non-active control (0.5 ml)

Placebo-Md = Non-active control (0.15 ml)

Placebo-Hd = Non-active control (0.5 ml)

\*AEs related to spontaneous or excessive bleeding will be identified based on the list of preferred terms described in section 12 –Annex

AESI: AEs of Special Interest - Spontaneous or excessive bleeding identified by the Investigator

28-MAR-2018 

204838 (RSV PED-002) Statistical Analysis Plan Final

### Template 36 Listing of adverse events, SAEs and solicited symptoms leading to withdrawal from the study or treatment from vaccination dose 1 up to Day X visit/study end <Exposed Set>

| Group | Subject No. | Country | Gender | Race | AE Description | SAE | Causality | Outcome | Type of discontinuation |
|---|---|---|---|---|---|---|---|---|---|

RSV-Ld = Low dose ChAd155-RSV vaccine (5 x 109 vp)

RSV-Md = Middle dose ChAd155-RSV vaccine (1.5 x 10<sup>10</sup> vp)

RSV-Hd = High dose ChAd155-RSV vaccine (5  $\times$  10<sup>10</sup> vp)

Placebo-Ld = Non-active control (0.5 ml)

Placebo-Md = Non-active control (0.15 ml)

Placebo-Hd = Non-active control (0.5 ml)

28-MAR-2018 

204838 (RSV PED-002) Statistical Analysis Plan Final

### Template 37 Number and percentage of subjects with anti-RSV-A neutralising antibody titre equal to or above <cut-off> and GMTs <PPS for analysis of immunogenicity at Day X>

| | | | | | ≥cut- | off un | it | | GMT | Ī | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | 95 | % CI | | 9 | 95% CI | | |
| Antibody | Group | Timing | N | n | % | LL | UL | value | LL | UL | Min | Max |
| Anti-RSV-A<br>Neutralizing<br>Antibody | <each<br>group&gt;</each<br> | PRE | | | | | | | | | | |
| • | | PI(D31) | | | | | | | | | | |
| | | PII(D61) | | | | | | | | | | |
| | | PII(D366) | | | | | | | | | | |

#### <each group>:

RSV-Ld = Low dose ChAd155-RSV vaccine (5 x 109 vp)

RSV-Md = Middle dose ChAd155-RSV vaccine (1.5 x 10<sup>10</sup> vp)

RSV-Hd = High dose ChAd155-RSV vaccine (5 x  $10^{10}$  vp)

Placebo-Ld = Non-active control (0.5 ml)

Placebo-Md = Non-active control (0.15 ml)

Placebo-Hd = Non-active control (0.5 ml)

GMT = geometric mean antibody titre calculated on all subjects

N = Number of subjects with available results

95% CI = 95% confidence interval; LL = lower limit, UL = upper limit

n/% = number/percentage of subjects with titer equal to or above specified value

MIN/MAX = Minimum/Maximum

PRE= Pre-vaccination at Day 1

PI(D31) = Post-vaccination dose 1 at Day 31

PII(D61) = Post-vaccination dose 2 at Day 61

204838 (RSV PED-002) Statistical Analysis Plan Final

### Template 38 Vaccine response for anti-RSV-A neutralising antibody titre at each post-vaccination timepoint <PPS for analysis of immunogenicity at Day X>

| | | | | | <each gro<="" th=""><th>oup&gt;</th><th></th></each> | oup> | |
|---|---|---|---|---|---|---|---|
| | | | | | | . ( | 95% CI |
| Antibody | Timing | Pre-vaccination status | N | n | % | LL | UL |
| <each antibody=""></each> | PII(D61) | <128 | | | | | |
| • | , , | ≥128 - ≤256 | | | | | |
| | | >256-≤1024 | | | | | |
| | | >1024 | | | | | |
| | | Total | | | | | |
| | PII(D366) | <128 | | | | | |
| | | ≥128 - ≤256 | | | | | |
| | | >256-≤1024 | | | | | |
| | | >1024 | | | | | |
| | | Total | | | | | |

#### <each group>:

RSV-Ld = Low dose ChAd155-RSV vaccine (5 x 109 vp)

RSV-Md = Middle dose ChAd155-RSV vaccine (1.5 x 10<sup>10</sup> vp)

RSV-Hd = High dose ChAd155-RSV vaccine (5 x 10<sup>10</sup> vp)

Placebo-Ld = Non-active control (0.5 ml)

Placebo-Md = Non-active control (0.15 ml)

Placebo-Hd = Non-active control (0.5 ml)

Total = all subjects with pre-and post- vaccination result available

Vaccine response defined as:

For subjects with pre-vaccination titer <128: antibody titer at post-vaccination>= 4 fold the pre-vaccination antibody titer For subjects with pre-vaccination titer in ≥128 - ≤256: antibody titer at post-vaccination >= 3 fold the pre-vaccination antibody titer

For subjects with pre-vaccination titer in >256-≤1024: antibody titer at post-vaccination>= 2.5 fold the pre-vaccination antibody titer

For subjects with pre-vaccination titer >1024: antibody titer at post-vaccination >= 1 fold the pre-vaccination antibody titer

N = number of subjects with both pre- and post-vaccination results available

n/% = number/percentage of responders

95% CI = exact 95% confidence interval, LL = Lower Limit, UL = Upper Limit

PII(D61) = Post-vaccination dose 2 at Day 61

204838 (RSV PED-002) Statistical Analysis Plan Final

### Template 39 Distribution of anti-RSV-A neutralising antibody titer <PPS for analysis of immunogenicity at Day X>

| | | | | Each gro | up |
|----------------------------------|--------|-------|---|----------|----|
| Antibody | Timing | Titre | N | n | % |
| Anti-RSV A Neutralizing Antibody | PRE | <128 | | | |
| | | ≥128 | | | |
| | | ≥256 | | | |
| | | ≥512 | | | |
| | | ≥1024 | | | |
| | | ≥2048 | | | |
| | | ≥4098 | | | |

#### <each group>:

RSV-Ld = Low dose ChAd155-RSV vaccine (5 x 109 vp)

RSV-Md = Middle dose ChAd155-RSV vaccine (1.5 x 10<sup>10</sup> vp)

RSV-Hd = High dose ChAd155-RSV vaccine (5 x  $10^{10}$  vp)

Placebo-Ld = Non-active control (0.5 ml)

Placebo-Md = Non-active control (0.15 ml)

Placebo-Hd = Non-active control (0.5 ml)

N = number of subjects with available results

n/% = number/percentage of subjects with titre within the specified criterion

PRE = Pre-vaccination at Day 1

PI(D31) = Post-vaccination dose 1 at Day 31

PII(D61) = Post-vaccination dose 2 at Day 61

204838 (RSV PED-002) Statistical Analysis Plan Final

#### Template 40 Distribution of fold of anti-RSV-A neutralising antibody titer by prevaccination titer category <PPS for analysis of immunogenicity at Day X>

| | | | | E | ach g | roup |
|---|---|---|---|---|---|---|
| Antibody | Fold change | Pre-vaccination status | Timing | N | n | % |
| Anti-RSV A Neutralizing<br>Antibody | <1 | <128 | PI(D31) | | | |
| | | | PII(D61) | | | |
| | | | PII(D366) | | | |
| | | ≥128-≤256 | , | | | |
| | | >256-≤512 | | | | |
| | | >1024-≤2048 | | | | |
| | | >2048-≤4096 | | | | |
| | | >4096 | | | | |
| | | Total | | | | |
| | ≥1 | | | | | |
| | ≥2 | | | | | |
| | ≥2.5 | | | | | |
| | ≥3 | | | | | |
| | ≥4 | | | | | |
| | ≥6 | | | | | |
| | ≥8 | | | | | |
| | ≥10 | | | | | |
| | ≥11 | | | | | |
| | ≥12 | | | | | |

#### <each group>:

RSV-Ld = Low dose ChAd155-RSV vaccine (5 x 109 vp)

RSV-Md = Middle dose ChAd155-RSV vaccine (1.5 x 10<sup>10</sup> vp)

RSV-Hd = High dose ChAd155-RSV vaccine (5 x 10<sup>10</sup> vp)

Placebo-Ld = Non-active control (0.5 ml)

Placebo-Md = Non-active control (0.15 ml)

Placebo-Hd = Non-active control (0.5 ml)

N = number of subjects with pre and corresponding post-vaccination results available

n/% = number/percentage of subjects with titre fold change meeting the specified criterion

PI(D31) = Post-vaccination dose 1 at Day 31

PII(D61) = Post-vaccination dose 2 at Day 61

204838 (RSV PED-002) Statistical Analysis Plan Final

# Template 41 Geometric mean of the individual ratio of anti-RSV-A neutralising antibody titers at each post-vaccination timepoint compared to prevaccination with 95% CI <PPS for analysis of immunogenicity at Day X>

| | | | | | | GMT ratio | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | 9 | 5% CI |
| Group | N | Time point description | GMT | Time point description | GMT | Ratio order | Value | LL | UL |
| <each group=""></each> | | PI(D31) | | PRE | | PI(D31) / PRE | | | |
| | | PII(D61) | | PRE | | PII(D61) / PRE | | | |
| | | PII(D366) | | PRE | | PII(D366) / PRE | | | |

#### <each group>:

RSV-Ld = Low dose ChAd155-RSV vaccine (5 x 109 vp)

RSV-Md = Middle dose ChAd155-RSV vaccine (1.5 x 10<sup>10</sup> vp)

RSV-Hd = High dose ChAd155-RSV vaccine (5 x 10<sup>10</sup> vp)

Placebo-Ld = Non-active control (0.5 ml)

Placebo-Md = Non-active control (0.15 ml)

Placebo-Hd = Non-active control (0.5 ml)

GMT = geometric mean antibody titer

N = Number of subjects with available results at the two considered time points

95% CI = 95% confidence interval; LL = Lower Limit, UL = Upper Limit

PRE= Pre-vaccination at Day 1

PI(D31) = Post-vaccination dose 1 at Day 31

PII(D61) = Post-vaccination dose 2 at Day 61

Figure 3 Reverse cumulative distribution curves for anti-RSV-A neutralising antibody titres in each group at baseline and <D60/D365> <PPS for analysis of immunogenicity at Day X>



RSV-Ld = Low dose ChAd155-RSV vaccine (5 x 109 vp)

RSV-Md = Middle dose ChAd155-RSV vaccine (1.5 x 10<sup>10</sup> vp)

RSV-Hd = High dose ChAd155-RSV vaccine (5 x 10<sup>10</sup> vp)

Placebo-Ld = Non-active control (0.5 ml)

Placebo-Md = Non-active control (0.15 ml)

Placebo-Hd = Non-active control (0.5 ml)

Note: This graph is provided as an example. The same graph will be provided in colour for each time point and each assay comparing the values of the groups

Figure 4 Individual results of anti-RSV-A neutralising antibody titre at Day <60/365> versus pre-vaccination in <each group> and Control group> <PPS for analysis of immunogenicity at Day X>



#### <each group>:

RSV-Ld = Low dose ChAd155-RSV vaccine (5 x 109 vp)

RSV-Md = Middle dose ChAd155-RSV vaccine (1.5 x 10<sup>10</sup> vp)

RSV-Hd = High dose ChAd155-RSV vaccine (5 x 10<sup>10</sup> vp)

Placebo-Ld = Non-active control (0.5 ml)

Placebo-Md = Non-active control (0.15 ml)

Placebo-Hd = Non-active control (0.5 ml)

Note: This graph is provided as an example. The same graph will be generated for each assay and each timepoint separately (Days 61, 366):

204838 (RSV PED-002) Statistical Analysis Plan Final

Template 42 Descriptive statistics on the frequency of CD4+ T-cells expressing at least two markers among CD40L, IL-2, TNF-α, and IFN-γ upon stimulation with <RSV F/ N /M2-1/combined> peptide pool <PPS for analysis of immunogenicity at Day X>

| | | | | <each g<="" th=""><th>group&gt;</th><th>•</th></each> | group> | • |
|---|---|---|---|---|---|---|
| Stimulation | Group | Timing | Paramter | Value | LĹ | UL |
| FNg protein – RSV F pool 15/11 Ag | | PRE | n | | | |
| | | | NMiss | | | |
| | | | GM | | | |
| | | | Mean | | | |
| | | | SD | | | |
| | | | Min | | | |
| | | | Q1 | | | |
| | | | Median | | | |
| | | | Q3 | | | |
| | | | Max | | | |
| | | PI(D31) | | | | |
| | | PII(D61) | | | | |
| | | PII(D366) | | | | |
| FNg protein – RSV N pool 15/11 Ag | | PRE | | | | |
| | | PI(D31) | | | | |
| | | PII(D61) | | | | |
| | | PII(D366) | | | | |
| FNg protein – RSV M2-1 pool 15/11 Ag | | PRE | | | | |
| | | PI(D31) | | | | |
| | | PII(D61) | | | | |
| | | PII(D366) | | | | |
| Combined (F,N and M2-1) | | PRE | | | | |
| | PI(D3 | | | | | |
| | | PII(D61) | | | | |
| | | PII(D366) | | | | |

RSV-Ld = Low dose ChAd155-RSV vaccine (5 x 109 vp)

RSV-Md = Middle dose ChAd155-RSV vaccine (1.5 x 10<sup>10</sup> vp)

RSV-Hd = High dose ChAd155-RSV vaccine (5 x 10<sup>10</sup> vp)

Placebo-Ld = Non-active control (0.5 ml)

Placebo-Md = Non-active control (0.15 ml)

Placebo-Hd = Non-active control (0.5 ml)

N = number of subjects with available results;

Nmiss = number of subjects with missing results

GM= Geometric Mean

SD = Standard Deviation

Q1,Q3 = First and third quartiles

Min/Max = Minimum/Maximum

PRE = Pre-vaccination at Day 1

PI(D31) = Post-vaccination dose 1 at Day 31

PII(D61) = Post-vaccination dose 2 at Day 61

PII(D366) = Post-vaccination dose 2 at Day 366

Please note that for combined peptide pool, we will only consider subjects who has data available for the three peptide pools

Figure 5 Boxplots of individual data for CD4+ T-cells expressing at least two markers among CD40L, IL-2, TNF-α, and IFN-γ upon stimulation with <RSV F/ N /M2-1/combined> peptide pool <from pre-vaccination to Day 61/Day 366> <PPS for analysis of immunogenicity at Day X>



RSV-Ld = Low dose ChAd155-RSV vaccine (5 x 109 vp)

RSV-Md = Middle dose ChAd155-RSV vaccine (1.5 x 10<sup>10</sup> vp)

RSV-Hd = High dose ChAd155-RSV vaccine (5 x 10<sup>10</sup> vp)

Placebo-Ld = Non-active control (0.5 ml)

Placebo-Md = Non-active control (0.15 ml)

Placebo-Hd = Non-active control (0.5 ml)

PRE= Pre-vaccination at Day 1

PI(D31) = Post-vaccination dose 1 at Day 31

PII(D61) = Post-vaccination dose 2 at Day 61

PII(D366) = Post-vaccination dose 2 at Day 366

Note: This graph is provided as an example. Template will be adapted to display the 3 RSV or 3Control groups together and the 4 timepoints: PRE, PI(D31), PII(D61) and PII(D366).

Please note – To present the information on pooled RSV and pooled Placebo after looking at the data of Day 61 analysis.

Figure 6 Co-expression profile of the RSV <F/N/M2-1> specific <CD4+> T-cells expressing at least two markers among CD40L, IL-2, TNF- $\alpha$ , and IFN-  $\gamma$  in <RSV-Ld group> <PPS for analysis of immunogenicity at Day X>



RSV-Ld = Low dose ChAd155-RSV vaccine (5 x 109 vp)

RSV-Md = Middle dose ChAd155-RSV vaccine (1.5 x 10<sup>10</sup> vp)

RSV-Hd = High dose ChAd155-RSV vaccine (5 x  $10^{10}$  vp)

Placebo-Ld = Non-active control (0.5 ml)

Placebo-Md = Non-active control (0.15 ml)

Placebo-Hd = Non-active control (0.5 ml)

Note: This graph is given as an example. Template will be adapted to display Q1-Median-Q3 for each combination of atleast 2 markers out of (CD40L, IL-2, TNF- $\alpha$ , and IFN- $\gamma \rightarrow 11$  combinations) for each timepoint: PRE, PI(D31), PII(D61) and PII(D366). It will be generated for each vaccine group and each RSV pool of peptides (RSV F/N/M2-1).

204838 (RSV PED-002) Statistical Analysis Plan Final

Template 43 Number and percentage of subjects with at least one RSV infection, RSV-RTI, RSV-LRTI, RSV-severe LRTI, RSV-very severe LRTI, All-cause LRTI and RSV hospitalization from vaccination dose 1 up to D366/D731 visit <Exposed Set>

| | | Total<br>N = | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | 95 | % CI | | | | 95% | <b>6 CI</b> |
| Categories | n** | n | % | LL | UL | n** | n | % | LL | UL |
| No Infection | | | | | | | | | | |
| RSV infection - symptomatic or asymptomatic* | | | | | | | | | | |
| RSV-RTI | | | | | | | | | | |
| RSV-LRTI | | | | | | | | | | |
| RSV-severe LRTI | | | | | | | | | | |
| RSV-very severe LRTI | | | | | | | | | | |
| All-cause LRTI | | | | | | | | | | |
| RSV hospitalization\$ | | | | | | | | | | |

RSV-Ld = Low dose ChAd155-RSV vaccine (5 x 109 vp)

RSV-Md = Middle dose ChAd155-RSV vaccine (1.5 x 10<sup>10</sup> vp)

RSV-Hd = High dose ChAd155-RSV vaccine (5 x 10<sup>10</sup> vp)

Placebo-Ld = Non-active control (0.5 ml)

Placebo-Md = Non-active control (0.15 ml)

Placebo-Hd = Non-active control (0.5 ml)

RSV = ChAd155-RSV vaccine (low/ middle/high dose pooled groups)

Placebo = Non-active control (0.5/0.15/0.5 ml pooled groups)

\$Confirmed RSV infection and hospitalized for acute medical condition

N = number of subjects in each group

n\*\* = number of cases in each category

n/%= number/percentage of subjects reporting at least once the case

95%CI= Exact 95% confidence interval; LL = lower limit, UL = upper limit

Please note - Single episode can be considered in multiple category depending on the symptom experienced

<sup>\*</sup> Association to RSV based on central testing only for asymptomatic visit (no local test available)

204838 (RSV PED-002) Statistical Analysis Plan Final

## Template 44 Number and percentage of subjects reporting the RSV infection of different severity by number of events experienced between vaccination dose 1 up to D366/D731 visit <Exposed Set>

| | | | <e< th=""><th>ach gro</th><th>up&gt;</th></e<> | ach gro | up> |
|---|---|---|---|---|---|
| | | | | 9 | 95% CI |
| Characteristics | Categories | n | % | LL | UL |
| RSV infection-symptomatic or asymptomatic* | 0 | | | | |
| | 1 | | | | |
| | 2 | | | | |
| RSV-RTI | 0 | | | | |
| | 1 | | | | |
| RSV-LRTI | 0 | | | | |
| | 1 | | | | |
| | 2 | | | | |
| RSV-Severe LRTI | 0 | | | | |
| | 1 | | | | |
| RSV-very severe LRTI | 0 | | | | |
| • | 1 | | | | |
| All cause LRTI | 0 | | | | |
| | 1 | | | | |
| | 2 | | | | |
| | 3 | | | | |
| RSV hospitalization\$ | 0 | | | | |
| · | 1 | | | | |
| | 2 | | | | |
| | 3 | | | | |

RSV-Ld = Low dose ChAd155-RSV vaccine (5 x 109 vp)

RSV-Md = Middle dose ChAd155-RSV vaccine (1.5 x 10<sup>10</sup> vp)

RSV-Hd = High dose ChAd155-RSV vaccine (5 x 10<sup>10</sup> vp)

Placebo-Ld = Non-active control (0.5 ml)

Placebo-Md = Non-active control (0.15 ml)

Placebo-Hd = Non-active control (0.5 ml)

RSV = ChAd155-RSV vaccine (low/ middle/high dose pooled groups)

Placebo = Non-active control (0.5/0.15/0.5 ml pooled groups)

N = number of subjects in each group

n = number of subjects in a given category

% =100\*n/N

LL, UL for percentage = Exact 95% Lower and Upper confidence limits

Please note – Single episode can be considered in multiple category depending on the symptom experienced

<sup>\*</sup> Association to RSV based on central testing only for asymptomatic visit (no local test available)

<sup>\$</sup>Confirmed RSV infection and hospitalized for acute medical condition

204838 (RSV PED-002) Statistical Analysis Plan Final

### Template 45 Number and percentage of RSV infections and associated disease severity between vaccination dose 1 up to D366/D731 visit <Exposed Set>

| | | | Grou<br>N = | • | | - | otal<br>N = | |
|---|---|---|---|---|---|---|---|---|
| | 95% CI | | | | | | 9 | 5% CI |
| Categories | n | % | LL | UL | n | n % | | UL |
| RSV asymptomatic (Excluding RSV-RTI, LRTI, RSV-severe LRTI or RSV- | | | | | | | | |
| very severe LRTI) | | | | | | | | |
| RSV RTI (Excluding LRTI, RSV-severe or very severe LRTI) | | | | | | | | |
| RSV LRTI (Excluding RSV-severe or very severe LRTI) | | | | | | | | |
| RSV-severe LRTI (Excluding RSV-very severe LRTI) | | | | | | | | |
| RSV-very severe LRTI | | | | | | | | |

RSV-Ld = Low dose ChAd155-RSV vaccine (5 x 109 vp)

RSV-Md = Middle dose ChAd155-RSV vaccine (1.5 x 10<sup>10</sup> vp)

RSV-Hd = High dose ChAd155-RSV vaccine (5 x 10<sup>10</sup> vp)

Placebo-Ld = Non-active control (0.5 ml)

Placebo-Md = Non-active control (0.15 ml)

Placebo-Hd = Non-active control (0.5 ml)

RSV = ChAd155-RSV vaccine (low/ middle/high dose pooled groups)

Placebo = Non-active control (0.5/0.15/0.5 ml pooled groups)

N = number of RSV positive samples in each group

n\*\* = number of cases in each category

n/%= number/percentage of cases in each category

95%CI= Exact 95% confidence interval; LL = lower limit, UL = upper limit

Please note - Single episode is considered in single category of highest severity based on the symptom experienced

<sup>\*</sup> Association to RSV based on central testing only for asymptomatic visit (no local test available)

204838 (RSV PED-002) Statistical Analysis Plan Final

### Template 46 Number and percentage of RSV infections requiring hospitalization between vaccination dose 1 up to D366/D731 <Exposed Set>

| | | Group<br>N = | | | Total<br>N = | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | 95 | % CI | | | | 959 | % CI |
| Categories | n** | n | % | LL | UL | n** | N | % | LL | UL |
| RSV RTI*(Excluding LRTI, severe or very severe LRTI) | | | | | | | | | | |
| RSV LRTI (Excluding severe or very severe LRTI) | | | | | | | | | | |
| RSV-severe LRTI (Excluding very severe LRTI) | | | | | | | | | | |
| RSV-very severe LRTI | | | | | | | | | | |

RSV-Ld = Low dose ChAd155-RSV vaccine (5 x 109 vp)

RSV-Md = Middle dose ChAd155-RSV vaccine (1.5 x 10<sup>10</sup> vp)

RSV-Hd = High dose ChAd155-RSV vaccine (5 x 10<sup>10</sup> vp)

Placebo-Ld = Non-active control (0.5 ml)

Placebo-Md = Non-active control (0.15 ml)

Placebo-Hd = Non-active control (0.5 ml)

RSV = ChAd155-RSV vaccine (low/ middle/high dose pooled groups)

Placebo = Non-active control (0.5/0.15/0.5 ml pooled groups)

N = number of RSV infections in each group

n\*\* = number of cases in each category

n/%= number/percentage of subjects reporting at least once the case

95%CI= Exact 95% confidence interval; LL = lower limit, UL = upper limit

204838 (RSV PED-002) Statistical Analysis Plan Final

### Template 47 Descriptive statistics of viral load calculated on all qRT-PCR confirmed RSV infection episodes with varying disease severity from vaccination dose 1 up to D366/D731 <Exposed Set>

| Symptoms | Parameters | Value | LL | UL |
|---|---|---|---|---|
| RSV asymptomatic* (Excluding RSV-RTI, RSV-LRTI, RSV-severe LRTI or RSV-very severe LRTI) | n | | | |
| | GM | | | |
| | 95% CI | | | |
| | SD | | | |
| | Q1 | | | |
| | Median | | | |
| | Q3 | | | |
| | Min/Max | | | |
| RSV RTI (Excluding RSV-LRTI, RSV-severe LRTI or RSV-very severe LRTI) | | | | |
| RSV LRTI (Excluding RSV-severe or RSV-very severe LRTI) | | | | |
| RSV-severe LRTI (Excluding RSV-very severe LRTI) | | | | |
| RSV-very severe LRTI | | | | |
| RSV hospitalization\$ | | | | |

RSV-Ld = Low dose ChAd155-RSV vaccine (5 x 109 vp)

RSV-Md = Middle dose ChAd155-RSV vaccine (1.5 x 10<sup>10</sup> vp)

RSV-Hd = High dose ChAd155-RSV vaccine (5 x  $10^{10}$  vp)

Placebo-Ld = Non-active control (0.5 ml)

Placebo-Md = Non-active control (0.15 ml)

Placebo-Hd = Non-active control (0.5 ml)

RSV = ChAd155-RSV vaccine (low/ middle/high dose pooled groups)

Placebo = Non-active control (0.5/0.15/0.5 ml pooled groups)

N = number of RSV infections episodes in each group

n= Number of events in each category

SD=Standard Deviation

Q1 and Q3 = 1st and 3rd quantiles

Min/Max = Minimum/Maximum

GM = Geometric mean

LL, UL for GM = Exact 95% Lower and Upper confidence limits

Total RSV viral load computed as RSV A Viral load + RSV B Viral load

\* Association to RSV based on central testing only for asymptomatic visit (no local test available)

\$Confirmed RSV infection and hospitalized for acute medical condition

Please note: each episode for a subject is considered to be independent. We may have multiple swab for one episode. We have considered the swab with maximum viral load from one episode for the table

Please note – Except for RSV hospitalization, single episode is considered in single category of highest severity based on the symptom experienced

Please check:- To check for cases where asymptomatic swab has been taken but the subject hasve symptoms of RTI or LRTI. In this case, asymptomatic is also considered as RSV RTI/LRTI and maximum viral load of all the episode should be considered.

204838 (RSV PED-002) Statistical Analysis Plan Final

## Template 48 Descriptive statistics of maximum viral load per subjects based on qRT-PCR confirmed episode with varying disease severity form vaccination dose 1 up to D366/D731 <Exposed Set>

| | | Ea | ch Grou <sub>l</sub><br>N= | ) |
|---|---|---|---|---|
| | | | 95 | % CI |
| Symptoms | Parameters | Value | LL | UL |
| RSV asymptomatic* (Excluding RSV-RTI, RSV-LRTI, RSV-severe LRTI or RSV-very severe LRTI) | n | | | |
| • | GM | | | |
| | 95% CI | | | |
| | SD | | | |
| | Q1 | | | |
| | Median | | | |
| | Q3 | | | |
| | Min/Max | | | |
| RSV RTI (Excluding RSV-LRTI, RSV-severe or RSV-very severe LRTI) | | | | |
| RSV LRTI (Excluding RSV-severe or RSV-very severe LRTI) | | | | |
| RSV-severe LRTI (Excluding RSV-very severe LRTI) | | | | |
| RSV-very severe LRTI | | | | |
| RSV hospitalization\$ | | | | |

RSV-Ld = Low dose ChAd155-RSV vaccine (5 x 109 vp)

RSV-Md = Middle dose ChAd155-RSV vaccine (1.5 x 10<sup>10</sup> vp)

RSV-Hd = High dose ChAd155-RSV vaccine (5 x  $10^{10}$  vp)

Placebo-Ld = Non-active control (0.5 ml)

Placebo-Md = Non-active control (0.15 ml)

Placebo-Hd = Non-active control (0.5 ml)

RSV = ChAd155-RSV vaccine (low/ middle/high dose pooled groups)

Placebo = Non-active control (0.5/0.15/0.5 ml pooled groups)

N = number of RSV positive subjects in each group

n= Number of subjects in each category

SD=Standard Deviation

Q1 and Q3 = 1st and 3rd quantiles

Min/Max = Minimum/Maximum

GM = Geometric mean

LL, UL for GM = Exact 95% Lower and Upper confidence limits

Total RSV viral load computed as RSV A Viral load + RSV B Viral load

Please note: Except of RSV hospitalization, the subject has been considered only once in one of the category based on the maximum severity of event experienced

<sup>\*</sup> Association to RSV based on central testing only for asymptomatic visit (no local test available)

<sup>\$</sup>Confirmed RSV infection and hospitalized for acute medical condition

204838 (RSV PED-002) Statistical Analysis Plan Final

### Template 49 Frequency of multiple respiratory pathogen for qRT-PCR confirmed RSV-RTI episodes from vaccination dose 1 up to D366/D731 visit <Exposed Set>

| | | | Gro<br>N | • | Total<br>N = | | | |
|---|---|---|---|---|---|---|---|---|
| | | | 9 | 5% CI | | | 9 | 5% CI |
| Categories | n | % | LL | UL | n | % | LL | UL |
| Influenza Virus A/California/7/2009(H1N1) | | | | | | | | |
| Adenovirus | | | | | | | | |
| Human Coronavirus OC43 | | | | | | | | |
| Human Coronavirus 229E | | | | | | | | |
| Human Coronavirus NL63 | | | | | | | | |
| Human Coronavirus HKU1 | | | | | | | | |
| Enterovirus + Rhinovirus | | | | | | | | |
| Influenza Virus A | | | | | | | | |
| Influenza Virus B | | | | | | | | |
| Influenza Virus A (H1N1) | | | | | | | | |
| Influenza Virus A (H3N2) | | | | | | | | |
| Human bocavirus | | | | | | | | |
| Human metapneumovirus | | | | | | | | |
| Parainfluenza virus 1 | | | | | | | | |
| Parainfluenza virus 2 | | | | | | | | |
| Parainfluenza virus 3 | | | | | | | | |
| Parainfluenza virus 4 | | | | | | | | |

RSV-Ld = Low dose ChAd155-RSV vaccine (5 x 109 vp)

RSV-Md = Middle dose ChAd155-RSV vaccine (1.5 x 10<sup>10</sup> vp)

RSV-Hd = High dose ChAd155-RSV vaccine (5 x  $10^{10}$  vp)

Placebo-Ld = Non-active control (0.5 ml)

Placebo-Md = Non-active control (0.15 ml)

Placebo-Hd = Non-active control (0.5 ml)

RSV = ChAd155-RSV vaccine (low/ middle/high dose pooled groups)

Placebo = Non-active control (0.5/0.15/0.5 ml pooled groups)

N = number of qRT-PCR confirmed RSV-RTI infection episodes in each group

n = number of episodes in a given category

% =100\*n/N

LL, UL for percentage = Exact 95% Lower and Upper confidence limits

204838 (RSV PED-002) Statistical Analysis Plan Final

### Template 50 Frequency of multiple respiratory pathogen for confirmed LRTI episodes from vaccination dose 1 up to D366/D731 visit <Exposed Set>

| | | | Gro<br>N : | | Total<br>N = | | | |
|---|---|---|---|---|---|---|---|---|
| | | | 9 | 5% CI | | | 9 | 5% CI |
| Categories | n | % | LL | UL | n | % | LL | J |
| Respiratory syncytial virus | | | | | | | | |
| Influenza Virus A/California/7/2009(H1N1) | | | | | | | | |
| Adenovirus | | | | | | | | |
| Human Coronavirus OC43 | | | | | | | | |
| Human Coronavirus 229E | | | | | | | | |
| Human Coronavirus NL63 | | | | | | | | |
| Human Coronavirus HKU1 | | | | | | | | |
| Enterovirus + Rhinovirus | | | | | | | | |
| Influenza Virus A | | | | | | | | |
| Influenza Virus B | | | | | | | | |
| Influenza Virus A (H1N1) | | | | | | | | |
| Influenza Virus A (H3N2) | | | | | | | | |
| Human bocavirus | | | | | | | | |
| Human metapneumovirus | | | | | | | | |
| Parainfluenza virus 1 | | | | | | | | |
| Parainfluenza virus 2 | | | | | | | | |
| Parainfluenza virus 3 | | | | | | | | |
| Parainfluenza virus 4 | | | | | | | | |

RSV-Ld = Low dose ChAd155-RSV vaccine (5 x 109 vp)

RSV-Md = Middle dose ChAd155-RSV vaccine (1.5 x 10<sup>10</sup> vp)

RSV-Hd = High dose ChAd155-RSV vaccine (5 x 10<sup>10</sup> vp)

Placebo-Ld = Non-active control (0.5 ml)

Placebo-Md = Non-active control (0.15 ml)

Placebo-Hd = Non-active control (0.5 ml)

RSV = ChAd155-RSV vaccine (low/ middle/high dose pooled groups)

Placebo = Non-active control (0.5/0.15/0.5 ml pooled groups)

N = number of confirmed LRTI infection episodes in each group

n = number of episodes in a given category

% =100\*n/N

LL, UL for percentage = Exact 95% Lower and Upper confidence limits

204838 (RSV PED-002) Statistical Analysis Plan Final

#### Template 51 Listing of RSV-RTI cases identified according to case definitions <Exposed Set>

| Gro | oup | Sub.<br>No. | Sex | Age at<br>episode(month) | Country | Site | Surveillance<br>type | Episode<br>nb | Dose . | Onset<br>day | SpO2 | Irate | test | tact . | RSV-<br>RTI | RSV-<br>LRTI | IRSV- | RSV-<br>very<br>severe<br>LRTI | Hospitalization | RVP<br>result |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | | | | | | | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | |

#### <each group>:

RSV-Ld = Low dose ChAd155-RSV vaccine (5 x 109 vp)

Placebo-Ld = Non-active control (0.5 ml)

RSV-Md = Middle dose ChAd155-RSV vaccine (1.5 x 10<sup>10</sup> vp)

Placebo-Md = Non-active control (0.15 ml)

RSV-Hd = High dose ChAd155-RSV vaccine (5 x 10<sup>10</sup> vp)

Placebo-Hd = Non-active control (0.5 ml)

RSV-LM=ChAd155-RSV vaccine (low/ middle dose pooled groups)

Placebo-LM= Non-active control (0.5/0.15 ml pooled groups)

RSV = ChAd155-RSV vaccine (low/ middle/high dose pooled groups)

Placebo = Non-active control (0.5/0.15/0.5 ml pooled groups)

28-MAR-2018 

204838 (RSV PED-002) Statistical Analysis Plan Final

#### Template 52 Listing of RSV-RTI requiring hospitalization and type of inpatient facility required <Exposed Set>

| ( | iroun l | Sub.<br>No. | Sex | Age at<br>episode(month) | Country | Classification<br>of episode<br>per WHO* | Total days<br>hospitalized | No. of<br>days of<br>monitoring<br>or nursing | nasogastric<br>or | No. of days<br>oxygen<br>administered | days<br>respiratory | No. of days<br>mechanical<br>ventilation<br>given | kept in | RVP<br>result | Pathogen<br>identified<br>in RVP |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | | | | | | Yes/No | |

RSV-Ld = Low dose ChAd155-RSV vaccine (5 x 109 vp)

Placebo-Ld = Non-active control (0.5 ml)

RSV-Md = Middle dose ChAd155-RSV vaccine (1.5 x 10<sup>10</sup> vp)

Placebo-Md = Non-active control (0.15 ml)

RSV-Hd = High dose ChAd155-RSV vaccine (5 x  $10^{10}$  vp)

Placebo-Hd = Non-active control (0.5 ml)

RSV-LM=ChAd155-RSV vaccine (low/ middle dose pooled groups)

Placebo-LM= Non-active control (0.5/0.15 ml pooled groups)

RSV = ChAd155-RSV vaccine (low/ middle/high dose pooled groups)

Placebo = Non-active control (0.5/0.15/0.5 ml pooled groups)

\*subject will be classified per maximum severity experienced

28-MAR-2018 

204838 (RSV PED-002) Statistical Analysis Plan Final

### Template 53 Number and percentage of subjects with highest associated severity of RSV infection from vaccination dose 1 up to D366/D731 visit <Exposed Set>

| Group<br>N = | | | | Total<br>N = | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | | 95 | % CI | ;i | | 959 | 95% CI | |
| n** | n | % | LL | UL | n** | n | % | LL | UL |
| | | | | | | | | | 1 |
| | n** | | N | N = 95 | N = 95% CI | N = 95% CI | N = 95% CI | N = N = N = | N = N = 95% CI 95° |

RSV-Ld = Low dose ChAd155-RSV vaccine (5 x 109 vp)

RSV-Md = Middle dose ChAd155-RSV vaccine (1.5 x 10<sup>10</sup> vp)

RSV-Hd = High dose ChAd155-RSV vaccine (5 x 10<sup>10</sup> vp)

Placebo-Ld = Non-active control (0.5 ml)

Placebo-Md = Non-active control (0.15 ml)

Placebo-Hd = Non-active control (0.5 ml)

RSV = ChAd155-RSV vaccine (low/ middle/high dose pooled groups)

Placebo = Non-active control (0.5/0.15/0.5 ml pooled groups)

N = number of subjects in each group

n\*\* = number of cases in each category

n/%= number/percentage of subjects reporting at least once the case

95%CI= Exact 95% confidence interval; LL = lower limit, UL = upper limit

Please note – Single episode can be considered in single category depending on the highest severity symptom experienced

204838 (RSV PED-002) Statistical Analysis Plan Final

### Template 54 Number and percentage of subjects reporting the RSV infection of maximum severity by number of events experienced between vaccination dose 1 up to D366/D731 visit <Exposed Set>

| | | | otal | | | |
|---|---|---|---|---|---|---|
| | | | | | 95% CI | |
| Characteristics | Categories | N | n | % | LL | UL |
| RSV asymptomatic (Excluding RSV-RTI, RSV-LRTI, RSV-severe LRTI or RSV-very severe LRTI) | 0 | | | | | |
| • , | 1 | | | | | |
| | 2 | | | | | |
| RSV-RTI (Excluding RSV-LRTI, RSV severe or very severe LRTI) | 0 | | | | | |
| , | 1 | | | | | |
| RSV-LRTI (Excluding RSV severe or very severe LRTI) | 0 | | | | | |
| | 1 | | | | | |
| RSV-Severe LRTI Excluding RSV very severe LRTI) | 0 | | | | | |
| | 1 | | | | | |
| RSV-very severe LRTI | 0 | | | | | |
| | 1 | | | | | |

RSV-Ld = Low dose ChAd155-RSV vaccine (5 x 109 vp)

RSV-Md = Middle dose ChAd155-RSV vaccine (1.5 x 10<sup>10</sup> vp)

RSV-Hd = High dose ChAd155-RSV vaccine (5 x 10<sup>10</sup> vp)

Placebo-Ld = Non-active control (0.5 ml)

Placebo-Md = Non-active control (0.15 ml)

Placebo-Hd = Non-active control (0.5 ml)

RSV = ChAd155-RSV vaccine (low/ middle/high dose pooled groups)

Placebo = Non-active control (0.5/0.15/0.5 ml pooled groups)

N = number of subjects in each group

n = number of subjects in a given category

% =100\*n/N

LL, UL for percentage = Exact 95% Lower and Upper confidence limits

Please note – Single episode will be considered in single category depending on the maximum severity experienced

204838 (RSV PED-002) Statistical Analysis Plan Final

## Template 55 Number (%) of subjects reported solicited local symptoms during the 7-day (Days 1-7) post-vaccination period following each dose and across doses <Exposed Set>

| | | | <each group=""></each> | | | | |
|---|---|---|---|---|---|---|---|
| | | | | | | 9: | 5 % CI |
| Dose | Symptom | Туре | N | n | % | LL | UL |
| DOSE 1 | Pain | All | | | | | |
| | | Grade 3 | | | | | |
| | Redness (mm) | All | | | | | |
| | | >20 | | | | | |
| | Swelling (mm) | All | | | | | |
| | | >20 | | | | | |
| DOSE 2 | Pain | | | | | | |
| | Redness (mm) | | | | | | |
| | Swelling (mm) | | | | | | |
| ACROSS DOSEs | Pain | | | | | | |
| | Redness (mm) | | | | | | |
| | Swelling (mm) | | | | | | |

#### <each group>:

RSV-Ld = Low dose ChAd155-RSV vaccine (5 x 109 vp)

RSV-Md = Middle dose ChAd155-RSV vaccine (1.5 x 10<sup>10</sup> vp)

RSV-Hd = High dose ChAd155-RSV vaccine (5 x 10<sup>10</sup> vp)

Placebo-Ld = Non-active control (0.5 ml)

Placebo-Md = Non-active control (0.15 ml)

Placebo-Hd = Non-active control (0.5 ml)

For each dose:

N = number of subjects with the corresponding documented dose

n/% = number/percentage of subjects reporting the type of symptom at least once following the corresponding dose For Across dose:

N = number of documented doses

n/% = number/percentage of doses followed by at least one type of symptom

95%CI= Exact 95% confidence interval; LL = lower limit, UL = upper limit

The maximum intensity of local injection site redness/swelling was coded as follows:

- 1: > 0.1 mm to < 5 mm
- $2: \geq 5 \text{ mm to} \leq 20 \text{ mm}$
- 3: > 20 mm

204838 (RSV PED-002) Statistical Analysis Plan Final

### Template 56 Number (%) of subjects reported solicited general symptoms during the 7-day (Days 1-7) post-vaccination period following each dose and across dose <Exposed Set>

| Dose | | | <each group=""></each> | | | | |
|---|---|---|---|---|---|---|---|
| | | | | | | 95 % C | |
| | Symptom | Туре | N | n | % | LL | UL |
| DOSE 1 | Drowsiness | All | | | | | |
| | | Grade 3 | | | | | |
| | | Related | | | | | |
| | Irritability/Fussiness | All | | | | | |
| | | Grade 3 | | | | | |
| | | Related | | | | | |
| | Loss of appetite | All | | | | | |
| | | Grade 3 | | | | | |
| | | Related | | | | | |
| | Fever (Axillary) (°C) | All (≥37.5) | | | | | |
| | | >39.5 | | | | | |
| | | Related | | | | | |
| DOSE 2 | Drowsiness | | | | | | |
| | Irritability/Fussiness | | | | | | |
| | Loss of appetite | | | | | | |
| | Fever (Axillary) (°C) | | | | | | |
| ACROSS DOSE | Drowsiness | | | | | | |
| | Irritability/Fussiness | | | | | | |
| | Loss of appetite | | | | | | |
| | Fever (Axillary) (°C) | | | | | | |

#### <each group>:

RSV-Ld = Low dose ChAd155-RSV vaccine (5 x 109 vp)

RSV-Md = Middle dose ChAd155-RSV vaccine (1.5 x 10<sup>10</sup> vp)

RSV-Hd = High dose ChAd155-RSV vaccine (5 x 10<sup>10</sup> vp)

Placebo-Ld = Non-active control (0.5 ml)

Placebo-Md = Non-active control (0.15 ml)

Placebo-Hd = Non-active control (0.5 ml)

For each dose:

N = number of subjects with the corresponding documented dose

n/% = number/percentage of subjects reporting the symptom at least once following the corresponding dose For Across dose:

N = number of documented doses

n/% = number/percentage of doses followed by at least one type of symptom

95%CI= Exact 95% confidence interval; LL = lower limit, UL = upper limit

Temperatures were coded as follows:

1: ≥ 37.5 °C to ≤ 38.5 °C

2: > 38.5 °C to  $\leq 39.5$  °C

3: > 39.5°C